### 1. TITLE PAGE

A Double-Blind, Controlled by Conventional BCG, Dose-escalation Phase I Study, to Evaluate Safety, Tolerability and Immunogenicity of a *Mycobacterium bovis* BCG (Bacillus Calmette-Guérin) Vaccine, 1331 Danish Strain, Live Attenuated and Recombinant for the Expression of Human Respiratory Syncytial Virus Nucleoprotein (N) in Healthy Males Within 18 and 50 Years of Age

### Final Integrated Clinical/Statistical Report

**Trial Number code:** 1) Public Health Institute of Chile Registry (N° 4060).

2) Clinicaltrials.gov identifier: NCT03213405.

**Development Phase:** Phase I

**Indication Studied:** Respiratory Syncytial Virus Infections

**Product:** rBCG-N-hRSV 001

Form/Route: Intradermal

**Sponsor:** Pontificia Universidad Católica de Chile

**Principal Investigator:** Alexis M. Kalergis, PhD

Clinical/Medical Monitor: Katia Abarca, MD
Laboratory Monitor: Susan Bueno, PhD

Pharmacovigilance (Safety Jose Vice

Narratives):

Biostatistician:

Jose Vicente Gonzalez, PhD

Clinical Trial Initiation

Date:

June 27 2017

Jaime Cerda, MD

**Clinical Trial Completion** 

January 8 2018

Date:

**Date of the report:** January 8 2018

Version Number: 0.2

This study was performed in compliance with Good Clinical Practice

## 2. TABLE OF CONTENTS

| | | <u>Page</u> |
|---|---|---|
| 1. | TITLE PAGE | I |
| 2. | TABLE OF CONTENTS | II |
| 3. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | VI |
| 4. | LIST OF TABLES | VII |
| 5. | LIST OF FIGURES | IX |
| 6. | ETHICS | 1 |
| 6.1. | Independent Ethics Committee (IEC) or Institutional Review Board (IRB) 1 | |
| 6.2. | Ethical Conduct of the Study | 1 |
| 6.3. | Subject Information and Consent | 1 |
| 7. | INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE | 2 |
| 7.1. | Administrative Structure at the Clinical Sites | 2 |
| 7.2 | Administrative Structure for the Trial | 2 |
| 8. | INTRODUCTION | 3 |
| 9. | STUDY OBJECTIVES | 5 |
| 10. | INVESTIGATIONAL PLAN | 6 |
| 10.1. | Overall Study Design and Plan Description | 6 |
| 10.2. | Rationale for Study Design | 7 |
| 10.3. | Selection of Study Population | 8 |
| 10.3.1. | Inclusion Criteria | 8 |
| 10.3.2. | Exclusion Criteria | 8 |
| 10.3.3. | Removal of Subjects from Therapy or Assessment | 10 |
| 10.4. | Vaccinations/Treatments | 11 |
| 10.4.1. | Vaccinations/Treatments Administered | 11 |
| 10.4.2. | Identity of Investigational Product(s) | 11 |
| 10.4.3. | Method of Assigning Subjects to Study Groups | 11 |
| 10.4.4. | Selection of Doses in the Study | 11 |
| 10.4.5. | Selection and Timing of Dose for Each Subject | 12 |
| 10.4.6. | Blinding 12 | |
| 10.4.7. | Prior and Concomitant Therapy 12 | |

| 10.4.8. | . Treatment Compliance | 12 |
|---|---|---|
| 10.5. | Efficacy/Immunogenicity and Safety Variables | 12 |
| 10.5.1. Efficacy/Immunogenicity and Safety Measurements Assessed and Flow Chart | | |
| 10.5.2. | . Appropriateness of Measurements | 13 |
| 10.5.3. | . Primary Efficacy/Immunogenicity Endpoints | 13 |
| 10.5.4. | . Primary Safety Endpoints | 13 |
| 10.5.5. | . Secondary Efficacy/Immunogenicity and Safety Endpoints | 14 |
| 9.5.6. | Drug Concentration Measurements | 14 |
| 10.6. | Data Quality Assurance | 14 |
| 10.6.1. | . Data Collection and Management | 14 |
| 10.6.1. | .1. Data Recording Methods | 15 |
| 10.6.1. | .2. Subject Identifiers | 15 |
| 10.6.2. | . Monitoring, Auditing, and Archiving | 15 |
| 10.6.3. | . Database Lock | 16 |
| 10.7. | Statistical Methods Planned in the Protocol and Determination of Sample Size | 16 |
| 10.7.1. | . Sample Size | 16 |
| 10.7.2. | . Statistical Analysis Plan | 17 |
| 11. | STUDY SUBJECTS | 18 |
| 11.1. | Disposition of Subjects | 18 |
| 11.1.1 | Demographic Data by Study Group | 18 |
| 11.1.2. | . Summary of Prior and Concurrent Medical Conditions | 18 |
| 11.1.3. | . Visit Schedule | 18 |
| 11.1.4. | . Vital Signs Grading 19 | |
| 11.2. | Protocol Deviations 20 | |
| 12. | EFFICACY/IMMUNOGENICITY EVALUATION 21 | |
| 12.1. | Analysis Populations 21 | |
| 12.2. | Demographics and Other Baseline Characteristics 21 | |
| 12.2.1. | . Prior and Concurrent Medical Conditions 22 | |
| 12.2.2. | . Prior and Concomitant Medications 22 | |
| 12.3. | Measurements of Treatment Compliance 22 | |
| 12.4. | Efficacy/Immunogenicity Results and Tabulations of Individual Subject Data | 22 |
| 12.4.1. | . Methodology and Primary Statistical Analysis of Efficacy/ Immunogenicity Data | 22 |

| 12.4.1. 1 Handli | ing of Dropouts or Missing Data 23 | |
|---|---|---|
| 12.4.2. Tabulation of Individual Response Data 23 | | |
| 12.4.3. Efficacy/Immunogenicity Conclusions 24 | | |
| 13. SAFETY | Y EVALUATION 25 | |
| 13.1. Extent o | f Exposure 25 | |
| 13.2. Adverse | Events (AEs)25 | |
| 13.2.1. Brief Su | mmary of Adverse Events 25 | |
| 13.2.2. Display | of Adverse Events 26 | |
| 13.2.2.1. S | Solicited AEs 28 | |
| 12.2.2.2. U | Unsolicited AEs 28 | |
| 13.2.3. Analysis | s of Adverse Events 30 | |
| 13.3. Deaths, | Other Serious Adverse Events, and | Other Significant Adverse Events 30 |
| _ | of Deaths, Other Serious Adverse E<br>30 | vents, and Other Significant Adverse Events |
| 13.3.1.1. Deaths | s 31 | |
| 13.3.1.2. Seriou | s Adverse Events 31 | |
| 13.3.1.3. | Other Significant Adverse Events | 31 |
| 13.3.2. Narrativ<br>Events | es of Deaths, Other Serious Advers | e Events, and Other Significant Adverse 31 |
| 13.3.3. Analysis<br>Adverse Events | | erious Adverse Events, and Other Significant |
| 13.4. Clinical | Laboratory Evaluation 32 | |
| 13.4.1. Individu | al Laboratory Measurements and A | bnormal Laboratory Values 32 |
| 133.4.2. H | Evaluation of Each Laboratory Para | meter 34 |
| 12.4.2.1. I | Laboratory Values over Time 34 | |
| 13.4.2.2. I | Individual Subject Changes 34 | |
| 13.4.2.3. I | Display of Laboratory Results | 36 |
| 13.4.2.4. | Chemistry Results | 36 |
| 13.4.2.5. H | Hematology Results | 36 |
| 13.4.2.6. U | Urinalysis Results 38 | |
| 13.5. Vital Sig | gns, Physical Exam Findings, and C | other Observations Related to Safety 38 |
| 13.5.1. Vital Signs Grading 39 | | |
| 13.5.2. Abnorm | al Vital Signs 39 | |

- 13.6. Concomitant Medications 40
- 12.7. Pregnancies (if applicable) 40
- 12.8. Safety Conclusions 40
- 14. DISCUSSIONS AND OVERALL CONCLUSION 41
- 15. TABLES, FIGURES, AND GRAPHS REFERRED TO BUT NOT INCLUDED IN THE TEXT 44
- 16. REFERENCE LIST 70

### 3. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE: Adverse Events

ARTIs: Acute Respiratory Tract Infections

BCG: Bacillus Calmette-Guérin

BCG-WT: Nonrecombinant, wild type Bacillus Calmette-Guérin

**CFU: Colony Forming Units** 

IC: Informed Consent DSMB: Data and Safety Monitoring Board

FI-rRSV: Formalin-inactivated vaccine

ID: Identification Number

HRP: Horseradish Peroxidase

hRSV: Human Respiratory Syncytial Virus

IFN-γ: Interferon Gamma

IL-2: Interleukin 2

NA: Not Applicable

N-RSV: Respiratory Syncytial Virus Nucleoprotein

PPD: purified protein derivative of Mycobacterium tuberculosis

rBCG-N-hRSV: recombinant Mycobacterium bovis BCG vaccine expressing the nucleoprotein

of hRSV

Th: T helper cells

TNF-α: Tumor necrosis factor alpha

### 4. LIST OF TABLES

| | <u>Page</u> |
|---|---|
| 1 Table I: Study design | 7 |
| 2 Table II: Safety and Efficacy/Immunogenicity evaluation | 13 |
| 3 Table III: Subjects receiving investigational product | 17 |
| 4 Table IV: Protocol deviation by each subject | 19 |
| 5 Table V: Immunogenicity individual response | 22 |
| 6 Table VI: SAE from the three cohorts, to date January 3, 2018 | 25 |
| 7 Table VII: Cohorts A, B and C, at day 30 | 25 |
| 8 Table VIII: Cohorts A, B and C, to date January 8th, 2018 | 26 |
| 9 Table IX: Listing of local adverse events by subjects | 27 |
| 10 Table X: Listing of general adverse events by subjects | 32 |
| 11 Table XI: Serious adverse events | 48 |
| 12 Table XII: Laboratory adverse events from cohort A, B and C at day 30 | 50 |
| 13 Table XIII: Vital signs grading | 52 |
| 14 Table XIV: Abnormal vital signs | 53 |
| 15 Table XV: Cohort by subject's number | 58 |
| 16 Table XVI: Demographic data by study group | 59 |
| 17Table XVII. Study Visit Schedule | 59 |
| 18 Table XVIII: Immunogenicity individual response | 61 |
| 19 Table XIX: Solicited general adverse events grade 3 | 64 |
| 20 Table XX: Number of Non-Solicited clinical adverse events | 64 |

| 21 Table XXI: Grade 3 laboratory adverse events and follow-up (to date) | 66 |
|-------------------------------------------------------------------------|----|
| 22 Table XXII: Biochemistry results from the 3 laboratory cohorts | 68 |
| 23 Table XXIII: Haematology results from all laboratory cohorts | 69 |
| 24 Table XXIV: Haematology results from all 3 clinical cohorts | 70 |
| 25 Table XXV: Urinalysis results from all laboratory cohorts | 70 |
| 26 Table XXVI: Urinalysis results from all clinical cohorts | 71 |
| 27 Table XXVI: Vital signs from all clinical cohorts | 71 |

| 5. | LIST OF FIG | URES | | | |
|---|---|---|---|---|---|
| | | | | | Page |
| 1 <u>F</u> i | igure 1: Clinical study | flow diagram | • | | 17 |
| | The phase 1 stud | y was a double blind, dos | se escalation tr | ial performed in heal | thy male |
| | adults. Each cohort incl | uded 6 volunteers vaccina | ated with escala | ating doses of rBCG- | N-hRSV |
| | $(5x10^3 \text{ CFU}; 5x10^4 \text{ CF})$ | U; 1x10 <sup>5</sup> CFU) and 2 vo | olunteers vacci | nated with the standa | ard BCG |
| | (BCG-WT) (2x10 <sup>5</sup> CFU | ). Furthermore, the safety | data for each | cohort were evaluated | l after all |
| | subjects in each group escalation could continu | had reached 30 days pos | t-vaccination to | o determine whether | the dose |
| 2 <u>F</u> i | igure 2: Measurement o | of specific cellular imm | une responses | by flow cytometry | against PPD |
| antig | ens (in black) and hRS | V-N protein (in white). | 57 | | |
| | The results are ex | pressed as fold changes (le | og2) compared | l with visit 1 (day 0) f | or CD4+ |
| | and CD8+ T cells that se | ecreted IL-2 and TNF-α at | 14 and 30 days | s post-vaccination for | the three |
| | dose groups receiving rl | BCG-N-hRSV (5x10 <sup>3</sup> CFU | U, 5x10 <sup>4</sup> CFU, | 1x10 <sup>5</sup> CFU) and for E | 3CG-WT |
| | $(2x10^5 \text{ CFU}).$ | | | | |
| 3 <u>F</u> | igure 3: Measurement | of specific cellular in | nmune respor | nses by ELISPOT | against PPD |
| antig | ens (in black) and hRS | V-N protein (in white) | | 59 | |
| | The results are ex | pressed as fold changes (le | og2) compared | l with visit 1 (day 0) f | for CD4+ |
| | and CD8+ T cells that | secreted IFN-γ and IL-2 a | at times 14, 30 | and 180 days post-va | ccination |
| | for the three dose grou | ps receiving rBCG-N-hRS | SV (5x10 <sup>3</sup> CFU | , 5x10 <sup>4</sup> CFU, 1x10 <sup>5</sup> C | CFU) and |
| | for BCG-WT (2x10 <sup>5</sup> C | CFU). | | | |
| 4 <u>F</u> i | igure 4: Measurement o | of PPD- and hRSV-N-sp | ecific humora | ıl immune responses | s (in black or |
| <u>white</u> | e bars, | respectively) | by | indirect | ELISA |
| <u>assay</u> | <u></u> | | | | 60 |

The results are expressed as fold changes (log10) compared with visit 1 (day 0) at 60, 120 and 180 days post-vaccination for the three dose groups of rBCG-N-hRSV (5x10<sup>3</sup> CFU, 5x10<sup>4</sup> CFU,  $1x10^5$  CFU) and for BCG-WT ( $2x10^5$  CFU).

### 6. ETHICS

# 6.1. Independent Ethics Committee (IEC) or Institutional Review Board (IRB)

The first signed informed consent was provided to the Institutional Ethics Committee on June 19<sup>th</sup>, 2017. The trial was approved by both, the Institutional Ethical Committee of the Pontificia Universidad Católica de Chile (document number 15-216) and the Chilean Public Health Institute (Instituto de Salud Pública de Chile, document number EC819077/16).

### **6.2.** Ethical Conduct of the Study

The trial (clinicaltrials.gov NCT03213405) was conducted in Santiago of Chile, in a single center (Clinical Research Center of Pontificia Universidad Católica de Chile (CICUC)). The protocol was conducted according to the current Tripartite Guidelines of Good Clinical Practice, Declaration of Helsinki (17) and local regulations (Instituto de Salud Pública). Written informed consent was obtained from each participant prior to study entry. A Data Safety Monitoring Board (DSMB) evaluated safety data for each dose cohort after all subjects of the group reached day 30 of follow up to determine whether the dose escalation could continue.

### 6.3. Subject Information and Consent

The Informed Consent (IC) document version 3.0 dated March 10<sup>th</sup> of 2017 was used. During the screening visit, the study was explained to each individual and each subject signed the consent form in duplicate. One copy was provided to the subject and the other copy was archived in the subject file for this study. The identity of each participant was confirmed and documented using a unique, study-specific identification number (ID) which was archived in the study file.

All the volunteers signed the IC approved by the Institutional Ethic Committee of the Facultad de Medicina of the Pontificia Universidad Católica de Chile, before starting the first screening visit.

## 7. INVESTIGATORS AND STUDY ADMINISTRATIVE STRUCTURE

### 7.1. Administrative Structure at the Clinical Sites

**Lead Site** 

Principal Investigator: Alexis M. Kalergis, PhD

Clinic Manager: Katia Abarca, MD

Laboratory Manager: Susan Bueno, PhD

Study Coordinator: Carolina Iturriaga, RN

Laboratory Supervisor: Susan Bueno, PhD and Alexis M. Kalergis, PhD

#### 7.2. Administrative Structure for the Trial

Principal Investigator: Alexis M. Kalergis, PhD

Scientific Lead: Alexis M. Kalergis, PhD

Medical Monitor: Katia Abarca, MD

Laboratory Supervisor Susan Bueno, PhD

Clinical Project Manager: Carolina Iturriaga, RN

Biostatistician: Jaime Cerda, MD, Pontificia Universidad

Católica de Chile.

Pharmacovigilance (Safety Narratives): -Jose Vicente Gonzalez, PhD

Report Author: Alexis M. Kalergis, PhD

Statistical and Data Coordinating Center: Pontificia Universidad Católica de Chile

Clinical Monitoring: SMOLAM LTDA

### 8. INTRODUCTION

The human respiratory syncytial virus (hRSV) is of great public health significance causing acute respiratory tract infections (ARTIs) in children worldwide (1). hRSV can cause mild manifestations such as rhinorrhea, cough and congestion, to severe manifestations such as alveolitis, bronchiolitis and pneumonia (2). Importantly, worldwide hRSV infections are responsible for more than 3 million hospitalizations and more than 33 million ARTI episodes each year among children up to five years (1).

No licensed vaccine is currently available to prevent hRSV infection. The only current hRSV treatment is a humanized monoclonal antibody that targets the F protein of the virus. This approach is only used as a prophylactic treatment, mainly for high-risk infants to prevent the most severe symptoms of hRSV infection (4). An early hRSV vaccine attempt utilized a formalininactivated vaccine (FI-hRSV) in the 1960s (5). Unfortunately, the administration of this vaccine caused hospitalization in up to 80% of vaccinated children, triggering an exacerbation of the disease upon exposure to natural infection (6, 7). Therefore, there is a need to develop a safe and effective hRSV vaccine that induces a protective immunological response, but without enhancing pulmonary disease after hRSV infection. It has been shown that in children with acute hRSV bronchiolitis a predominantly T helper (Th)-2 cell biased response occurs and may be responsible for the pathologic outcomes (8). Further, a reduction in the frequency of  $\gamma\delta$  T cells producing IFNy has also been observed in samples from children presenting hRSV disease (9). These previous studies suggest that immunologic protection against hRSV involves a type 1-biased immune response (including CD4+ Th1 cells producing IFN-γ, TNF-α and IL-2), whereas enhanced hRSV disease is associated with a type 2-biased immune response (including CD4+ Th2 cells producing IL-4, IL-5 and IL-13). Therefore, a current view is that optimal hRSV vaccines should induce potent CD4<sup>+</sup> Th1 cell responses, and not CD4<sup>+</sup> Th2 cell responses. According to the 2017 report from Program for Appropriate Technology in Health (PATH, www.path.org), multiple hRSV vaccine candidates are in clinical evaluation including live-attenuated, particle-based and adenovirus-vectored approaches (10).

A vaccine candidate consisting on a recombinant *Mycobacterium bovis* (BCG) that expresses the nucleoprotein (N) of hRSV (rBCG-N-hRSV) has been developed by the team of Dr. Alexis Kalergis at the Pontificia Universidad Católica de Chile (11). BCG has been historically

used to prevent tuberculous meningitis and miliary TB disease and has been applied more than 4 billon times since its introduction in most countries around the world (12). In addition, BCG induces strong Th1, and not Th2 immune responses in both, animal models and in humans, and therefore is hypothesized to be an ideal vector for a vaccine directed against hRSV infection (13). Importantly, immunization with rBCG-N-hRSV in mice prevented lung associated damage from hRSV infection, decreased inflammatory cell infiltrations and induced an early recruitment of CD4<sup>+</sup> and CD8<sup>+</sup>T cells to the lungs (11, 14, 15). In addition, rBCG-N-hRSV generated an effective neutralizing antibody response in RSV-infected mice (16).

### 9. STUDY OBJECTIVES

The primary objective of this study was to characterize the safety and tolerability of escalating doses of the rBCG-N-hRSV vaccine, including doses of  $5x10^3$ ,  $5x10^4$  and  $1x10^5$  CFU in healthy adult males 18 to 50 years of age.

The secondary objectives included characterization of the immune responses induced against the hRSV-N and against mycobacterial antigens with escalating doses of the rBCG-N-hRSV vaccine.

### 10. INVESTIGATIONAL PLAN

### 10.1. Overall Study Design and Plan Description

This was a phase I, double blind trial to evaluate the safety, tolerability and immunogenicity of an investigational recombinant BCG vaccine expressing hRSV-N compared to a control, nonrecombinant wild type BCG vaccine (conventional BCG) within each cohort, performed in healthy adult males 18 to 50 years of age.

After a full clinical and laboratory evaluation to exclude those with underlying diseases, immunodeficiency and latent tuberculosis infection per inclusion and exclusion criteria, the participants were enrolled into three cohorts. Within each cohort, the participants were randomly and in a blinded-manner assigned to receive the tested vaccine (rBCG-N-hRSV) or the control vaccine (conventional BCG).

Each cohort was vaccinated according to their assigned groups followed by a period of 6 months of follow-up. Safety data was evaluated by a Data and Safety Monitoring Board (DSMB), that determined whether, according to previously defined parameters, the escalation to the next cohort was possible, or whether the study needed to be halted due to safety concerns. Blood, saliva and urine samples were obtained pre-vaccination and on days 14, 30 and 180 post-vaccination, and (peripheral blood mononuclear cells) PBMCs were purified from the blood for cellular immune assays and serum isolated for humoral immune assays. The study design can be seen in Table I.

Table I: Study design

| Cohort | Number of vaccinated | Safety analysis by<br>CIMD | Follow up | Study completion |
|---|---|---|---|---|
| A | n=8 6 rBCG-N-hRSV 5x10^3 2 BCG 2x10^5 | Day 30 | Until day 180 | n=8 per group<br>TOTAL<br>VACCINATED THAT |
| В | n=8 6 rBCG-N-hRSV 5x10^4 2 BCG 2x10^5 | Day 30 | Chartary 100 | COMPLETED THE<br>STUDY=24 |

| С | n=8 |
|---|-------------------------|
| | 6 rBCG-N-hRSV<br>1x10^5 |
| | 2 BCG 2x10^5 |

Samples were taken from all enrolled subjects at different time-points for the following purposes:

- Day 0: Venous blood for basal immunogenicity assays (cellular and humoral, 26 ml total).
- Day 7: Venous blood (16 ml) for laboratory adverse events study. Venous blood (4 ml), urine (10 ml) and saliva (>1 ml) for BCG excretion studies.
- Day 14: Venous blood (16 ml) for laboratory adverse events study. Venous blood immunogenicity assays (cellular and humoral, 26 ml total). Venous blood (4 ml), urine (10 ml) and saliva (>1ml) for BCG excretion studies.
- Day 30: Venous blood (16 ml) for laboratory adverse events study. Venous blood immunogenicity assays (cellular and humoral, 26 ml total). Venous blood (4 ml), urine (10 ml) and saliva (>1ml) for BCG excretion studies.
- Day 60: Venous blood (16 ml) for laboratory adverse events study. Venous blood immunogenicity assays (cellular and humoral, 26 ml total). Venous blood (4 ml), urine (10 ml) and saliva (>1 ml) for BCG excretion studies.
- Day 120: Venous blood (16 ml) for laboratory adverse events study. Venous blood immunogenicity assays (cellular and humoral, 26 ml total). Venous blood (4 ml), urine (10 ml) and saliva (>1ml) for BCG excretion studies.
- Day 180: Venous blood (16 ml) for laboratory adverse events study. Venous blood immunogenicity assays (cellular and humoral, 26 ml total). Venous blood (4 ml), urine (10 ml) and saliva (>1ml) for BCG excretion studies.

### **10.2.** Rationale for Study Design

Because this was a first-in-human phase I trial to study a novel recombinant BCG vaccine designed to protect against both, hRSV and *Mycobacterium tuberculosis* infections, a careful dose escalation trial was designed with safety monitoring between escalation groups. The specific doses were selected based on the standard dose of BCG utilized in Chile for infant vaccination to protect against TB. The first group received a recombinant RSV-BCG vaccine dose that was equivalent to 1/100<sup>th</sup> of the standard dose of non-recombinant BCG licensed for use in infants in Chile. The second group received a recombinant RSV-BCG vaccine dose that was equivalent to 1/10<sup>th</sup> of the standard dose of non-recombinant BCG licensed for use in infants in Chile. The third group received a recombinant RSV-BCG vaccine dose that was equivalent to a full dose of non-recombinant BCG licensed for use in infants in Chile. The third group

could provide the advantage of inducing protective immunity against both, hRSV and TB infection and disease. If shown to be safe and effective, this one recombinant vaccine could replace standard BCG vaccination currently given to protect against TB. The reason to perform a double blind study was to assure that the study would not be biased. It is worth mentioning that, due that BCG vaccination is mandatory in Chile, all enrolled subjects were BCG-positive.

### **10.3.** Selection of Study Population

#### 10.3.1. Inclusion Criteria

The inclusion criteria were as follows:

- Chilean male between 18 and 50 years old.
- Evidence of voluntary participation through documentation of informed consent.
- Good health, according to the medical history, physical examination and normal laboratory test.
- A history of vaccination with BCG once or twice during the participant's life.

  In this population, the vaccine will work as a boost for BCG.

### 10.3.2. Exclusion Criteria

The exclusion criteria were as follows:

- Symptoms or diagnosis suggesting any type of systemic disease including renal, liver, cardiovascular or pulmonary impairment, immunodeficiency, autoimmune diseases, malignancies, psychiatric or other conditions that could interfere with the interpretation of the results or compromise the health of the participants.
- Body mass index lower than 19 and higher than 30 kg/m2 and/or weight under 50 kg.

- Not being able to attend all the study visits (face-to-face and telephone contacts)
  or follow the specified instructions (fasting, avoidance of intense physical
  exercise during the 24 hours preceding the study visits and 72 hours postvaccination).
- Signs of latent or active infection with *Mycobacterium tuberculosis*: QuantiFERON-TB positive test or Chest X-ray suggesting Tuberculosis (TB).
- Positive screening for the human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) and hepatitis C virus (HCV).
- Evidence of primary or secondary immunodeficiency, determined by history, physical test and levels of serum immunoglobulins and lymphocytes subpopulations at the screening.
- Use of immunosuppressing drugs during the last 6 months prior to, or during the study.
- Use of inhaled corticosteroids for bronchial hyper-reactivity during the last year.
- History of close contact exposure to patients with Tuberculosis or other mycobacterial infections, even if under treatment.
- History of substance abuse (drugs or alcohol), according to DMS IV (See footnote\*).
- Occurrence of any serious adverse events associated with previous BCG vaccination.
- History of severe allergic reactions or anaphylaxis to vaccines.
- History of severe infections (use of IV antibiotics, latent TB, herpes zoster) six months previous to screening.
- Refusal of condom use during sexual contact or abstinence from sexual activity during the study (See footnote\*\*).
- Administration of immunoglobulins or blood-derived products six months previous to participation in the study or planned use of these products during the study.
- Eczema at the vaccination site (deltoid zone).
- Antecedents of keloid scar.

- Being vaccinated with BCG during the last 10 years.
- History of being vaccinated with BCG three or more times or the presence of three BCG scars.
- Receipt of other investigational products 30 days previous to the study.
- Administration of any vaccine 8 weeks prior to recruitment.
- Administration of any other vaccine during the first 30 days after vaccination with the rBCG-hRSV.
- Acute illness symptoms and/or feverish symptoms at the time, or during the last seven days prior to enrollment (fever defined as an oral or axillary temperature of >38°C).
- (\*) Substance abuse (drugs or alcohol): Maladaptive pattern of substance abuse that leads to a clinically significant mental or physical deterioration during the previous twelve months. Clinically significant deterioration would include evidence of any of the following: inability to complete personal and/or professional obligations; use of drugs or alcohol in dangerous situations, such as driving a vehicle; and legal problems related to drug or alcohol use.
- (\*\*) Given the remote possibility of negative effects produced by the vaccination on sperm, only volunteers that are not planning on conceiving a child during the study duration were enrolled. During each visit, abstinence or the use of effective contraceptive device will be confirmed.

### 10.3.3. Removal of Subjects from Therapy or Assessment

18 subjects were not enrolled in the study because they presented one or more exclusion parameters, including: Gilbert Syndrome, hepatitis B and latent *Mycobacterium tuberculosis* infection, HIV infection, three (3) BCG scars and screening tests out of the normal range. All enrolled subjects completed the trial. This was due to good safety results. Subjects were not enrolled due to non-compatible clinical or laboratory screening results before enrollment for the trial. These data are in section 10.7.1 below.

### 10.4. Vaccinations/Treatments

#### 10.4.1. Vaccinations/Treatments Administered

Two vaccines were administrated during this study. Two volunteers per cohort were vaccinated with conventional BCG full dose ( $2x10^5$  CFU). Six volunteers per cohort were vaccinated with escalating doses of rBCG-N-hRSV (cohort A  $5x10^3$  CFU, cohort B  $5x10^4$  CFU, and cohort C  $1x10^5$  CFU). These vaccines were administered as an intradermal injection at study entry.

#### 10.4.2. Identity of Investigational Product(s)

The study vaccine consisted of a novel, live attenuated, recombinant *Mycobacterium bovis* BCG (Bacillus Calmette-Guérin), Danish strain 1331, expressing the nucleoprotein (N) from the human respiratory syncytial virus (hRSV serogroup A2, strain 13018-8, obtained from the Institute of Public Health of Chile (11)), called rBCG-N-hRSV. The vaccine was designed at the Pontificia Universidad Católica de Chile and manufactured under cGMP conditions at IDT Biologika (former AERAS TB Vaccine Foundation)(USA).

### 10.4.3. Method of Assigning Subjects to Study Groups

This phase I study was performed as a double blind, randomized trial. The study was organized in three groups, each including 8 subjects (total number of subjects was 24). Each group was created using the random.org software and the random-sequence-generator command for 8 numbers (1 to 8). The first 6 numbers were assigned to the vaccine under study and the last 2 numbers to the control vaccine.

### 10.4.4. Selection of Doses in the Study

The doses were selected according to the publications by Cautivo, K.M. *et al* and by Céspedes, P.C. *et al*. (14,15), which describe that 1x10^8 CFU and 3x10^5 CFU were used respectively to immunize mice, showing safety and efficacy in mice in both studies. Further, the current recommended dose for BCG was also considered as part of the dose selection (<a href="https://www.who.int/immunization\_standards/vaccine\_quality/118\_bcg/en/">https://www.who.int/immunization\_standards/vaccine\_quality/118\_bcg/en/</a>). Because this was a first-in-human phase I trial to study a novel recombinant BCG vaccine designed to protect against

both, hRSV and *Mycobacterium tuberculosis* infections, a careful dose escalation trial was designed with safety monitoring between escalation groups. The dose escalation in the clinical trial began with 1/100<sup>th</sup> of the standard full dose licensed for infant BCG vaccination in Chile, then proceeded to 1/10<sup>th</sup> of the standard full dose licensed for infant BCG vaccination in Chile, and then proceeded to the standard full dose licensed for infant BCG vaccination in Chile.

#### 10.4.5. Selection and Timing of Dose for Each Subject

This study followed a careful dose escalation strategy, with pauses by the DSMB to review the data after all subjects in each cohort had been evaluated for at least 30 days post-vaccination and before proceeding to the following escalation dose. In cohorts A, B and C the doses of rBCG-N-hRSV were  $5x10^3$  CFU,  $5x10^4$  CFU and  $1x10^5$  CFU, respectively. The BCG-WT dose for all control subjects was the same, which was the standard full dose ( $2x10^5$  CFU) licensed for use in infants in Chile.

### **10.4.6.** Blinding

This study was a double blinded study in which both, the participants and personnel were blinded to all the groups in the study.

### 10.4.7. Prior and Concomitant Therapy

NA

#### **10.4.8.** Treatment Compliance

N/A

### 10.5. Efficacy/Immunogenicity and Safety Variables

### 10.5.1. Safety Measurements Assessed and Flow Chart

To assess the safety of the vaccine, a series of clinical tests to assess possible adverse events was performed. These tests can be seen in Table II. Adverse events (severe, local, general) were recorded through day 180 and laboratory tests were performed at days 1, 2, 3, 7, 14, 30, 60, 120 and 180 post-vaccination.

Table II: Safety and Efficacy/Immunogenicity evaluation.

| Safety test | | |
|---|---|---|
| | Local adverse events | Pain, sensitivity (tenderness to touch)<br>erythema, scab, induration, abscess<br>and axillary lymphadenopathy |
| Clinical | General adverse events | Fever, tachycardia,<br>hypo/hypertension, headache, fatigue,<br>myalgia, nausea/vomiting and<br>diarrhea |
| | Hematological | Blood count (hemoglobin, leukocytes, neutrophils, lymphocytes and platelets count) |
| Laboratory | Biochemical | Transaminases, bilirubin, cholesterol, creatine, ureic nitrogen, plasmatic electrolytes, coagulation test, creatine phosphokinase and urine analyses |

### **10.5.2.** Appropriateness of Measurements

The above safety measurements were conducted to identify clinical symptoms or laboratory parameters that were uniquely related to the administration of the experimental rBCG-N-hRSV vaccine. Unusual local systemic clinical reactions were documented, and laboratory evidence for renal, liver, hematologic disease adverse events were recorded.

### 10.5.3. Primary Efficacy/Immunogenicity Endpoints

NA

### 10.5.4. Primary Safety Endpoints

The primary safety endpoints of the study were the following:

- Evaluation of reactogenicity (Local and systemics AE)
- Evaluation of laboratory AE
- Serious AE (SAE)
- Evaluation of the presence of the BCG vaccine (wild-type and recombinant) in body fluids (blood, urine and saliva were cultured).

#### 10.5.5. Secondary Efficacy/Immunogenicity and Safety Endpoints

The secondary efficacy/immunogenicity and safety endpoints were the following:

- Evaluation of the humoral and cellular immune responses against *M. bovis* BCG.
- Evaluation of the humoral and cellular immune responses against hRSV.

### 10.5.6. Drug Concentration Measurements

NA

### **10.6.** Data Quality Assurance

### **10.6.1.** Data Collection and Management

For the clinical and laboratory data collection, a handwritten and electronic Case Report File (CRF) was used for each visit. In addition, the local BCG lesion sites were photographed to document the local reactogenicity responses (pictures of the vaccine area were taken).

To look for evidence of disseminated and/or persistent BCG infection vaccinated donors provided samples of blood, urine and saliva.

For the cellular immunogenicity assays 20 ml of venous blood were collected in heparinized tubes (BD Vacutainer, New Jersey, USA), obtained from volunteers at day 0, 14, 30, 60, 120 and 180 post-vaccination. The venous blood was purified by gradient centrifugation with Leukocyte Separation Medium (LSM, Corning, Virginia, USA) for 30 minutes at 20°C/300g. Cells were collected, washed twice with 1X PBS (Gibco, New York, USA), counted in a Neubauer chamber and then frozen with DMSO in liquid nitrogen. All samples were stored in a -150°C Ultrafreezer until the assays were performed.

For the humoral immunogenicity assays, 6 ml of venous blood were collected in non-heparinized tubes (BD Vacutainer, New Jersey, USA), acquired from volunteers at day 0, 14, 30, 60, 120 and 180 days post-vaccination. The venous blood was incubated vertically at room temperature for at least 30 minutes, then serum obtained by centrifugation for 15 minutes at room temperature in an Eppendorf centrifuge with a horizontal rotor at 1,500 g. 1.8 ml of serum were collected, aliquoted in 6 vials and frozen at -80°C (Glacier<sup>TM</sup> -86°C Ultra low Freezer) until the assays were performed.

Assays to detect disseminated/persistent infection with the BCG vaccines included PCR and conventional culture, the cellular immunogenicity assays were assessed by ELISPOT and flow cytometry and the humoral immunogenicity assays were evaluated using indirect ELISA assays. These results were reported on specific study report forms

### 10.6.1.1. Data Recording Methods

The Source Documents used for documenting the clinical data were the institutional clinical records at PUCC hospital and clinical evaluating unit and for the volunteers. In each study visit the anamnesis-clinical record/history for each subject, physical exam and all the study procedures as described above were collected on the CRF to properly inform the clinician about the individual health history.

For the laboratory data, an electronic report issued by the clinical laboratory at PUCC hospital was generated.

### 10.6.1.2. Subject Identifiers

Each sample was identified with the number of each subject (i.e. the samples from RSV01 were identified as RSV01)

### 10.6.2. Monitoring, Auditing, and Archiving

Once the healthy volunteers met the inclusion and exclusion criteria, the subjects received a single dose of the vaccine intradermally in the deltoid area. They were observed in the study clinic for the next 3 hours. Participants were evaluated at days 1, 2, 3, 7, 14, 30, 60, 120 and 180 after vaccination. Follow-up phone calls were performed at days 4, 21, 45, 90 and 150 after vaccination.

### 10.6.3. Database Lock

The staff of the clinical team entered information from each participant into an electronic CRF using a software called FMED (generated by the company "Brain Up"), which automatically organizes the data into a single coded excel file.

## 10.7. Statistical Methods Planned in the Protocol and Determination of Sample Size

### 10.7.1. Sample Size

A total of 42 healthy males between ages 18 and 50 years of age were screened, and 24 were enrolled and vaccinated with 8 participants in each cohort. Table III shows the number and age of participants that were screened and vaccinated.

Table III: Subjects receiving investigational product.

| Subject number | Age | Received vaccine number | Subject number | Age | Received vaccine number |
|---|---|---|---|---|---|
| RSV01 | 31 | CL01 | RSV22 | 20 | NA |
| RSV02 | 32 | CL02 | RSV23 | 25 | NA |
| RSV03 | 22 | CL03 | RSV24 | 22 | CL12 |
| RSV04 | 22 | NA | RSV25 | 44 | CL13 |
| RSV05 | 21 | CL04 | RSV26 | 25 | CL14 |
| RSV06 | 35 | NA | RSV27 | 22 | CL15 |
| RSV07 | 36 | CL05 | RSV28 | 25 | NA |
| RSV08 | 26 | NA | RSV29 | 19 | NA |
| RSV09 | 22 | NA | RSV30 | 24 | CL16 |
| RSV10 | 25 | CL06 | RSV31 | 33 | NA |
| RSV11 | 27 | NA | RSV32 | 21 | CL17 |
| RSV12 | 24 | NA | RSV33 | 21 | CL18 |
| RSV13 | 20 | CL07 | RSV34 | 21 | CL19 |
| RSV14 | 34 | CL08 | RSV35 | 20 | NA |
| RSV15 | 24 | NA | RSV36 | 25 | CL20 |
| RSV16 | 24 | CL09 | RSV37 | 29 | NA |
| RSV17 | 20 | CL10 | RSV38 | 19 | CL21 |
| RSV18 | 28 | CL11 | RSV39 | 27 | NA |
| RSV19 | 48 | NA | RSV40 | 21 | CL22 |
| RSV20 | 25 | NA | RSV41 | 21 | CL23 |
| RSV21 | 21 | NA | RSV42 | 20 | CL24 |

<sup>\*</sup>NA: non applicable; CL-number: refers to the vaccine code received

### 10.7.2. Statistical Analysis Plan

This was a phase I clinical trial to evaluate safety and was not statistically powered. For the clinical data obtained the Student's *t*-test was used. For immunogenicity assays, statistical significance was assessed using One-way ANOVA with a posteriori Tukey test or Two-way ANOVA test with a posteriori Tukey test.

### 11. STUDY SUBJECTS

### 11.1. Disposition of Subjects

Once inclusion criteria were met, volunteers were enrolled into three cohorts. Each cohort included 6 volunteers vaccinated with escalating doses of rBCG-N-hRSV (5x10<sup>3</sup> CFU; 5x10<sup>4</sup> CFU; 1x10<sup>5</sup> CFU) and 2 volunteers vaccinated with the standard BCG (BCG-WT) (full dose of 2x10<sup>5</sup> CFU). Figure 1 shows the clinical study flow diagram.



**Figure 1: Clinical study flow diagram.** The phase 1 study was a double blind dose ranging study. Each cohort included 6 volunteers vaccinated with escalating doses of rBCG-N-hRSV (5 x  $10^3$  CFU; 5 x  $10^4$  CFU; 1 x  $10^5$  CFU) and 2 volunteers vaccinated with the standard BCG (BCG-WT) (2 x  $10^5$  CFU). Furthermore, the DSMB evaluated safety data of each cohort after the first 30 days of follow up and decided if escalation could continue.

Table IV show the disposition of subjects according to the cohort in which they were (from all the subjects including the ones that were excluded from the study).

Table IV: Cohort by subject's number.

| Cohort | Subject number | Cohort | Subject number |
|--------|----------------|--------|----------------|
| | RSV01 | | RSV22 |
| | RSV02 | | RSV23 |
| | RSV03 | | RSV24 |
| | RSV04 | | RSV25 |
| | RSV05 | В | RSV26 |
| | RSV06 | | RSV27 |
| | RSV07 | | RSV28 |
| A | RSV08 | | RSV29 |
| | RSV09 | | RSV30 |
| | RSV10 | | RSV31 |
| | RSV11 | | RSV32 |
| | RSV12 | | RSV33 |
| | RSV13 | | RSV34 |
| | RSV14 | | RSV35 |
| | RSV15 | C | RSV36 |
| | RSV16 | C | RSV37 |
| | RSV17 | | RSV38 |
| D | RSV18 | | RSV39 |
| В | RSV19 | | RSV40 |
| | RSV20 | | RSV41 |
| | RSV21 | | RSV42 |

### 11.1.1. Demographic Data by Study Group

The Table V show the demographic data of subjects according to study group (from all subjects including the ones that were excluded from the study).

Table V: Demographic data by study group.

| Study group | Age range | Sex/Gender |
|-------------|-----------|------------|
| Cohort A | 20-36 | |
| Cohort B | 20-44 | Male |
| Cohort C | 19-25 | |

### 11.1.2. Summary of Prior and Concurrent Medical Conditions

NA

### 11.1.3. Study Visit Schedule

The Table VI show the study visit schedule for the participants.

Table VI. Study visit Schedule

| Name/number of<br>visit | Screening<br>Day -3<br>to -10 | Visit 1<br>Day 0 | Visit 2<br>Day 1<br>(+1) | Visit 3<br>Day 2<br>(+1) | Visita 4<br>Día 3<br>(+1) | Call<br>Day 4 | Visita 5<br>Day 7<br>(±2) | Visit 6<br>Day 14<br>(±3) | Call<br>Day 21 | Visit 7<br>Day 30<br>(±5) | Call<br>Day 45 | Visit 8<br>Day 60<br>(±7) | Call<br>Day 90 | Visit 9<br>Day 120<br>(±7) | Call<br>Day 150 | Visit<br>10<br>Day<br>180<br>(±7) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Description of the visit | Screening | Vaccinati<br>on | Follow up<br>Visit | Follow up<br>Visit | Follow up<br>Visit | Telephonic contact | Follow up<br>Visit | Follow up<br>Visit | Telephonic contact | Follow up<br>Visit | Telephonic contact | Follow up<br>Visit | Telephonic contact | Follow up<br>Visit | Telephonic contact | Final visit |
| Informed Consent | x | | | | | | | | | | | | | | | |
| Medical History | х | | | | | | | | | | | | | | | |
| Physical exam | х | х | x | х | х | | х | x | | х | | х | | х | | х |
| Vital Signs | x | X | × | x | X | | x | X | | x | | x | | X | | x |
| Verification of inclusion criteria | x | × | ~ | ~ | ~ | | ~ | | | ~ | | ^ | | ^ | | ~ |
| Designation of study # | х | | | | | | | | | | | | | | | |
| Eligibility tests | х | | | | | | | | | | | | | | | |
| Verification of Inclusion criteria | | х | | | | | | | | | | | | | | |
| Randomization | | X | | | | | | - | | | | | | | | |
| Samples for immunogenicity tests | | х | | | | | | х | | х | | х | | х | | Х |
| Vaccine<br>administration | | x | | | | | | 1 | | | | | | | | |
| Observation for 3 h | | х | | | | | | | | | | | | | | |
| Daily Chart deliver | | x | | | | | x | x | | x | | х | | x | | |
| Safety contact | | | | | | х | | | х | | х | | х | | x | |
| Daily chart revision | | | x | x | х | | х | х | | х | | x | | x | | х |
| Evaluation of papule | | | х | х | х | | X | х | | X | | X | | X | | х |
| Safety Tests | | | х | х | х | | х | х | | х | | х | | х | | х |
| Transmisibility tests | | | | | | | х | | | х | | | | | | х |
| AE, SAEs | | | | | | х | x | x | х | x | х | x | х | х | х | х |

### 11.1.4. Vital Signs Grading

The vital signs were graded from 1 to 4.

Table VII: Vital signs grading.

| Vital signs | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potential life risk (Grade 4) |
|---|---|---|---|---|
| Fever (°C) (oral or axillary) | 38.0-38.4 | 38.5-38.9 | 39.0-40.0 | >40.0 |
| Tachycardia – beats<br>per minute | 101-115 | 116-130 | >130 | Emergency visit or hospitalization due to arrhythmia |

| Bradycardia – beats<br>per minute | 50-54 | 45-49 | < 45 | Emergency visit or hospitalization due to bradyarrhythmia |
|---|---|---|---|---|
| Hypertension<br>(systolic) – mmHg | 141-150 | 151-155 | >155 | Emergency visit or<br>hospitalization due to<br>malignant<br>hypertension |
| Hypertension<br>(diastolic) - mmHg | 91-95 | 96-100 | >100 | Emergency visit or<br>hospitalization due to<br>malignant<br>hypertension |
| Hypotension<br>(systolic) – mmHg | 85-89 | 80-84 | < 80 | Emergency visit or hospitalization due to shock |
| Respiratory<br>frequency – breaths<br>per minute | 17-20 | 21-25 | >25 | Intubation |

### 11.2. Protocol Deviations

Table VIII shows the protocol deviations for each subject, all of which took place during the eligibility exams. The deviations were reported to the institutional ethics committee and to the Data and Safety Monitoring Board (DSMB).

The DSMB analyzed these deviations and requested additional information on the lymphocytic subpopulations. Upon review, the DSMB concluded that the protocol deviations did not have any impact on the safety of the subjects and recommended that the study continue.

Table VIII: Protocol deviation by each subject

| Subject | Deviation | Corrective action |
|---|---|---|
| RSV01 | Albumin at baseline (eligibility tests) out of the range indicated in amendment 2 (5.1 mg/dl, value indicated is 3.5-5.0) | All study personnel were trained to rigorously adhere |

| | I | 1 1 0 1 |
|---|---|---|
| RSV01 | Cholesterol at baseline (eligibility tests) out of the range indicated in amendment 2, 200 mg/dl (the amendment 2 indicated, by mistake, the normal value is <200, being ≤200 correct) | to the values of the laboratory |
| RSV01 | Missing values for CD16 or CD56/19 in the lymphocytic populations at baseline (eligibility tests) | The laboratory was trained to report these values of the study subjects |
| RSV02 | Missing values for CD16 or CD56/19 in the lymphocytic populations at baseline (eligibility tests) | stady subjects |
| RSV03 | Missing values for CD16 or CD56/19 in the lymphocytic populations at baseline (eligibility tests) | |
| RSV05 | Missing values for CD16 or CD56/19 in the lymphocytic populations at baseline (eligibility tests) | |
| RSV07 | Missing values for CD16 or CD56/19 in the lymphocytic populations at baseline (eligibility tests) | |
| RSV25 | From day 9, the subject did not register appropriately the measurements for erythema and induration, but all of these were less than 25 mm | The subject and study personnel were retrained to ensure these measurements were performed until day 30 |
| RSV27 | In Visit 6 (day 14 post-vaccination) the PT and PTT were not measured. | Study personnel were retrained on the correct tubes to be used for these measurements |
| RSV 36 | Visit 7, 1 day out of the window period | The subject was further educated as to the importance of following study procedures |

### 12. EFFICACY/IMMUNOGENICITY EVALUATION

### 12.1. Analysis Populations

The population analyzed were healthy male adults, between 18 and 50 years of age.

### 12.2. Demographics and Other Baseline Characteristics

The participants were healthy Chilean males 18 to 50 years old, who were vaccinated with BCG once or twice during their life, prior to study participation. The information was recording by an objective evaluation of the BCG vaccination scar or scars in each subject. It is not possible to determine which BCG strain the participant received previous to this study, because the Chilean Government obtain different vaccines from different sources (Statens Serum Institut or Serum Institute of India)

#### 12.2.1. Prior and Concurrent Medical Conditions

The subjects were healthy and tested negative for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG) and hepatitis C virus (HCV), and had no evidence of primary or secondary immunodeficiency.

#### 12.2.2. Prior and Concomitant Medications

The subjects had to meet the inclusion and exclusion criteria prior to enrolling in the trial. Prior to the study, the subjects were not allowed to use inhaled corticosteroids or immunosuppressors, had not received treatment for tuberculosis or other mycobacteria, had not used illegal drug substances and had not been administered immunoglobulins or blood-derived products.

### **12.3.** Measurements of Treatment Compliance

Since the treatment is an immunization with a single dose of either, control BCG vaccine provided by the Ministry of Health in Chile (Serum Institute of India, Bacillus Calmette Guerin Moscow strain 361- I) or rBCG-N-hRSV, no measurements of treatment compliance were required.

## 12.4. Efficacy/Immunogenicity Results and Tabulations of Individual Subject Data

### 12.4.1. Methodology and Primary Statistical Analysis of Efficacy/ Immunogenicity Data

The immune responses were measured as follows: Peripheral blood mononuclear cells (PBMC) and serum samples from twenty four subjects were collected on visits 1 (day 0), 6 (day 14), 7 (day 30) and 10 (day 180) post-vaccination and stored. The 24 subjects were divided in three groups of 8 according to the dose of rBCG-N-hRSV used: Cohort A (5x10³ CFU), cohort B (5x10⁴ CFU) and cohort C (1x10⁵ CFU). To evaluate the cellular response, the cells obtained from peripheral blood were thawed, counted and stimulated *in vitro* with PPD and N-RSV antigens to measure the antigen-specific immune response. Total cells that secreted IL-2 and/or IFN-γ were measured by ELISPOT and cellular subpopulations of CD4⁺/CD8⁺ producers of IL-2⁺ IFN-γ were measured by flow cytometry. To evaluate the humoral response, sera were thawed and incubated in pre-activated ELISA plates with PPD and N-RSV antigens. Afterwards, they were incubated

with human anti-IgG secondary antibody conjugated to horseradish peroxidase (HRP). The specific immunoglobulins against PPD and N-RSV were quantified using a standard curve with the humanized anti-F antibody (Palivizumab). The results were obtained based on the absorbance of the product generated by the anti-IgG HRP antibody and TMB substrate (3,3',5,5'-Tetramethylbenzidine) in a spectrophotometer.

All statistical analyses for the immunogenicity assays were performed using GraphPad Prism version 7.0 Software. Statistical significance was assessed using One-way ANOVA with a *posteriori* Tukey test, or two-way ANOVA test with a *posteriori* Tukey test.

### 12.4.1.1. Handling of Dropouts or Missing Data

Data for some time points for ELISPOT evaluation in cohort A was missing, as described in table V.

### 12.4.2. Tabulation of Individual Response Data

Table IX: Immunogenicity Individual Response

| | | IFN-y and IL-2 SFC/million cells against PPD | | | | | | | IFN-y and IL-2 SFC/million cells against hRSV N protein | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | BCG-W | VT 2x10 <sup>5</sup> | | | | | |
| | VRS01 | VRS 13 | VRS18 | VRS24 | VRS34 | VRS38 | VRS01 | VRS 13 | VRS18 | VRS24 | VRS34 | VRS38 |
| 0 dpi | 0 | 23.3 | 110 | 10 | 60 | 123.3 | 0 | 0 | 13.3 | 0 | 0 | 0 |
| 14 dpi | 23.3 | | 103.3 | 3.3 | 63.3 | 196.7 | 0 | * | * | 0 | 0 | 6.7 |
| 30 dpi | 120 | 73.3 | 140 | 3.3 | 86.7 | 120 | 10 | 3.3 | 0 | 0 | 0 | 3.3 |
| 60 dpi | 86.7 | 130 | 126.7 | 33.3 | 73.3 | 110 | 3.3 | 3.3 | 0 | 0 | 3.3 | 0 |
| 120 dpi | 70 | 96.7 | 256.7 | 46.7 | 6.7 | 113.3 | 10 | 0 | 6.7 | 0 | 0 | 10 |
| 180 dpi | 53.3 | 6.7 | 160 | 93.3 | 0 | 56.7 | 3.3 | 0 | 3.3 | 3.3 | 3.3 | 0 |
| | COHORT A | | | | | | | | | | | |
| | VRS02 | VRS03 | VRS05 | VRS07 | VRS10 | VRS14 | VRS02 | VRS03 | VRS05 | VRS07 | VRS10 | VRS14 |
| 0 dpi | * | 36.7 | 90 | 20 | 70 | 266.7 | * | 3.3 | 46.7 | 0 | 0 | 16.7 |
| 14 dpi | * | * | * | 36.7 | | 200 | * | * | * | 3.3 | * | 13.3 |
| 30 dpi | * | 150 | 33.3 | 110 | 263.3 | 126.7 | * | 0 | 16.7 | 3.3 | 0 | 6.7 |
| 60 dpi | 56.7 | 50 | 10 | 33.3 | 156.7 | 66.7 | 0 | 0 | 3.3 | 10 | 0 | 3.3 |
| 120 dpi | 6.7 | 146.7 | 40 | 83.3 | 83.3 | 143.3 | 0 | 10 | 20 | 0 | 0 | 0 |
| 180 dpi | 23.3 | 70 | 13.3 | 46.7 | 16.7 | 43.3 | 0 | 0 | 13.3 | 6.7 | 0 | 0 |
| | | | | | | СОНО | RT B | | | | | |
| | VRS16 | VRS27 | VRS17 | VRS25 | VRS26 | VRS30 | VRS16 | VRS27 | VRS17 | VRS25 | VRS26 | VRS30 |
| 0 dpi | 33.3 | 0 | 90 | 20 | 46.7 | 10 | 10 | 0 | 6.7 | 0 | 6.7 | 10 |
| 14 dpi | 106.7 | 253.3 | 236.7 | 13.3 | 63.3 | 46.7 | 6.7 | 0 | 3.3 | 0 | 0 | 3.3 |
| 30 dpi | 106.7 | 306.7 | 300 | 60 | 136.7 | 46.7 | 6.7 | 0 | 3.3 | 3.3 | 23.3 | 6.7 |
| 60 dpi | 180 | 413.3 | 216.7 | 146.7 | 106.7 | 20 | 6.7 | 16.7 | 3.3 | 3.3 | 10 | 3.3 |

| 120 dpi | 93.3 | 176.7 | 143.3 | 6.7 | 90 | 13.3 | 10 | 13.3 | 0 | 0 | 3.3 | 0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 180 dpi | 100 | 100 | 113.3 | 73.3 | 50 | 13.3 | 0 | 0 | 0 | 3.3 | 10 | 0 |
| | COHORT C | | | | | | | | | | | |
| | VRS32 | VRS33 | VRS36 | VRS40 | VRS41 | VRS42 | VRS32 | VRS33 | VRS36 | VRS40 | VRS41 | VRS42 |
| 0 dpi | 6.7 | 43.3 | 110 | 46.7 | 10 | 440 | 0 | 6.7 | 23.3 | 46.7 | 10 | 0 |
| 14 dpi | 66.7 | 276.7 | 180 | 153.3 | 26.7 | 543.3 | 0 | 0 | 56.7 | 46.7 | 10 | 6.7 |
| 30 dpi | 103.3 | 126.7 | 166.7 | 106.7 | 13.3 | 340 | 6.7 | 3.3 | 66.7 | 33.3 | 16.7 | 10 |
| 60 dpi | 50 | 46.7 | 20 | 70 | 16.7 | 223.3 | 3.3 | 3.3 | 3.3 | 46.7 | 6.7 | 3.3 |
| 120 dpi | 16.7 | 36.7 | 383.3 | 103.3 | 0 | 76.7 | 0 | 3.3 | 0 | 46.7 | 10 | 23.3 |
| 180 dpi | 36.7 | 73.3 | 280 | 63.3 | 0 | 116.7 | 6.7 | 13.3 | 3.3 | 36.7 | 13.3 | 23.3 |

<sup>\*</sup>Missing data

dpi: Days post-immunization.

### 12.4.3. Efficacy/Immunogenicity Conclusions

Cellular immunogenicity measurements showed that 14 days after vaccination all volunteers increased cellular production of IFN-γ and IL-2 upon *in vitro* stimulation with PPD antigen by ELISPOT (Figure 2). The cellular response against the RSV N protein was increased 30 days after vaccination, indicating the induction of a specific immune response against antigens included in the vaccine.



Figure 2: Measurement of the specific cellular response by ELISPOT against the PPD antigens (in black) and N protein (in white) of the human respiratory syncytial virus. The results are expressed as the fold change (log2) with respect to visit 1 (day 0) for IFN-g and IL-2 secretory cells at times 14, 30 and 180 days after vaccination for the three doses of rBCG-N-hRSV (5x10<sup>3</sup> CFU, 5x10<sup>4</sup> CFU, 1x10<sup>5</sup> CFU) and for BCG-WT (2x10<sup>5</sup> CFU).

Furthermore, the amount of specific IgG response against PPD and N in the serum increased 60 days post-vaccination (Figure 3). In summary, rBCG-N-hRSV showed a good safety profile in healthy adults and induced specific cellular and humoral immune responses.



Figure 3: Measurement of the specific humoral immune response by indirect ELISA assay against the N protein (in white) and PPD antigens (in black) of the human respiratory syncytial virus. The result is expressed in fold change (log10) with respect to visit 1 (day 0) in the detection of specific IgG at times 60, 120 and 180 days after vaccination for the three doses of rBCG- N-hRSV (5x10<sup>3</sup> CFU, 5x10<sup>4</sup> CFU, 1x10<sup>5</sup> CFU) and for BCG-WT (2x10<sup>5</sup> CFU).

### 13. SAFETY EVALUATION

### 13.1. Extent of Exposure

From the total of 24 participants, there were 524 adverse events.

### 13.2. Adverse Events (AEs)

### 13.2.1. Brief Summary of Adverse Events

Overall, 524 adverse events were registered for the 24 participants: 244 local adverse events (46.6%), 157 general adverse events (30.0%) and 123 laboratory adverse events (23.5%). Importantly, no participants were discontinued due to an AE. The most frequent local solicited adverse events were abscess, scabbing and tenderness at the BCG injection sites, occurring in all participants. The most common solicited adverse events were headache, fatigue, diarrhea and myalgia. As for the laboratory adverse events (as defined by a significant deviation from normal ranges for laboratory tests), 56.9% were classified as not related to vaccine and 43.1% as possibly

related to vaccine because no definitive etiology was found. The most common laboratory adverse event was decreased hemoglobin (see Table XII).

### 13.2.2. Display of Adverse Events

A severe laboratory adverse event (SAE) G4 was presented during the study of cohort C. This event relates to subject RSV34 that on day 14 (December 06 2017), while being asymptomatic, presented a rise in CPK values (20.488 U/L). The subject did intense exercise at the gym on December 03th, 2017 for 1.5 hour, resulting in fatigue at the end of his exercise and myalgias for the next few days. This was accompanied by a grade 3 rise in SGOT (276 U/L). On December 11, 2017 the subject was found to have a CPK of 3.827 U/L and SGOT of 186 U/L. On visit day 30 (December 21, 2017), both values had normalized (CPK 134 U/L and SGOT 18 U/L). The SAE from this study are shown in Table VI. This event was considered to be unrelated to the study vaccine, by the investigator as well as the sponsor's security delegate, Dr. Fernando Altermatt. The SAE was reported to the institutional ethics committee (CEC-MedCUC) and to the sponsor's security delegate, who notified the Institute for Public Health of Chile (Instituto de Salud Pública de Chile).

Table X: SAE from the three cohorts, at January 8 2018, completion of day 30 post vaccination Cohort C

| Cohort | SAEs | SAE type | Relation with the vaccine | Final Disposition |
|---|---|---|---|---|
| A | 0 | None | None | None |
| В | 0 | None | None | None |
| С | 1 | Grade 4 rise of CPK | Not related | Resolved |
| Total | 1 | Laboratory abnormality | Not related | All resolved |

Clinical adverse events (CAE) were presented at day 30 and are shown in Table XI. A rise of local AEs was observed in cohort B as compared to cohort A, and in cohort C as compared to cohort B, being significant only for the difference between cohort A and C (p=0.04 test U Mann Whitney). As for the total AEs, there were no significant differences between cohorts.

Table XI: Clinical Adverse Events Cohorts A, B and C, at day 30 at January 8 2018, completion of day 30 post vaccination Cohort C

| Event | Cohort A | Cohort B | Cohort C | Total |
|--------------------------|----------|----------|----------|-------|
| Solicited local AE | 51 | 70 | 83 | 204 |
| Non solicited local AE | 8 | 6 | 8 | 22 |
| Subtotal local AE | 59 | 76 | 91 | 226 |
| Solicited general AE | 21 | 19 | 28 | 68 |
| Non solicited general AE | 15 | 2 | 11 | 28 |
| Subtotal general AE | 36 | 21 | 39 | 96 |
| Total AE | 95 | 97 | 130 | 322 |

Clinical adverse events (CAE) identified by January 8<sup>th</sup> 2018, which is completion of day 30 post vaccination of Cohort C, are shown in table XII.

Table XII: Clinical adverse events for Cohorts A, B and C at the day of the inform (January 8th 2018), completion of day 30 post vaccination Cohort C.

| | Cohort A | Cohort B | Cohort C | Total |
|--------------------------|-------------|----------|----------|-------|
| Event | Day 150-180 | Day 60 | Day 30 | |
| Solicited local AE | 57 | 72 | 83 | 212 |
| Non solicited local AE | 11 | 6 | 8 | 25 |
| Subtotal local AE | 68 | 78 | 91 | 237 |
| Solicited general AE | 22 | 20 | 28 | 70 |
| Non solicited general AE | 38 | 6 | 11 | 55 |
| Subtotal general AE | 60 | 26 | 39 | 125 |
| Total AE | 128 | 104 | 130 | 258 |
#### 13.2.2.1. Solicited AEs

Clinical solicited adverse events were followed through day 30 post-vaccination. Local solicited AE included pain, sensitivity, erythema, scab, induration, abscess and axillary lymphadenopathy. General solicited AE included fever, tachycardia, hypo/hypertension, headache, fatigue, myalgia, nausea/vomiting and diarrhea. Local solicited grade 3 AE were identified only in cohort C, and included 2 grade 3 reactions (1 pain and 1 sensitivity) at the vaccination site. Both events were resolved.

Table XIII: Solicited general adverse events grade 3. The number of low, moderate and severe events per cohort and per type of event is shown in the Table. The vital risk events are not included in this Table.

| Event | Cohort A | | | | Cohort B | | | Cohort C | |
|---|---|---|---|---|---|---|---|---|---|
| | low | moderate | severe | low | moderate | severe | low | moderate | severe |
| Headache | 3 | 0 | 0 | 0 | 0 | 0 | 9 | 2 | 0 |
| Fatigue | 2 | 0 | 0 | 3 | 0 | 0 | 4 | 1 | 0 |
| Nausea/vomiting | 7 | 2 | 0 | 5 | 1 | 0 | 4 | 0 | 0 |
| Diarrhea | 6 | 0 | 0 | 4 | 0 | 0 | 5 | 0 | 0 |
| Myalgia | 1 | 0 | 0 | 6 | 0 | 0 | 3 | 0 | 0 |
| Fever | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| TOTAL | 19 | 2 | 0 | 18 | 1 | 0 | 25 | 3 | 0 |

#### 13.2.2.2. Unsolicited AEs

Clinical unsolicited adverse events were recorded through day 30. The episodes of high blood pressure and tachycardia did not occur in the period immediately after vaccination, but at the beginning of subsequent visits. In Cohort A, these measurements were not repeated by the staff. In Cohort B, these measurements were repeated and the values were repeatedly high.

Table XIV: Number of Non-Solicited Clinical Adverse events.

| Event | Cohorts A (5x10^3) | Cohorts A (5x10^4) | Cohorts A (1x10^5) | Control BCG<br>WT<br>(2x10^5) | TOTAL |
|---|---|---|---|---|---|
| Viral upper respiratory infection | 4 | 4 | 7 | 3 | 18 |
| Headache | 1 | 2 | 0 | 14 | 17 |
| Other events respiratory tract | 7 | 0 | 3 | 1 | 11 |
| Diarrhea/gastroenteritis | 1 | 0 | 4 | 0 | 5 |
| Toothache | 3 | 0 | 0 | 0 | 3 |
| Ecchymosis injection site | 1 | 0 | 1 | 0 | 2 |
| Bruise on hand | 1 | 0 | 1 | 0 | 2 |
| Contusion of hand/wrist | 0 | 0 | 1 | 1 | 2 |
| Cellulitis tight | 0 | 1 | 0 | 1 | 2 |
| Muscular contraction back | 0 | 1 | 0 | 1 | 2 |
| Abdominal pain | 0 | 0 | 0 | 1 | 1 |
| Arterial hypertension | 0 | 0 | 1 | 0 | 1 |
| Foot injury due to beat | 0 | 0 | 0 | 1 | 1 |
| General malaise | 0 | 0 | 1 | 0 | 1 |
| Urethritis | 0 | 0 | 1 | 0 | 1 |
| Urticaria | 0 | 0 | 1 | 0 | 1 |
| Sclap ache | 0 | 0 | 1 | 0 | 1 |
| Retro ocular ache | 1 | 0 | 0 | 0 | 1 |

| Fever | 1 | 0 | 0 | 0 | 1 |
|-----------------------------|----|---|----|----|----|
| Epistaxis | 0 | 0 | 0 | 1 | 1 |
| Nausea | 0 | 0 | 1 | 0 | 1 |
| Ansiety | 0 | 0 | 1 | 0 | 1 |
| Insomnia | 0 | 0 | 1 | 0 | 1 |
| Myalgia | 0 | 0 | 1 | 0 | 1 |
| Leg pain | 0 | 0 | 0 | 1 | 1 |
| Scratch in vaccination site | 1 | 0 | 0 | 0 | 1 |
| TOTAL | 20 | 6 | 25 | 25 | 76 |

#### 13.2.3. Analysis of Adverse Events

There were more solicited local grade 2 and grade 3 clinical AEs (severe and moderate) in Cohort B and C compared to Cohort A (p = 0.012 and p = 0.001, respectively), but there were no significant differences between Cohort B and Cohort C (p = 0.362): Cohort A (3/51 = 5.9%), Cohort B (16/70 = 22.9%), Cohort C (25/83 = 30.1%). There were no significant differences in the solicited general AEs between cohorts, and therefore there was no association with increasing doses of the study vaccine. There were no significant differences in unsolicited clinical AEs between the groups.

The listing of local adverse events by subjects, can be seen in Table XXV (annex).

The listing of general adverse events by subjects, can be seen in Table XXVI (annex).

# 13.3. Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

# 13.3.1. Listing of Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

No deaths occurred in any study subject during the trial observation period.

Two Serious Adverse Events were registered during the study.

#### 13.3.1.1. Deaths

No deaths were occurred in this study.

#### 13.3.1.2. Serious Adverse Events

The listing of serious adverse events, can be seen in Table XV.

Table XV: Serious adverse events.

| Subject | Age | Diagnosis | Vaccination<br>Date | Start Date (days post-vaccination) | Resolution Date (days post-vaccination) | Severity<br>Criterion | Vaccine | Assigned<br>Cause | Related to vaccination |
|---|---|---|---|---|---|---|---|---|---|
| RSV34 | 22 | Increase in CPK | 21-11-17 | 17 | 31 | Lab AE G4 | Control | Intense<br>exercises<br>the day<br>before | No |
| RSV42 | 20 | Precordial pain<br>secondary to<br>Supraventricular<br>Tachycardia | 04-12-17 | 51 | 53 | Hospitalization | 5x10 <sup>5</sup> | Previous<br>pre-<br>excitation<br>syndrome | No |

#### 13.3.1.3. Other Significant Adverse Events

NA

## 13.3.2. Narratives of Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

There were no deaths.

RSV34:

One SAE laboratory grade 4 AE occurred in subject RSV34 enrolled in cohort C, who was vaccinated on day November 21<sup>st</sup>, 2017 and on day 14 (December 06<sup>th</sup>, 2017 17 days after vaccination) presented to the clinic and was found to have an asymptomatic grade 4 increase in CPK (20,488 U/L). The subject had engaged in intense exercise at a gym on December 03, 2017 for 1.5 hours, and experienced marked fatigue at the end of the exercise and myalgia for the next few days. This was associated with a grade 3 increase in SGOT (276 U/L). At follow up on

December 11, 2017, the subject was found to have decreased levels of CPK (3,827 U/L) and SGOT (186 U/L). At his next scheduled visit on day 30 post-vaccination (December 21, 2017) both values had normalized (CPK of 134 U/L and SGOT of 18 U/L). The events were considered not to be related to the study vaccine by both, the investigator and the security delegate sponsor, Dr. Fernando Altermatt. The SAE was reported to the institutional ethic committee (CEC-MedUC) and the security delegate sponsor notified the Instituto de Salud Pública de Chile (ISP). The event was not related to the vaccination.

#### **RSV42**:

A second subject was hospitalized on January 25<sup>th</sup>, 2018 (51 days post vaccination) when he presented precordial pain beginning the night before. At the hospital, his EKG was essentially normal (only abnormality was a delta wave compatible with pre-excitation, which was a previous condition identified in the patient). However, he was found to have elevated cardiac enzymes. Echocardiogram findings were normal. The physicians determined that the precordial pain was most likely secondary to a supra-ventricular tachycardia due to a pre-excitation pathway that had been diagnosed when the subject was an infant. The final diagnosis for this SAE was pre-cordial pain secondary to a supra-ventricular tachycardia due to a pre-existing pre-excitation syndrome. The event was resolved the day of his medical release (January 26, 2018, day 53 post-vaccination). The event was not related to the vaccination.

# 13.3.3. Analysis and Discussion of Deaths, Other Serious Adverse Events, and Other Significant Adverse Events

According to the narrative, the Serious Adverse Events detected were not related to immunization. No deaths were reported in this study.

## 13.4. Clinical Laboratory Evaluation

#### 13.4.1. Individual Laboratory Measurements and Abnormal Laboratory Values

Laboratory adverse events (LAE) are presented in table XVI. No significant differences were observed comparing the 3 cohorts.

Table XVI: Laboratory adverse events from cohort A, B and C at day January 8<sup>th</sup>, 2018( 30 days after Cohort C vaccination)

| | Coh | ort A | Coh | ort B | Col | nort C |
|---|---|---|---|---|---|---|
| Event | Total | Grade 1/2/3 | Total | Grade 1/2/3 | Total | Grade 1/2/3 |
| Decrease of Hb | 7* | 5/1/1 | 5** | 5/0/0 | 8 | 7/1/0 |
| Increase in CPK | 6 | 3/2/1 | 2 | 2/0/0 | 4 | 2/2/0 |
| Leukopenia | 5# | 5/0/0 | 1 | 1/0/0 | 0 | NA |
| Increase in cholesterol | 2 | 2/0/0 | 1 | 1/0/0 | 0 | NA |
| Proteinuria <sup>S</sup> | 2 | 0/2/0 | 1 | 1/0/0 | 1 | 1/0/0 |
| Leukocytosis | 1 | 1/0/0 | 0 | NA | 0 | NA |
| Neutropenia | 1 | 0/1/0 | 0 | NA | 0 | NA |
| Increased SGOT or SGPT | 1 | 1/0/0 | 1 | 1/0/0 | 1 | 0/0/1 |
| Hypoproteinemia | 1 | 1/0/0 | 0 | NA | 0 | NA |
| Hyperglycemia <sup>&amp;</sup> | 1 | 1/0/0 | 0 | NA | 0 | NA |
| Hypophosphatemia | 1 | 1/0/0 | 1 | 1/0/0 | 1 | 1/0/0 |
| Increase in prothrombin | 1 | 1/0/0 | 0 | NA | 0 | NA |
| Pyuria | 0 | NA | 1 | 1/0/0 | 2 | 1/1/0 |
| Eosinophilia | 0 | NA | 1 | 1/0/0 | 1 | 1/0/0 |
| Hematuria | 0 | NA | 0 | NA | 1 | 0/1/0 |
| Increased LDH | 0 | NA | 0 | NA | 1 | 1/0/0 |
| Hypokalemia | 0 | NA | 0 | NA | 1 | 1/0/0 |
| Increase alkaline phosphatases | 0 | NA | 0 | NA | 1 | 1/0/0 |
| Total | 29 | 22/5/2 | 14 | 14/0/0 | 22 | 16/5/1 |

<sup>\*7</sup> episodes in 6 subjects, \*\*5 episodes in 4 subjects. Two recovered and presented again.

There was no relation of frequency and intensity of some laboratory AE with the type of vaccine received.

<sup>#5</sup> episodes in 4 subjects, one recovered and presented again.

<sup>§</sup>Proteinuria +- is considered mild and +, moderate

<sup>&</sup>amp;Patient was not fasting

#### 13.4.2. Evaluation of Each Laboratory Parameter

Hematological and biochemical parameters were measured at days 7, 14, 30, 60, 120 and 180 post-vaccination.

#### 13.4.2.1. Laboratory Values over Time

All grade 3 events reported decreased over time.

#### 13.4.2.2. Individual Subject Changes

Subject RSV01 presented 3 grade 3 events and only 2 of them returned to normal values. Subject RSV14 presented 1 grade 3 event and at day 30 was back to normal. Subject RSV25 presented 1 grade 3 events and at day 60 it continued as a grade 3. It normalized at visit 10 (day 180 post vaccination). Finally, subject RSV34 presented 2 events which at day 30 were back to normal.

Table XVII: Grade 3 laboratory adverse events and follow-up

| N | Cohort | Event<br>(Subject) | Association<br>with the<br>vaccine | Visit<br>when<br>event<br>presented | Evolution over time | Clinical<br>Manifestation | Observations |
|---|---|---|---|---|---|---|---|
| 1 | A | Hb decreased (RSV01) | Likely. Alternative cause: blood samples | V5 (Day 7) | Basal: 17.4 Day 07: 15.9 (G1) Day 14: 15.1 (G3) Day 30: 15.2 (G3) Day 60: 16.7 (G1) | None | Initial Hb was above the upper limit (17.4) because of potential dehydration at enrollment. The participant did not have anemia. |
| 2 | A | CPK increased (RSV14) | Likely. Alternative cause: exercise in | V5 (Day 7) | Day 7: 972 (G3) Day 14: 168 (N) Day 30: 126 (N) | None | Limit values established by PUCC were twice those established by the USA and France. Taking |

| | | | previous<br>days | | | | this information into consideration, the AE corresponds to Grade 2. |
|---|---|---|---|---|---|---|---|
| 3 | A | Hematuria<br>(RSV01) | Likely. Alternative cause: micro lithiasis | V8 (Day 60) | Day 60: 170 GR (G3) Day 62: 14 GR (G1) Day 120: 4 GR (N) | None | Family history of lithiasis. Culture negative. |
| 4 | A | Hypernatremia | Likely. Alternative cause: dehydration by fasting | V9 (Day<br>120) | Day 60: 150<br>mEq/L (G3)<br>Day 62: 143<br>mEq/L (N) | None | Normal repeated fasting |
| 5 | В | Hypophosphatemia<br>(RSV25) | Likely. Alternative cause: Low ingestion of phosphorus | V8 (Day 60) | Day 60: 1.8 mEq/L (G3) | None | At day 7 shows<br>Grade 1,<br>normalized at day<br>14. |
| 6 | С | CPK increased (RSV34) | Unrelated. Alternative cause: extreme exercise | V6 (Day 14) | Day 14:20.488 U/L<br>(G4)<br>Day 19: 3.827 U/L<br>(G3)<br>Day 30: 134 U/L<br>(N) | None | Normal at day 30 (V7) |
| 7 | С | SGTO increased (RSV34) | Unrelated. Alternative cause: exercise in previous days | V6 (Day 14) | Day 14: 276 U/L (G3) Day 19: 186 U/L (G2) Day 30: 18 U/L (N) | None | Normal at day 30 (V7) |

#### 13.4.2.3. Displays of Laboratory Results

#### 13.4.2.4. Chemistry Results

The biochemistry results from the 3 laboratory Cohorts, can be seen in Table XVIII.

Table XVIII: Biochemistry results from all laboratory cohorts. The total number of non-solicited clinical adverse events is shown per cohort ("Total" column). Also, the number of subjects that were categorized under a specific grade (1-low/2-moderate/3-severe) is shown in the Grades column.

| Event | Cohort A | | Cohort B | | Cohort C | |
|---|---|---|---|---|---|---|
| | Total | Grades | Total | Grades | Total | Grades 1/2/3 |
| Hb decreased | 7* | 5/1/1 | 6** | 6/0/0 | 8 | 7/1/0 |
| CPK increased | 6 | 3/2/1 | 2 | 2/0/0 | 4 | 2/2/0 |
| Alkaline phosphatases | 0 | NA | 0 | NA | 1 | 1/0/0 |
| TOTAL | 13 | 8/3/2 | 8 | 8/0/0 | 13 | 10/3/0 |

<sup>\*7</sup> episodes in 6 subjects, one recovered and presented again

#### 13.4.2.5. Hematology Results

The hematology results from the 3 laboratory Cohorts, can be seen in Table XIX.

Table XIX: Hematology results from all laboratory cohorts. The total number of non-solicited clinical adverse events is shown per cohort ("Total" column). Also, the number of subjects that were categorized under a specific grade (1-low/2-moderate/3-severe) is shown in the Grades column.

| Event | Cohort A | | Cohort B | | Cohort C | |
|---|---|---|---|---|---|---|
| | Total Grades | | Total | Grades | Total | Grades 1/2/3 |
| | | 1/2/3 | | 1/2/3 | | |
| Leukopenia | 5# | 5/0/0 | 1 | 1/0/0 | 0 | NA |
| Cholesterol increased | 2 | 2/0/0 | 1 | 1/0/0 | 0 | NA |

<sup>\*\*6</sup> episodes in 5 subjects, one recovered and presented again.

| Leukocytosis | 1 | 1/0/0 | 0 | NA | 0 | NA |
|----------------------------|----|--------|---|-------|---|-------|
| Neutropenia | 1 | 0/1/0 | 0 | NA | 0 | NA |
| SGOT or SGPT increased | 1 | 1/0/0 | 1 | 1/0/0 | 1 | 0/0/1 |
| Hypoproteinemia | 1 | 1/0/0 | 0 | NA | 0 | NA |
| Hyperglycemia & | 1 | 1/0/0 | 0 | NA | 0 | NA |
| Hypophosphatemia | 1 | 1/0/0 | 1 | 1/0/0 | 1 | 1/0/0 |
| Prothrombin time increased | 1 | 1/0/0 | 0 | NA | 0 | NA |
| Leucocituria | 0 | NA | 1 | 1/0/0 | 2 | 1/1/0 |
| Eosinophilia | 0 | NA | 1 | 1/0/0 | 1 | 1/0/0 |
| LDH increase | 0 | NA | 0 | NA | 1 | 1/0/0 |
| Hypokalemia | 0 | NA | 0 | NA | 1 | 1/0/0 |
| TOTAL | 14 | 13/1/0 | 6 | 6/0/0 | 7 | 5/1/1 |

<sup># 5</sup> episodes in 4 subjects, one recovered and presented again

The hematology results from the 3 clinical Cohorts, can be seen in Table XX.

Table XX: Hematology results from all 3 clinical cohorts. The total number of non-solicited clinical adverse events is shown per cohort ("Total" column). Also, the number of subjects that were categorized under a specific grade (1-low/2-moderate) is shown in the Grades column.

| Event | Cohort A | | Cohort B | | Cohort C | |
|---|---|---|---|---|---|---|
| | Total | Grades | Total | Grades | Total | Grades |
| Viral upper respiratory infection* | 5 | 5/0 | 1 | 1/0 | 2 | 2/0 |
| Other events respiratory system and ORL | 3 | 0/3 | 0 | NA | 1 | 1/0 |
| Lipothymia due to blood sampling | 1 | 0/1 | 0 | NA | 0 | NA |

| TOTAL | 9 | 5/4 | 1 | 1/0 | 3 | 3/0 |
|-------|---|-----|---|-----|---|-----|
|-------|---|-----|---|-----|---|-----|

#### 13.4.2.6. Urinalysis Results

The urinalysis results from the 3 laboratory Cohorts, can be seen in Table XXI.

Table XXI: Urinalysis results from all laboratory cohorts. The total number of non-solicited clinical adverse events is shown per cohort ("Total" column). Also, the number of subjects that were categorized under a specific grade (1-low/2-moderate/3-severe) is shown in the Grades column.

| Event | Coho | rt A | Cohort B | | Cohort C | |
|---|---|---|---|---|---|---|
| | Total | Grades | Total | Grades | Total | Grades 1/2/3 |
| Proteinuria <sup>§</sup> | 2 | 0/2/0 | 1 | 1/0/0 | 1 | 1/0/0 |
| Hematuria | 0 | NA | 0 | NA | 1 | 0/1/0 |
| TOTAL | 2 | 0/2/0 | 1 | 1/0/0 | 2 | 1/1/0 |

The urinalysis results from the 3 clinical Cohorts, can be seen in Table XXII.

Table XXII: Urinalysis results from all clinical cohorts. The total number of non-solicited clinical adverse events is shown per cohort ("Total" column). Also, the number of subjects that were categorized under a specific grade (1-low/2-moderate) is shown in the Grades column.

| Event | Cohe | ort A | Coh | ort B | Cohort C | |
|------------|--------------|-------|-------|--------|----------|--------|
| | Total Grades | | Total | Grades | Total | Grades |
| Urethritis | 0 | NA | 0 | NA | 1 | 1/0 |
| TOTAL | 0 | 0 NA | | NA | 1 | 1/0 |

# 13.5. Vital Signs, Physical Exam Findings, and Other Observations Related to Safety

#### 13.5.1. Vital Signs Grading

The vital signs from the 3 clinical Cohorts, can be seen in Table XXIII.

Table XXIII: Vital signs from all clinical cohorts. The total number of non-solicited clinical adverse events is shown per cohort ("Total" column). Also, the number of subjects that were categorized under a specific grade (1-low/2-moderate) is shown in the Grades column.

| Event | Coh | ort A | Coh | ort B | Cohort C | |
|---|---|---|---|---|---|---|
| | Total | Grades | Total | Grades | Total | Grades |
| Arterial hypertension | 2 | 2/0 | 1 | 1/0 | 0 | NA |
| Tachycardia | 1 | 1/0 | 0 | NA | 0 | NA |
| Systolic hypotension | 0 | NA | 0 | NA | 2 | 1/1 |
| TOTAL | 3 | 3/0 | 1 | 1/0 | 2 | 1/1 |

#### 13.5.2. Abnormal Vital Signs

The abnormal vital signs can be seen in table XXIV.

Table XXIV: Abnormal vital signs.

| Subject<br>N° | Cohort | Vaccine<br>Type* | Vaccine<br>Dose | AE<br>N°*<br>** | Diagnosis | AD<br>Type<br>*** | Vaccination<br>day | AE<br>Starts (day post<br>vaccination) | AE<br>Ends(day post<br>vaccination) |
|---|---|---|---|---|---|---|---|---|---|
| RSV03 | Cohort A | 1 | $5x10^{3}$ | 22 | Tachycardia | 3 | 1 | 1 | 1 |
| RSV05 | Cohort A | 1 | $5x10^{3}$ | 2 | Hypertension | 3 | 2 | 2 | 2 |
| RSV07 | Cohort A | 1 | $5x10^{3}$ | 6 | Hypotension | 3 | 7 | 7 | 7 |
| RSV07 | Cohort A | 1 | $5x10^{3}$ | 12 | Tachycardia | 3 | 2 | 2 | 2 |
| RSV14 | Cohort A | 1 | $5x10^{3}$ | 12 | Hypertension | 3 | 2 | 2 | 2 |
| RSV30 | Cohort B | 1 | 5x 10 <sup>4</sup> | 5 | Hypertension | 3 | 2 | 2 | 2 |
| RSv38 | Cohort C | 2 | 5x 10 <sup>5</sup> | 1 | Hypotension | 3 | 0 | 0 | 0 |
| RSV42 | Cohort C | 1 | 5x 10 <sup>5</sup> | 9 | Hypotension | 3 | 1 | 1 | 1 |

<sup>\*</sup> rBCG-N-hRSV (1) or WT-BCG (2).

<sup>\*\*</sup>AE number indicates the relative total AE numbers registered up to the point of that AE.

<sup>\*\*\*</sup> local solicited AE (1), local non-solicited AE (2), general solicited AE (3), general non-solicited AE (4), laboratory registered AE (5).

#### 13.6. Concomitant Medications

The use of concomitant medications was recorded. The concomitant medications used were associated with general adverse events (eg-upper respiratory infections) and general discomfort. No subject used any forbidden medications (corticosteroids, other live attenuated vaccines) throughout the protocol period.

### 13.7. Pregnancies (if applicable)

NA

## 13.8. Safety Conclusions

Clinical results indicated that both vaccines, rBCG-N-hRSV and BCG-WT, were safe and well tolerated. A higher reactogenicity in terms of abscess and scab formation at the vaccination sites was noted with dose escalation of the vaccine study, but none of these reactions were unexpected in the context of normal reactogenicity related to licensed intradermal BCG vaccines.

#### 14. DISCUSSIONS AND OVERALL CONCLUSION

The rBCG-N-hRSV vaccine has shown to be safe, well tolerated and immunogenic in healthy male adult volunteers. In terms of safety and tolerability, no related SAE were reported through the 180 days of follow-up post-vaccination. A higher reactogenicity was observed with the dose escalation of the vaccine study in terms of time of appearance and severity of abscess and scabbing. Other local events were not increased in association with dose escalations of the study vaccine.

In terms of immunogenicity, rBCG-N-hRSV elicited antigen-specific IgG and cellular immune responses against PPD and N-hRSV. Therefore, the rBCG-N-hRSV is a promising vaccine to prevent hRSV infection/disease as well as tuberculosis infection/disease in children and the elderly.

HRSV may cause severe cases of pneumonia and bronchiolitis in young children and the elderly (2). Unfortunately, the only licensed treatment to date for use in preventing severe hRSV disease is the monoclonal antibody Palivizumab, mainly indicated for high-risk infants (4). However, such treatment is costly and requires repeated doses to be effective (19). Further, although high numbers of prototype vaccines against hRSV infection are under development, few of them are on clinical trials (10). In the current study, we present the results of a Phase I clinical trial of a recombinant BCG that expresses the nucleoprotein of hRSV. BCG is a safe and immunogenic vaccine, being a suitable vector for hRSV vaccine (12, 13). Because our vaccine was designed using BCG as the vector, as well as to provide Th1 cell-inducing adjuvant properties, we evaluated the cellular immune responses of participants against mycobacterial PPD antigens. As shown in the cellular immunogenicity assays (Figures 2 to 4), before vaccination all participants displayed a modest frequency of cells that secreted IFN-γ and IL-2 in response to PPD stimulation. These baseline modest levels of immune response were likely due to the fact that all enrolled participants had been vaccinated in childhood with BCG. Therefore, we expected specific "recall" immune responses after in vitro cell stimulation with PPD (20). Once participants were vaccinated with the study vaccines (independently of the vaccine used), all demonstrated a sustained increase in IFN-y and IL-2 secretion, starting from 14th day post-vaccination and persisting at least until day 30 post-vaccination. We also found that the number of Spot Forming Cells by ELISpot, and the frequency by flow cytometry of CD4+ and CD8+ T cells secreting IFN-γ, IL-2 and TNF-α after PPD stimulation, increased as higher doses of the rBCG-N-hRSV vaccine were tested. These results indicate that the rBCG-N-hRSV vaccine can induce relevant antigen-specific T cell responses protective against TB, and suggest that these TB-specific responses are dose-dependent.

In contrast to the conventional BCG vaccine, this phase I study was the first time that the rBCG-N-hRSV was tested in healthy volunteers, and hRSV-specific immune responses were measured to determine the cellular and humoral immune responses directed against the N-hRSV protein. Prior to vaccination, we measured the baseline immune response to N protein and found that cells from all participants responded to N protein in vitro by secreting IFN-y, IL-2 and/or TNFα (Figures 3, 4, and Suppl. Figure 1). These baseline N-RSV-specific responses are likely due to previous hRSV exposures (3). Similarly, increased anti-F IgG antibody responses were found in all subjects enrolled into Cohort A, also suggesting that those subjects had been previously exposed to hRSV. It is known that after hRSV infection, cellular and humoral immune responses can be increased against hRSV antigens, such as the N protein (21). However, these immune responses appear to be ineffective, as recurrent infections can occur (22). We previously described that low single doses of BCG-N-hRSV vaccine (3x10<sup>5</sup> CFUs) were enough to induce Th1 immune responses in mice that protected animals against hRSV challenge (15). This antiviral immune response was characterized by the secretion of high levels of IFN-y and IL-17 from T cells after in vitro stimulation with hRSV antigens. In accordance with preclinical data, we found that all participants given BCG-N-hRSV vaccines increased the numbers of Spot Forming Cells and the frequencies of CD4<sup>+</sup> and CD8<sup>+</sup> T cells producing IFN-γ after hRSV nucleoprotein antigen in vitro stimulation. These levels increased from 14th day post vaccination and remained high at least until day 60, and in some cases even until day 180 post-vaccination. As seen with PPD measurements, the hRSV-specific immune responses increased with dose escalation. Polyfunctional T cell responses (producing combinations of both IFN-γ and IL-2) were more pronounced at day 30 postvaccination.

All available data to date suggest that protective hRSV immune responses must include strong CD4+ Th1 responses, and these Th1 responses are not associated with RSV disease exacerbation. This latter point is important since the first FI-hRSV vaccine failed to prevent hRSV infection, and even worse vaccinated children had an increased risk of severe disease after hRSV infection (7). As described above, we have previously observed in our clinical work that rBCG-N-hRSV is immunogenic without causing immune enhancement disease in mice (11, 15). Further, in

the present phase I clinical study, we did not find any related severe adverse events in response to the rBCG-N-hRSV in healthy adult donors. All subjects had a follow-up for 180 days, during which they could have been exposed to hRSV infection, and importantly, no severe disease was found in any subject.

# 15. TABLES, FIGURES, AND GRAPHS REFERRED TO BUT NOT INCLUDED IN THE TEXT

Table XXV: Listing of local adverse events by subjects.

<sup>\*\*</sup>AE type: local solicited AE (1), local non-solicited AE (2), general solicited AE (3), general AE (4), laboratory registered AE (5).

| Subject | | Vaccine | | AE | Day post | AE | Total AE |
|---|---|---|---|---|---|---|---|
| Number | Cohort | Type* | Diagnosis | type** | Vaccine | Start | Duration |
| RSV01 | Cohort A | 2 | Vaccine site sensitivity | 1 | 27-06-2017 | 27-06-2017 | 9 |
| RSV01 | Cohort A | 2 | Pain vaccination site | 1 | 28-06-2017 | 28-06-2017 | 1 |
| RSV01 | Cohort A | 2 | Erythema vaccination site | 1 | 29-06-2017 | 29-06-2017 | 1 |
| RSV01 | Cohort A | 2 | Vaccination site abscess | 1 | 18-07-2017 | 18-07-2017 | 65 |
| RSV01 | Cohort A | 2 | Vaccination site crust | 1 | 18-07-2017 | 18-07-2017 | 123 |
| RSV02 | Cohort A | 1 | Vaccine site sensitivity | 1 | 28-06-2017 | 28-06-2017 | 38 |
| RSV02 | Cohort A | 1 | Erythema vaccination site | 1 | 01-07-2017 | 01-07-2017 | 2 |
| RSV02 | Cohort A | 1 | Induration vaccination site | 1 | 30-06-2017 | 30-06-2017 | 1 |
| RSV02 | Cohort A | 1 | Pain vaccination site | 1 | 07-07-2017 | 07-07-2017 | 5 |
| RSV02 | Cohort A | 1 | Vaccination site abscess | 1 | 11-07-2017 | 11-07-2017 | 2 |
| RSV02 | Cohort A | 1 | Vaccination site crust | 1 | 11-07-2017 | 11-07-2017 | 67 |
| RSV03 | Cohort A | 1 | Pruritus vaccination site | 2 | 30-06-2017 | 30-06-2017 | 7 |
| RSV03 | Cohort A | 1 | Flaking vaccination site | 2 | 02-07-2017 | 02-07-2017 | 25 |
| RSV03 | Cohort A | 1 | Vaccine site sensitivity | 1 | 28-06-2017 | 28-06-2017 | 74 |
| RSV03 | Cohort A | 1 | Pain vaccination site | 1 | 29-06-2017 | 29-06-2017 | 3 |
| RSV03 | Cohort A | 1 | Vaccination site crust | 1 | 06-08-2017 | 06-08-2017 | 40 |
| RSV03 | Cohort A | 1 | Vaccination site abscess | 1 | 27-07-2017 | 27-07-2017 | 10 |
| RSV05 | Cohort A | 1 | Erythema vaccination site | 1 | 06-07-2017 | 06-07-2017 | 2 |
| RSV05 | Cohort A | 1 | Vaccine site sensitivity | 1 | 05-07-2017 | 05-07-2017 | 10 |
| RSV05 | Cohort A | 1 | Pain vaccination site | 1 | 07-07-2017 | 07-07-2017 | 5 |
| RSV05 | Cohort A | 1 | Vaccination site abscess | 1 | 22-07-2017 | 22-07-2017 | 3 |
| RSV05 | Cohort A | 1 | Vaccination site crust | 1 | 25-07-2017 | 25-07-2017 | 33 |
| RSV07 | Cohort A | 1 | Pain vaccination site | 1 | 13-07-2017 | 13-07-2017 | 10 |
| RSV07 | Cohort A | 1 | Vaccine site sensitivity | 1 | 16-07-2017 | 16-07-2017 | 11 |
| RSV07 | Cohort A | 1 | Pruritus vaccination site | 2 | 13-07-2017 | 13-07-2017 | 15 |
| RSV07 | Cohort A | 1 | Vaccination site abscess | 1 | 18-07-2017 | 18-07-2017 | 7 |
| RSV07 | Cohort A | 1 | Vaccination site crust | 1 | 23-07-2017 | 23-07-2017 | 74 |
| RSV10 | Cohort A | 1 | Tiredness in vaccinated arm | 2 | 10-07-2017 | 10-07-2017 | 1 |
| RSV10 | Cohort A | 1 | Vaccine site sensitivity | 1 | 10-07-2017 | 10-07-2017 | 17 |
| RSV10 | Cohort A | 1 | Pruritus vaccination site | 2 | 12-07-2017 | 12-07-2017 | 12 |
| RSV10 | Cohort A | 1 | Erythema vaccination site | 1 | 12-07-2017 | 12-07-2017 | 2 |

<sup>\*</sup>Vaccine type: rBCG-N-hRSV (1), WT-BCG (2).

| RSV10 | Cohort A | 1 | Pain vaccination site | 1 | 12-07-2017 | 12-07-2017 | 15 |
|---|---|---|---|---|---|---|---|
| RSV10 | Cohort A | 1 | Vaccination site abscess | 1 | 20-07-2017 | 20-07-2017 | 7 |
| RSV10 | Cohort A | 1 | Vaccination site crust | 1 | 20-07-2017 | 20-07-2017 | 131 |
| RSV10 | Cohort A | 1 | Induration vaccination site | 1 | 11-07-2017 | 11-07-2017 | 1 |
| RSV13 | Cohort A | 2 | Pruritus vaccination site | 2 | 18-07-2017 | 18-07-2017 | 6 |
| RSV13 | Cohort A | 2 | Vaccine site sensitivity | 1 | 18-07-2017 | 18-07-2017 | 2 |
| RSV13 | Cohort A | 2 | Erythema vaccination site | 1 | 18-07-2017 | 18-07-2017 | 3 |
| RSV13 | Cohort A | 2 | Vaccination site abscess | 1 | 27-07-2017 | 27-07-2017 | 15 |
| RSV13 | Cohort A | 2 | Vaccination site crust | 1 | 27-07-2017 | 27-07-2017 | 137 |
| RSV13 | Cohort A | 2 | Pain vaccination site | 1 | 24-07-2017 | 24-07-2017 | 3 |
| RSV14 | Cohort A | 1 | Pain vaccination site | 1 | 19-07-2017 | 19-07-2017 | 17 |
| RSV14 | Cohort A | 1 | Vaccine site sensitivity | 1 | 19-07-2017 | 19-07-2017 | 28 |
| RSV14 | Cohort A | 1 | Vaccination site abscess | 1 | 02-08-2017 | 02-08-2017 | 1 |
| RSV14 | Cohort A | 1 | Vaccination site crust | 1 | 03-08-2017 | 03-08-2017 | 11 |
| RSV14 | Cohort A | 1 | Pruritus vaccination site | 2 | 22-07-2017 | 22-07-2017 | 5 |
| RSV14 | Cohort A | 1 | Flaking vaccination site | 2 | 16-08-2017 | 16-08-2017 | 8 |
| RSV16 | Cohort B | 1 | Vaccine site sensitivity | 1 | 02-10-2017 | 02-10-2017 | 11 |
| RSV16 | Cohort B | 1 | Induration vaccination site | 1 | 03-10-2017 | 03-10-2017 | 20 |
| RSV16 | Cohort B | 1 | Pruritus vaccination site | 2 | 06-10-2017 | 06-10-2017 | 1 |
| RSV16 | Cohort B | 1 | Left axillary lymphadenopathy | 1 | 06-10-2017 | 06-10-2017 | 3 |
| RSV16 | Cohort B | 1 | Vaccination site crust | 1 | 14-10-2017 | 14-10-2017 | 170 |
| RSV16 | Cohort B | 1 | Vaccination site abscess | 1 | 15-10-2017 | 15-10-2017 | 4 |
| RSV17 | Cohort B | 1 | Erythema vaccination site | 1 | 03-10-2017 | 03-10-2017 | 4 |
| RSV17 | Cohort B | 1 | Vaccine site sensitivity | 1 | 03-10-2017 | 03-10-2017 | 13 |
| RSV17 | Cohort B | 1 | Induration vaccination site | 1 | 03-10-2017 | 03-10-2017 | 4 |
| RSV17 | Cohort B | 1 | Pain vaccination site | 1 | 03-10-2017 | 03-10-2017 | 13 |
| RSV17 | Cohort B | 1 | Vaccination site abscess | 1 | 12-10-2017 | 12-10-2017 | 75 |
| RSV17 | Cohort B | 1 | Vaccination site crust | 1 | 13-10-2017 | 13-10-2017 | 92 |
| RSV18 | Cohort B | 2 | Vaccine site sensitivity | 1 | 04-10-2017 | 04-10-2017 | 13 |
| RSV18 | Cohort B | 2 | Erythema vaccination site | 1 | 04-10-2017 | 04-10-2017 | 4 |
| RSV18 | Cohort B | 2 | Induration vaccination site | 1 | 05-10-2017 | 05-10-2017 | 9 |
| RSV18 | Cohort B | 2 | Pain vaccination site | 1 | 10-10-2017 | 10-10-2017 | 3 |
| RSV18 | Cohort B | 2 | Vaccination site abscess | 1 | 09-10-2017 | 09-10-2017 | 7 |
| RSV18 | Cohort B | 2 | Vaccination site crust | 1 | 14-10-2017 | 14-10-2017 | 142 |
| RSV24 | Cohort B | 2 | Pain vaccination site | 1 | 03-10-2017 | 03-10-2017 | 12 |
| RSV24 | Cohort B | 2 | Vaccine site sensitivity | 1 | 03-10-2017 | 03-10-2017 | 15 |
| RSV24 | Cohort B | 2 | Erythema vaccination site | 1 | 04-10-2017 | 04-10-2017 | 7 |
| RSV24 | Cohort B | 2 | Induration vaccination site | 1 | 04-10-2017 | 04-10-2017 | 6 |
| RSV24 | Cohort B | 2 | Vaccination site abscess | 1 | 14-10-2017 | 14-10-2017 | 13 |
| RSV24 | Cohort B | 2 | Vaccination site crust | 1 | 18-10-2017 | 18-10-2017 | 34 |
| RSV25 | Cohort B | 1 | Pain vaccination site | 1 | 05-10-2017 | 05-10-2017 | 1 |
| RSV25 | Cohort B | 1 | Vaccine site sensitivity | 1 | 05-10-2017 | 05-10-2017 | 1 |

| RSV25 | Cohort B | 1 | Erythema vaccination site | 1 | 06-10-2017 | 06-10-2017 | 8 |
|---|---|---|---|---|---|---|---|
| RSV25 | Cohort B | 1 | Vaccination site abscess | 1 | 06-10-2017 | 06-10-2017 | 6 |
| RSV25 | Cohort B | 1 | Induration vaccination site | 1 | 07-10-2017 | 07-10-2017 | 37 |
| RSV25 | Cohort B | 1 | Vaccination site crust | 1 | 08-10-2017 | 08-10-2017 | 51 |
| RSV26 | Cohort B | 1 | Pain vaccination site | 1 | 04-10-2017 | 04-10-2017 | 8 |
| RSV26 | Cohort B | 1 | Vaccine site sensitivity | 1 | 04-10-2017 | 04-10-2017 | 13 |
| RSV26 | Cohort B | 1 | Erythema vaccination site | 1 | 05-10-2017 | 05-10-2017 | 16 |
| RSV26 | Cohort B | 1 | Vaccination site abscess | 1 | 11-10-2017 | 11-10-2017 | 5 |
| RSV26 | Cohort B | 1 | Ulcer vaccination site | 2 | 17-10-2017 | 17-10-2017 | 2 |
| RSV26 | Cohort B | 1 | Vaccination site crust | 1 | 15-10-2017 | 15-10-2017 | 91 |
| RSV27 | Cohort B | 1 | Induration vaccination site | 1 | 18-10-2017 | 18-10-2017 | 11 |
| RSV27 | Cohort B | 1 | Erythema vaccination site | 1 | 05-10-2017 | 05-10-2017 | 15 |
| RSV27 | Cohort B | 1 | Pain vaccination site | 1 | 04-10-2017 | 04-10-2017 | 14 |
| RSV27 | Cohort B | 1 | Vaccine site sensitivity | 1 | 04-10-2017 | 04-10-2017 | 11 |
| RSV27 | Cohort B | 1 | Pruritus vaccination site | 2 | 09-10-2017 | 09-10-2017 | 2 |
| RSV27 | Cohort B | 1 | Vaccination site abscess | 1 | 12-10-2017 | 12-10-2017 | 7 |
| RSV27 | Cohort B | 1 | Vaccination site crust | 1 | 18-10-2017 | 18-10-2017 | 143 |
| RSV30 | Cohort B | 1 | Vaccine site sensitivity | 1 | 10-10-2017 | 10-10-2017 | 10 |
| RSV30 | Cohort B | 1 | Pruritus vaccination site | 2 | 11-10-2017 | 11-10-2017 | 7 |
| RSV30 | Cohort B | 1 | Left axillary pain | 2 | 10-10-2017 | 10-10-2017 | 1 |
| RSV30 | Cohort B | 1 | Vaccination site crust | 1 | 21-10-2017 | 21-10-2017 | 19 |
| RSV30 | Cohort B | 1 | Pain vaccination site | 1 | 18-10-2017 | 18-10-2017 | 5 |
| RSV30 | Cohort B | 1 | Vaccination site abscess | 1 | 19-10-2017 | 19-10-2017 | 3 |
| RSV32 | Cohort C | 1 | Pain vaccination site | 1 | 21-11-2017 | 21-11-2017 | 15 |
| RSV32 | Cohort C | 1 | Vaccine site sensitivity | 1 | 22-11-2017 | 22-11-2017 | 18 |
| RSV32 | Cohort C | 1 | Erythema vaccination site | 1 | 22-11-2017 | 22-11-2017 | 12 |
| RSV32 | Cohort C | 1 | Vaccination site abscess | 1 | 27-11-2017 | 27-11-2017 | 110 |
| RSV32 | Cohort C | 1 | Induration vaccination site | 1 | 23-11-2017 | 23-11-2017 | 32 |
| RSV32 | Cohort C | 1 | Vaccination site crust | 1 | 27-11-2017 | 27-11-2017 | 202 |
| RSV33 | Cohort C | 1 | Pain vaccination site | 1 | 21-11-2017 | 21-11-2017 | 10 |
| RSV33 | Cohort C | 1 | Vaccine site sensitivity | 1 | 21-11-2017 | 21-11-2017 | 10 |
| RSV33 | Cohort C | 1 | Erythema vaccination site | 1 | 23-11-2017 | 23-11-2017 | 4 |
| RSV33 | Cohort C | 1 | Vaccination site abscess | 1 | 26-11-2017 | 26-11-2017 | 5 |
| RSV33 | Cohort C | 1 | Vaccination site crust | 1 | 28-11-2017 | 28-11-2017 | 67 |
| RSV33 | Cohort C | 1 | Induration vaccination site | 1 | 28-11-2017 | 28-11-2017 | 1 |
| RSV34 | Cohort C | 2 | Pain vaccination site | 1 | 21-11-2017 | 21-11-2017 | 18 |
| RSV34 | Cohort C | 2 | Vaccine site sensitivity | 1 | 22-11-2017 | 22-11-2017 | 5 |
| RSV34 | Cohort C | 2 | Erythema vaccination site | 1 | 22-11-2017 | 22-11-2017 | 3 |
| RSV34 | Cohort C | 2 | Induration vaccination site | 1 | 23-11-2017 | 23-11-2017 | 1 |
| RSV34 | Cohort C | 2 | Pruritus vaccination site | 2 | 24-11-2017 | 24-11-2017 | 17 |
| RSV34 | Cohort C | 2 | Vaccination site abscess | 1 | 04-12-2017 | 04-12-2017 | 63 |
| RSV34 | Cohort C | 2 | Vaccination site crust | 1 | 20-02-2018 | 20-02-2018 | 63 |

| RSV36 | Cohort C | 1 | Vaccine site sensitivity | 1 | 27-11-2017 | 27-11-2017 | 55 |
|---|---|---|---|---|---|---|---|
| RSV36 | Cohort C | 1 | Erythema vaccination site | 1 | 28-11-2017 | 28-11-2017 | 8 |
| RSV36 | Cohort C | 1 | Pain vaccination site | 1 | 28-11-2017 | 28-11-2017 | 11 |
| RSV36 | Cohort C | 1 | Vaccination site abscess | 1 | 01-12-2017 | 01-12-2017 | 5 |
| RSV36 | Cohort C | 1 | Vaccination site crust | 1 | 04-12-2017 | 04-12-2017 | 44 |
| RSV36 | Cohort C | 1 | Ulcer vaccination site | 2 | 15-12-2017 | 15-12-2017 | 14 |
| RSV38 | Cohort C | 2 | Vaccine site sensitivity | 1 | 27-11-2017 | 27-11-2017 | 38 |
| RSV38 | Cohort C | 2 | Pain vaccination site | 1 | 27-11-2017 | 27-11-2017 | 21 |
| RSV38 | Cohort C | 2 | Erythema vaccination site | 1 | 28-11-2017 | 28-11-2017 | 2 |
| RSV38 | Cohort C | 2 | Pruritus vaccination site | 2 | 29-11-2017 | 29-11-2017 | 7 |
| RSV38 | Cohort C | 2 | Vaccination site abscess | 1 | 05-12-2017 | 05-12-2017 | 6 |
| RSV38 | Cohort C | 2 | Vaccination site crust | 1 | 08-12-2017 | 08-12-2017 | 36 |
| RSV38 | Cohort C | 2 | Ulcer vaccination site | 2 | 27-12-2017 | 27-12-2017 | 10 |
| RSV40 | Cohort C | 1 | Vaccine site sensitivity | 1 | 28-11-2017 | 28-11-2017 | 19 |
| RSV40 | Cohort C | 1 | Pain vaccination site | 1 | 04-12-2017 | 04-12-2017 | 11 |
| RSV40 | Cohort C | 1 | Erythema vaccination site | 1 | 04-12-2017 | 04-12-2017 | 5 |
| RSV40 | Cohort C | 1 | Induration vaccination site | 1 | 06-12-2017 | 06-12-2017 | 1 |
| RSV40 | Cohort C | 1 | Vaccination site abscess | 1 | 04-12-2017 | 04-12-2017 | 28 |
| RSV40 | Cohort C | 1 | Vaccination site crust | 1 | 05-12-2017 | 05-12-2017 | 27 |
| RSV40 | Cohort C | 1 | Ulcer vaccination site | 2 | 01-01-2018 | 01-01-2018 | 15 |
| RSV41 | Cohort C | 1 | Vaccine site sensitivity | 1 | 28-11-2017 | 28-11-2017 | 15 |
| RSV41 | Cohort C | 1 | Pain vaccination site | 1 | 29-11-2017 | 29-11-2017 | 7 |
| RSV41 | Cohort C | 1 | Vaccination site abscess | 1 | 30-11-2017 | 30-11-2017 | 8 |
| RSV41 | Cohort C | 1 | Induration vaccination site | 1 | 01-12-2017 | 01-12-2017 | 1 |
| RSV41 | Cohort C | 1 | Vaccination site crust | 1 | 03-12-2017 | 03-12-2017 | 185 |
| RSV41 | Cohort C | 1 | Erythema vaccination site | 1 | 06-12-2017 | 06-12-2017 | 1 |
| RSV42 | Cohort C | 1 | Vaccine site sensitivity | 1 | 04-12-2017 | 04-12-2017 | 14 |
| RSV42 | Cohort C | 1 | Pain vaccination site | 1 | 05-12-2017 | 05-12-2017 | 6 |
| RSV42 | Cohort C | 1 | Erythema vaccination site | 1 | 05-12-2017 | 05-12-2017 | 6 |
| RSV42 | Cohort C | 1 | Vaccination site abscess | 1 | 06-12-2017 | 06-12-2017 | 7 |
| RSV42 | Cohort C | 1 | left axillary pain | 1 | 07-12-2017 | 07-12-2017 | 7 |
| RSV42 | Cohort C | 1 | Vaccination site crust | 1 | 11-12-2017 | 11-12-2017 | 103 |

### Table XXVI: Listing of general adverse events by subjects.

<sup>\*\*</sup>AE type: local solicited AE (1), local non-solicited AE (2), general solicited AE (3), general AE (4), laboratory registered AE (5).

| Subject | | Vaccine | AE | | AE | Day<br>post | AE | AE |
|---|---|---|---|---|---|---|---|---|
| N° | Cohort | Type* | N° | Diagnosis | Туре | Vaccine | Start | End |
| | Cohort | | | Hypophosphate | | | 05-07- | 13-07- |
| RSV01 | Α | 2 | 1 | mia | 5 | 8 | 2017 | 2017 |

<sup>\*</sup>Vaccine type: rBCG-N-hRSV (1), WT-BCG (2).

| i | | 1 1 | | Ī | | ı | | L 40.0= |
|---|---|---|---|---|---|---|---|---|
| DC)/04 | Cohort | | 0 | I long a mailte a maile | _ | 0 | 05-07- | 13-07- |
| RSV01 | Cohort | 2 | 2 | Hyperglycemia | 5 | 8 | 2017<br>10-07- | 2017<br>10-07- |
| RSV01 | A | 2 | 3 | Sickness | 3 | 13 | 2017 | 2017 |
| KSVUI | Cohort | 2 | 3 | Left wrist | 3 | 13 | 06-07- | 22-09- |
| RSV01 | A | 2 | 4 | contusion | 4 | 9 | 2017 | 2017 |
| KSVUI | Cohort | 2 | 4 | Vaccine site | 4 | 9 | 27-06- | 29-06- |
| RSV01 | A | 2 | 5 | sensitivity | 1 | 0 | 2017 | 2017 |
| 113701 | Cohort | | <u> </u> | Pain vaccination | ' | 0 | 28-06- | 28-06- |
| RSV01 | A | 2 | 6 | site | 1 | 1 | 2017 | 2017 |
| 110701 | Cohort | | | Erythema | | · · | 29-06- | 29-06- |
| RSV01 | A | 2 | 7 | vaccination site | 1 | 2 | 2017 | 2017 |
| | Cohort | _ | • | Decreased | | | 05-07- | Continu |
| RSV01 | A | 2 | 8 | hemoglobin | 5 | 8 | 2017 | es |
| | Cohort | | | Vaccination site | | - | 18-07- | 20-09- |
| RSV01 | Α | 2 | 9 | abscess | 1 | 21 | 2017 | 2017 |
| | Cohort | | | | | | 27-07- | 21-08- |
| RSV01 | Α | 2 | 10 | Proteinuria | 5 | 30 | 2017 | 2017 |
| | Cohort | | | | | | 27-07- | 21-08- |
| RSV01 | Α | 2 | 11 | Leukocytosis | 5 | 30 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 14-07- | 17-07- |
| RSV01 | Α | 2 | 12 | sensitivity | 1 | 17 | 2017 | 2017 |
| | Cohort | | | | | | 10-07- | 10-07- |
| RSV01 | Α | 2 | 13 | Abdominal pain | 4 | 13 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 18-07- | 17-11- |
| RSV01 | Α | 2 | 14 | crust | 1 | 21 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 20-07- | 21-07- |
| RSV01 | Α | 2 | 15 | sensitivity | 1 | 23 | 2017 | 2017 |
| | Cohort | | | | | | 21-08- | 24-10- |
| RSV01 | Α | 2 | 16 | Hematuria | 5 | 55 | 2017 | 2017 |
| 50,404 | Cohort | | | | _ | | 23-08- | 24-10- |
| RSV01 | A | 2 | 17 | Proteinuria | 5 | 57 | 2017 | 2017 |
| D0) (04 | Cohort | | 40 | D'andres | 0 | 40 | 09-07- | 09-07- |
| RSV01 | A | 2 | 18 | Diarrhea | 3 | 12 | 2017 | 2017 |
| RSV01 | Cohort | 2 | 19 | Haadaaha | 3 | 12 | 09-07- | 09-07-<br>2017 |
| KSVUI | A<br>Cohort | 2 | 19 | Headache | 3 | 12 | 2017<br>24-10- | 26-10- |
| RSV01 | A | 2 | 20 | Hypernatremia | 5 | 119 | 2017 | 2017 |
| 113701 | Cohort | | 20 | Пуретнапенна | J | 113 | 04-07- | 11-07- |
| RSV02 | A | 1 | 1 | Leukopenia | 5 | 6 | 2017 | 2017 |
| 110102 | Cohort | | • | Lounopoilla | | ŭ | 04-07- | 11-07- |
| RSV02 | A | 1 1 | 2 | Neutropenia | 5 | 6 | 2017 | 2017 |
| | Cohort | | | | | - | 04-07- | 11-07- |
| RSV02 | Α | 1 | 3 | Increase in CPK | 5 | 6 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 28-06- | 04-08- |
| RSV02 | Α | 1 | 4 | sensitivity | 1 | 0 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 01-07- | 01-07- |
| RSV02 | Α | 1 | 5 | vaccination site | 1 | 3 | 2017 | 2017 |
| | Cohort | 1 | | Induration | | | 30-06- | 30-06- |
| RSV02 | Α | 1 | 6 | vaccination site | 1 | 2 | 2017 | 2017 |
| | Cohort | _ | _ | Pain vaccination | | _ | 07-07- | 11-07- |
| RSV02 | A | 1 | 7 | site | 1 | 9 | 2017 | 2017 |
| DO: (22 | Cohort | | _ | Decrease | _ | 4.0 | 11-07- | 24-07- |
| RSV02 | A | 1 | 8 | hemoglobin | 5 | 13 | 2017 | 2017 |
| D67/00 | Cohort | | 0 | Vaccination site | 4 | 40 | 11-07-<br>2017 | 11-07- |
| RSV02 | A<br>Cohort | 1 | 9 | abscess | 1 | 13 | 11-07- | 2017<br>11-07- |
| RSV02 | A | 1 | 10 | Diarrhea | 3 | 13 | 2017 | 2017 |
| 113702 | Cohort | <u>'</u> | 10 | Diaiiiica | J | 13 | 13-07- | 13-07- |
| RSV02 | A | 1 1 | 11 | Diarrhea | 3 | 15 | 2017 | 2017 |
| 1.0002 | Cohort | <del> </del> | | Erythema | J | 10 | 04-07- | 04-07- |
| RSV02 | A | 1 | 12 | vaccination site | 1 | 6 | 2017 | 2017 |
| | Cohort | · | 14 | . acciation one | · | , | 24-07- | Continu |
| RSV02 | A | 1 | 13 | Leukopenia | 5 | 26 | 2017 | es |
| | Cohort | <u> </u> | | Vaccination site | | | 11-07- | 15-09- |
| RSV02 | A | 1 | 14 | crust | 1 | 13 | 2017 | 2017 |
| | <u> </u> | | | | | | | |

| | Cobort | l I | | | I I | | 22.00 | 1 25 10 |
|---|---|---|---|---|---|---|---|---|
| RSV02 | Cohort<br>A | 1 | 15 | Lymphopenia | 5 | 55 | 22-08-<br>2017 | 25-10-<br>2017 |
| 110102 | Cohort | | 10 | Бутрпоротіа | Ü | - 00 | 09-07- | 09-07- |
| RSV02 | Α | 1 | 16 | Diarrhea | 3 | 11 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 15-07- | 15-07- |
| RSV02 | A | 1 | 17 | crust | 1 | 17 | 2017 | 2017 |
| DCV02 | Cohort | 1 | 18 | Ingresses in CDV | 5 | 110 | 25-10-<br>2017 | 18-12- |
| RSV02 | A<br>Cohort | I | 10 | Increase in CPK | 5 | 119 | 18-12- | 2017<br>26-12- |
| RSV02 | A | 1 | 19 | Hyperglycemia | 5 | 173 | 2017 | 2017 |
| | Cohort | | - | Decreased | | | 18-12- | Continu |
| RSV02 | Α | 1 | 20 | hemoglobin | 5 | 173 | 2017 | es |
| | Cohort | | | Pruritus | | _ | 30-06- | 06-07- |
| RSV03 | A<br>Cohort | 1 | 1 | vaccination site | 2 | 3 | 2017<br>02-07- | 2017 |
| RSV03 | A | 1 | 2 | Flaking vaccination site | 2 | 5 | 2017 | 26-07-<br>2017 |
| 110 7 0 0 | Cohort | ' | | vaccination site | | | 08-07- | 24-07- |
| RSV03 | A | 1 | 3 | Common cold | 4 | 11 | 2017 | 2017 |
| | Cohort | | | | | | 04-07- | 10-07- |
| RSV03 | Α | 1 | 4 | Increase in CPK | 5 | 7 | 2017 | 2017 |
| RSV03 | Cohort | 1 | 5 | Hypoproteinemi | 5 | 7 | 04-07- | 10-07- |
| K5V03 | A<br>Cohort | I | ეე | Vaccine site | 5 | - 1 | 2017<br>28-06- | 2017<br>03-07- |
| RSV03 | A | 1 | 6 | sensitivity | 1 | 1 | 2017 | 2017 |
| 110100 | Cohort | · | | Pain vaccination | | | 29-06- | 30-06- |
| RSV03 | Α | 1 | 7 | site | 1 | 2 | 2017 | 2017 |
| | Cohort | | | Decrease | | | 04-07- | 10-07- |
| RSV03 | A | 1 | 8 | hemoglobin | 5 | 7 | 2017 | 2017 |
| RSV03 | Cohort<br>A | 1 | 9 | Fatigue | 3 | 22 | 19-07-<br>2017 | 19-07-<br>2017 |
| 113703 | Cohort | ' | 9 | i aligue | 3 | | 21-07- | 23-07- |
| RSV03 | A | 1 | 10 | Fatigue | 3 | 24 | 2017 | 2017 |
| | Cohort | | | <u> </u> | | | 18-07- | 19-07- |
| RSV03 | Α | 1 | 11 | Headache | 3 | 21 | 2017 | 2017 |
| DC//02 | Cohort | 1 | 12 | Haadaaha | 3 | 24 | 21-07- | 23-07- |
| RSV03 | A<br>Cohort | I | 12 | Headache | 3 | 24 | 2017<br>22-07- | 2017 |
| RSV03 | A | 1 | 13 | Myalgia | 3 | 25 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 07-07- | 09-07- |
| RSV03 | Α | 1 | 14 | sensitivity | 1 | 10 | 2017 | 2017 |
| DO: (00 | Cohort | | 4-5 | Vaccine site | | 4.4 | 11-07- | 16-07- |
| RSV03 | A<br>Cohort | 1 | 15 | sensitivity Vaccine site | 1 | 14 | 2017<br>18-07- | 2017<br>14-09- |
| RSV03 | A | 1 | 16 | sensitivity | 1 | 21 | 2017 | 2017 |
| | Cohort | | | Decrease | | | 31-07- | 31-08- |
| RSV03 | Α | 1 | 17 | hemoglobin | 5 | 34 | 2017 | 2017 |
| 50.400 | Cohort | | | | _ | | 31-07- | 27-12- |
| RSV03 | A | 1 | 18 | Leukopenia | 5 | 34 | 2017 | 2017 |
| RSV03 | Cohort<br>A | 1 | 19 | Vaccination site<br>crust | 1 | 40 | 06-08-<br>2017 | 14-09-<br>2017 |
| 110 000 | Cohort | 1 | 19 | Vaccination site | ' | 40 | 27-07- | 05-08- |
| RSV03 | A | 1 | 20 | abscess | 1 | 30 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 22-07- | 22-07- |
| RSV03 | Α | 1 | 21 | site | 1 | 25 | 2017 | 2017 |
| DC//02 | Cohort | | 22 | Tachyaardia | 2 | 4 | 28-06- | 28-06- |
| RSV03 | A<br>Cohort | 1 | 22 | Tachycardia | 3 | 1 | 2017<br>22-11- | 2017 |
| RSV03 | A | 1 | 23 | Headache | 4 | 148 | 2017 | 2017 |
| | Cohort | | | Puncture site | | | 05-07- | 10-07- |
| RSV05 | Α | 1 | 1 | ecchymosis | 4 | 1 | 2017 | 2017 |
| DOV (0.5 | Cohort | | _ | 11 ( | | _ | 06-07- | 06-07- |
| RSV05 | Cohort | 1 | 2 | Hypertension | 3 | 2 | 2017<br>06-07- | 2017<br>07-07- |
| RSV05 | Cohort<br>A | 1 | 3 | Erythema vaccination site | 1 | 2 | 2017 | 2017 |
| 1,0 000 | Cohort | <del>' </del> | <u> </u> | Vaccine site | <u>'</u> | | 05-07- | 08-07- |
| RSV05 | A | 1 | 4 | sensitivity | 1 | 1 | 2017 | 2017 |

| 1 | Louisia | 1 1 | | l per en en en en en en | i | Ī | 07.07 | 1 07 07 |
|---|---|---|---|---|---|---|---|---|
| RSV05 | Cohort | _ | 5 | Pain vaccination | 1 | 3 | 07-07-<br>2017 | 07-07- |
| RSVUS | A<br>Cohort | 1 | 5 | site | 1 | 3 | 12-07- | 2017<br>19-07- |
| RSV05 | | 1 | 6 | Decreased | 5 | 8 | 2017 | 2017 |
| K5V05 | A<br>Cohort | I | 0 | hemoglobin | 5 | 0 | 12-07- | 13-07- |
| RSV05 | | 1 | 7 | Headache | 3 | 8 | 2017 | 2017 |
| K5V05 | Cohort | I | | пеацаспе | 3 | 0 | 12-07- | 14-07- |
| RSV05 | | 1 | 8 | Bilateral Otalgia | 4 | 8 | 2017 | 2017 |
| K5V05 | Cohort | I | 0 | Retro ocular left | 4 | 0 | 12-07- | 13-07- |
| RSV05 | A | 1 | 9 | pain | 4 | 8 | 2017 | 2017 |
| N3V03 | Cohort | ' | 3 | pairi | 4 | 0 | 12-07- | 12-07- |
| RSV05 | A | 1 | 10 | Fatigue | 3 | 8 | 2017 | 2017 |
| 110 7 0 3 | Cohort | ' | 10 | Tauguc | <u> </u> | | 19-07- | 07-08- |
| RSV05 | A | 1 | 11 | Increase in CPK | 5 | 15 | 2017 | 2017 |
| 113703 | Cohort | ' | 11 | IIICICase III CI IX | J | 13 | 18-07- | 02-08- |
| RSV05 | A | 1 | 12 | Tonsillitis | 4 | 14 | 2017 | 2017 |
| 110 100 | Cohort | | 12 | Pain vaccination | | 17 | 20-07- | 23-07- |
| RSV05 | A | 1 | 13 | site | 1 | 16 | 2017 | 2017 |
| 110100 | Cohort | | 10 | Vaccine site | | 10 | 20-07- | 25-07- |
| RSV05 | A | 1 | 14 | sensitivity | 1 | 16 | 2017 | 2017 |
| 110 100 | Cohort | | 1-7 | Vaccination site | | 10 | 22-07- | 24-07- |
| RSV05 | A | 1 | 15 | abscess | 1 | 18 | 2017 | 2017 |
| 110100 | Cohort | | 10 | авссосс | | | 22-07- | 23-07- |
| RSV05 | A | 1 | 16 | Headache | 3 | 18 | 2017 | 2017 |
| 110100 | Cohort | • | | Tioddaciio | | 10 | 27-07- | 28-07- |
| RSV05 | A | 1 | 17 | Headache | 3 | 23 | 2017 | 2017 |
| 110100 | Cohort | · | | Tioddaciio | | 20 | 22-07- | 23-07- |
| RSV05 | A | 1 | 18 | Fatigue | 3 | 18 | 2017 | 2017 |
| 110100 | Cohort | | | rangao | | | 27-07- | 28-07- |
| RSV05 | A | 1 | 19 | Fatigue | 3 | 23 | 2017 | 2017 |
| | Cohort | · | | Vaccination site | | | 25-07- | 26-08- |
| RSV05 | A | 1 | 20 | crust | 1 | 21 | 2017 | 2017 |
| | Cohort | | | | - | | 12-07- | 12-07- |
| RSV05 | A | 1 | 21 | Sickness | 3 | 8 | 2017 | 2017 |
| | Cohort | | | | | | 07-09- | 10-09- |
| RSV05 | Α | 1 | 22 | Common cold | 4 | 65 | 2017 | 2017 |
| | Cohort | | | Decrease | | | 25-10- | Continu |
| RSV05 | Α | 1 | 23 | haemoglobin | 5 | 113 | 2017 | es |
| | Cohort | | | | | | 25-10- | 29-12- |
| RSV05 | Α | 1 | 24 | Increase in CPK | 5 | 113 | 2017 | 2017 |
| | Cohort | | | Acute | | | 25-12- | 01-01- |
| RSV05 | Α | 1 | 25 | gastroenteritis | 4 | 174 | 2017 | 2018 |
| | Cohort | | | | | | 10-07- | 12-07- |
| RSV07 | Α | 1 | 1 | Common cold | 4 | 0 | 2017 | 2017 |
| | Cohort | | | | | | 10-07- | 10-07- |
| RSV07 | Α | 1 | 2 | Headache | 3 | 0 | 2017 | 2017 |
| DO: 45- | Cohort | ] | _ | Pain vaccination | | | 13-07- | 14-07- |
| RSV07 | A | 1 | 3 | site | 1 | 3 | 2017 | 2017 |
| D0: 40= | Cohort | | | 11 | _ | _ | 13-07- | 13-07- |
| RSV07 | A | 1 | 4 | Headache | 3 | 3 | 2017 | 2017 |
| D0\/07 | Cohort | | _ | Vaccine site | | _ | 16-07- | 26-07- |
| RSV07 | A | 1 | 5 | sensitivity | 1 | 6 | 2017 | 2017 |
| DC) (0.7 | Cohort | | _ | Llumotara: | _ | _ | 17-07- | 17-07- |
| RSV07 | A | 1 | 6 | Hypotension | 3 | 7 | 2017 | 2017 |
| DC\/07 | Cohort | | - | Drotoinurio | _ | 7 | 17-07- | 26-07- |
| RSV07 | A | 1 | 7 | Proteinuria | 5 | 7 | 2017<br>17-07- | 2017 |
| RSV07 | Cohort | 1 | 8 | Increase in CPK | 5 | 7 | - | 26-07-<br>2017 |
| 13701 | A | '- | 0 | Pruritus | ິ | <del> </del> | 2017<br>13-07- | 26-07- |
| RSV07 | Cohort | 1 | 10 | | 2 | 3 | 13-07-<br>2017 | 26-07- |
| 13701 | A<br>Cohort | | 10 | vaccination site Hypercholestero | | 3 | 26-07- | 10-08- |
| RSV07 | A | 1 | 11 | lemia | 5 | 16 | 20-07- | 2017 |
| 10001 | Cohort | ' | 11 | TOTTILA | | 10 | 12-07- | 12-07- |
| RSV07 | A | 1 | 12 | Tachycardia | 3 | 2 | 2017 | 2017 |
| 1.0001 | Cohort | ' | 12 | racitycalula | | | 16-07- | 22-07- |
| RSV07 | A | 1 | 9 | Cough | 4 | 6 | 2017 | 22-07- |
| 110 4 0 1 | | 1 | 9 | Cougn | 4 | U | 2017 | 2011 |

| RSV07 | | 1 - | | | 1 | ı | | | |
|---|---|---|---|---|---|---|---|---|---|
| RSV07 | 501/05 | Cohort | | | Pain vaccination | | | 16-07- | 22-07- |
| RSV07 A | RSV07 | | 1 | 13 | site | 1 | 6 | | |
| RSV07 | | | | | | | | | |
| RSV07 A | RSV07 | | 1 | 14 | | 3 | 8 | | |
| Cohort | | Cohort | | | Vaccination site | | | | |
| RSV07 | RSV07 | | 1 | 15 | abscess | 1 | 8 | | |
| Cohort | | Cohort | | | Vaccination site | | | 23-07- | 04-10- |
| RSV07 A | RSV07 | Α | 1 | 16 | crust | 1 | 13 | 2017 | 2017 |
| RSV07 | | Cohort | | | Decreased | | | 10-08- | 08-09- |
| RSV07 | RSV07 | Α | 1 | 17 | haemoglobin | 5 | 31 | 2017 | 2017 |
| RSV07 | | Cohort | | | Vaccination site | | | 19-08- | |
| RSV07 | RSV07 | Α | 1 | 18 | abscess | 1 | 40 | | 2017 |
| Cohort | | Cohort | | | Pain vaccination | | | 19-08- | 19-08- |
| RSV07 | RSV07 | Α | 1 | 19 | site | 1 | 40 | 2017 | 2017 |
| RSV07 | | Cohort | | | Wisdom tooth | | | 17-08- | |
| RSV07 | RSV07 | Α | 1 | 20 | pain | 4 | 38 | 2017 | 2017 |
| RSV07 | | Cohort | | | Pruritus | | | 13-07- | 13-07- |
| RSV07 | RSV07 | Α | 1 | 21 | vaccination site | 2 | 3 | 2017 | 2017 |
| RSV07 | | Cohort | | | Wisdom tooth | | | 21-08- | |
| Cohort | RSV07 | | 1 | 22 | | 4 | 42 | | |
| RSV07 | | Cohort | | | Wisdom tooth | | | | |
| RSV07 | RSV07 | | 1 | 23 | | 4 | 54 | 2017 | |
| RSV07 | | Cohort | | | Scratch in crust | | | | |
| RSV07 | RSV07 | | 1 | 24 | | 4 | 48 | | |
| RSV07 | | Cohort | | | Vaccination site | | - | | |
| New Note | RSV07 | | 1 | 25 | | 1 | 48 | | |
| RSV07 | | Cohort | | | Hypercholestero | | | | |
| RSV07 | RSV07 | | 1 | 26 | | 5 | 60 | | |
| RSV07 | | | | | | - | | | |
| RSV07 | RSV07 | | 1 | 27 | Headache | 3 | 9 | | |
| RSV07 | | Cohort | | | | | | | |
| RSV07 | RSV07 | _ | 1 | 28 | | 5 | 120 | - | |
| RSV07 A | | Cohort | | | Ŭ | | | | |
| RSV07 | RSV07 | | 1 | 29 | Pyuria | 5 | 120 | 2017 | |
| RSV07 A | | Cohort | | | | | | | |
| RSV10 A | RSV07 | | 1 | 30 | Increased TTPA | 5 | 120 | 2017 | 2018 |
| RSV10 A | | | | | Tiredness in | | | | |
| RSV10 A | | Cohort | | | vaccinated arm | | | 10-07- | |
| RSV10 A | RSV10 | | 1 | 1 | (left) | 2 | 0 | 2017 | 2017 |
| RSV10 A | | Cohort | | | Vaccine site | | | 10-07- | 10-07- |
| RSV10 A | RSV10 | | 1 | 2 | sensitivity | 1 | 0 | | 2017 |
| Name | | Cohort | | | Pruritus | | | 12-07- | 23-07- |
| RSV10 A | RSV10 | | 1 | 3 | vaccination site | 2 | 2 | 2017 | 2017 |
| Cohort Frythema 12-07- 13-07- 2017 2017 | | Cohort | | | Vaccine site | | | 11-07- | 27-07- |
| RSV10 A 1 5 vaccination site 1 2 2017 2017 RSV10 A 1 6 site 1 2 2017 2017 RSV10 A 1 7 Sickness 3 0 2017 2017 RSV10 A 1 8 abscess 1 10 2017 2017 RSV10 A 1 9 haemoglobin 5 14 2017 2017 RSV10 A 1 1 9 haemoglobin 5 14 2017 2017 RSV10 A 1 1 10 Increase in CPK 5 14 2017 2017 RSV10 A 1 1 1 crustomation site 1 1 2017 2017 RSV10 A 1 1 1 1 1 2017 2017 RSV10 A 1 1 | RSV10 | Α | 1 | 4 | sensitivity | 1 | 1 | 2017 | 2017 |
| RSV10 | | Cohort | | | Erythema | | | 12-07- | 13-07- |
| RSV10 A 1 6 site 1 2 2017 2017 RSV10 A 1 7 Sickness 3 0 2017 2017 RSV10 A 1 8 abscess 1 10 2017 2017 RSV10 A 1 9 haemoglobin 5 14 2017 2017 RSV10 A 1 10 Increase in CPK 5 14 2017 2017 RSV10 A 1 10 Increase in CPK 5 14 2017 2017 RSV10 A 1 1 cust 1 10 2017 2017 RSV10 A 1 1 1 1 1 1 1 1 2017 2017 RSV10 A 1 1 1 2 2017 2017 2017 2017 RSV10 A 1 1 < | RSV10 | Α | 1 | 5 | vaccination site | 1 | 2 | 2017 | 2017 |
| Cohort RSV10 A | | Cohort | | | Pain vaccination | | | 12-07- | 15-07- |
| RSV10 A 1 7 Sickness 3 0 2017 2017 RSV10 A 1 8 abscess 1 10 2017 24-07- RSV10 A 1 9 haemoglobin 5 14 2017 2017 RSV10 A 1 10 Increase in CPK 5 14 2017 2017 RSV10 A 1 11 crust 5 14 2017 2017 RSV10 A 1 11 crust 1 10 2017 27-11- RSV10 A 1 11 crust 1 10 2017 2017 RSV10 A 1 12 site 1 7 2017 2017 RSV10 A 1 12 site 1 7 2017 2017 RSV10 A 1 13 vaccination site 1 1 <td< td=""><td>RSV10</td><td>Α</td><td>1</td><td>6</td><td>site</td><td>1</td><td>2</td><td>2017</td><td>2017</td></td<> | RSV10 | Α | 1 | 6 | site | 1 | 2 | 2017 | 2017 |
| RSV10 | | Cohort | | | | | | | |
| RSV10 A 1 8 abscess 1 10 2017 2017 Cohort | RSV10 | Α | 1 | 7 | Sickness | 3 | 0 | 2017 | |
| RSV10 A | | Cohort | | | | | | | |
| RSV10 A 1 9 haemoglobin 5 14 2017 2017 RSV10 A 1 10 Increase in CPK 5 14 2017 2017 Cohort Vaccination site 20-07- 27-11- RSV10 A 1 11 crust 1 10 2017 2017 RSV10 A 1 12 site 1 7 2017 2017 RSV10 A 1 13 vaccination 1 1-07- 11-07- RSV10 A 1 13 vaccination site 1 1 2017 2017 RSV10 A 1 13 vaccination site 1 1 2017 2017 RSV10 A 1 13 vaccination site 1 1 2017 2017 | RSV10 | | 1 | 8 | abscess | 1 | 10 | | |
| Cohort | | Cohort | | | | | | | |
| RSV10 A 1 10 Increase in CPK 5 14 2017 2017 RSV10 A 1 11 crust 1 10 2017 27-11- RSV10 A 1 11 crust 1 10 2017 2017 RSV10 A 1 12 site 1 7 2017 2017 RSV10 A 1 13 vaccination 1 11-07- 11-07- RSV10 A 1 13 vaccination site 1 1 2017 2017 RSV10 A 1 13 vaccination site 1 1 2017 2017 RSV10 A 1 13 vaccination site 1 1 2017 2017 | RSV10 | | 1 | 9 | haemoglobin | 5 | 14 | | |
| Cohort | | Cohort | | | | | | | |
| RSV10 A 1 11 crust 1 10 2017 2017 Cohort Pain vaccination 17-07- 27-07- RSV10 A 1 12 site 1 7 2017 2017 Cohort Induration 11-07- 11-07- RSV10 A 1 13 vaccination site 1 1 2017 2017 Cohort Acute rhinopharyngou 15-08- 25-08- | RSV10 | | 1 | 10 | | 5 | 14 | | |
| RSV10 A 1 12 site 1 7 2017 2017 Cohort A 1 13 vaccination 1 1-07- 27-07- RSV10 A 1 13 vaccination 1 1-07- 11-07- Acute rhinopharyngou 15-08- 25-08- | | | | | | | | | |
| RSV10 A 1 12 site 1 7 2017 2017 Cohort Induration 11-07- 11-07- RSV10 A 1 13 vaccination site 1 1 2017 2017 Cohort Acute rhinopharyngou 15-08- 25-08- | RSV10 | | 1 | 11 | | 1 | 10 | | |
| RSV10 A 1 13 vaccination 1 11-07- 11-07- 2017 Acute rhinopharyngou 15-08- 25-08- | | | | | | | | | |
| RSV10 A 1 13 vaccination site 1 1 2017 2017 | RSV10 | | 1 | 12 | | 1 | 7 | | |
| Cohort Acute rhinopharyngou 15-08- 25-08- | | | | | | | | | |
| Cohort rhinopharyngou 15-08- 25-08- | RSV10 | Α | 1 | 13 | | 1 | 1 | 2017 | 2017 |
| RSV10 A 1 14 sitis 4 36 2017 2017 | D01//0 | | | | | _ | | | |
| | RSV10 | A | 1 | 14 | sitis | 4 | 36 | 2017 | 2017 |

| İ | Cohort | | | | | | 15-08- | 16-08- |
|---|---|---|---|---|---|---|---|---|
| RSV10 | Α | 1 | 15 | Fever | 4 | 36 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 21-09- | 22-09- |
| RSV10 | Α | 1 | 16 | abscess | 1 | 73 | 2017 | 2017 |
| | Cohort | | | Acute | | | 04-11- | 23-11- |
| RSV10 | Α | 1 | 17 | pharyngitis | 4 | 117 | 2017 | 2017 |
| | Cohort | | | | | | 07-11- | 06-01- |
| RSV10 | Α | 1 | 18 | Hypoglycemia | 5 | 120 | 2017 | 2018 |
| | Cohort | | | | | | 07-11- | 06-01- |
| RSV10 | Α | 1 | 19 | Leukocytosis | 5 | 120 | 2017 | 2018 |
| | Cohort | | | Decreased | | | 06-01- | Continu |
| RSV10 | Α | 1 | 20 | hemoglobin | 5 | 180 | 2018 | es |
| | Cohort | | | Pruritus | | | 18-07- | 23-07- |
| RSV13 | Α | 2 | 1 | vaccination site | 2 | 1 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 18-07- | 19-07- |
| RSV13 | Α | 2 | 2 | sensitivity | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 18-07- | 20-07- |
| RSV13 | Α | 2 | 3 | vaccination site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | | | | 24-07- | 08-09- |
| RSV13 | Α | 2 | 4 | Leukopenia | 5 | 7 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 27-07- | 10-08- |
| RSV13 | Α | 2 | 5 | abscess | 1 | 10 | 2017 | 2017 |
| | Cohort | | | | | | 25-07- | 25-07- |
| RSV13 | Α | 2 | 6 | Headache | 3 | 8 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 27-07- | 07-09- |
| RSV13 | Α | 2 | 7 | crust | 1 | 10 | 2017 | 2017 |
| | Cohort | | | | | | 30-07- | 30-07- |
| RSV13 | Α | 2 | 8 | Headache | 3 | 13 | 2017 | 2017 |
| | Cohort | | | | | | 10-08- | 10-08- |
| RSV13 | Α | 2 | 9 | Odynophagia | 4 | 24 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 24-07- | 26-07- |
| RSV13 | Α | 2 | 10 | site | 1 | 7 | 2017 | 2017 |
| | Cohort | | | | | | 24-08- | 24-08- |
| RSV13 | Α | 2 | 11 | Headache | 4 | 38 | 2017 | 2017 |
| | Cohort | _ | | | | | 26-08- | 26-08- |
| RSV13 | A | 2 | 12 | Headache | 4 | 40 | 2017 | 2017 |
| | Cohort | _ | | | | | 31-08- | 15-09- |
| RSV13 | A | 2 | 13 | Common cold | 4 | 45 | 2017 | 2017 |
| D01/40 | Cohort | | | | | 40 | 04-09- | 11-09- |
| RSV13 | A | 2 | 14 | Epistaxis | 4 | 49 | 2017 | 2017 |
| D0\/40 | Cohort | | 4.5 | Vaccination site | | | 10-09- | 20-09- |
| RSV13 | A | 2 | 15 | crust | 1 | 55 | 2017 | 2017 |
| D0\/40 | Cohort | | 40 | Vaccination site | | 60 | 23-09- | 18-11-<br>2017 |
| RSV13 | A | 2 | 16 | crust | 1 | 68 | 2017<br>13-09- | 15-09- |
| RSV13 | Cohort | 2 | 17 | Lagrain | 4 | F0 | 2017 | 2017 |
| KSVIS | A | | 17 | Leg pain | 4 | 58 | | |
| RSV13 | Cohort<br>A | 2 | 18 | Headache | 4 | 75 | 30-09-<br>2017 | 30-09-<br>2017 |
| K3V13 | Cohort | 2 | 10 | Tieauache | 4 | 7.5 | 06-10- | 06-10- |
| RSV13 | A | 2 | 19 | Headache | 4 | 81 | 2017 | 2017 |
| 110713 | Cohort | | 13 | i icauaciie | 4 | 01 | 10-11- | 10-11- |
| RSV13 | A | 2 | 20 | Headache | 4 | 116 | 2017 | 2017 |
| 110110 | Cohort | | 20 | i icaudoli <del>c</del> | 4 | 110 | 14-11- | Continu |
| RSV13 | A | 2 | 21 | Leukopenia | 5 | 120 | 2017 | es |
| 1.0 / 13 | Cohort | - | ۷۱ | Vaccination site | | 120 | 18-11- | 26-11- |
| RSV13 | A | 2 | 22 | crust | 1 | 124 | 2017 | 2017 |
| 110110 | Cohort | | | Vaccination site | | 127 | 26-11- | 12-12- |
| RSV13 | A | 2 | 23 | crust | 1 | 132 | 2017 | 2017 |
| | Cohort | | | | · | 102 | 24-11- | 24-11- |
| RSV13 | A | 2 | 24 | Headache | 4 | 130 | 2017 | 2017 |
| 1.51.0 | Cohort | - | <b>4</b> -7 | | 7 | 100 | 01-12- | 01-12- |
| RSV13 | A | 2 | 25 | Headache | 4 | 137 | 2017 | 2017 |
| | Cohort | | | | | | 07-12- | 07-12- |
| RSV13 | A | 2 | 26 | Headache | 4 | 143 | 2017 | 2017 |
| | Cohort | | | | | | 30-12- | 30-12- |
| RSV13 | A | 2 | 27 | Headache | 4 | 166 | 2017 | 2017 |
| | -1 | | | · <del></del> | | | | |

| RSV13 A | ĺ | Cohort | Ĭ | I | Hypophosphate | ĺ | l | 08-01- | Continu |
|---|---|---|---|---|---|---|---|---|---|
| RSV14 | RSV13 | | 2 | 28 | | 5 | 175 | | |
| RSV14 | | | _ | | | | | | |
| RSV14 | RSV14 | | 1 | 1 | | 1 | 1 | | |
| RSV14 | | | · | | | | • | | |
| RSV14 | RSV14 | | 1 | 2 | | 1 | 1 | | |
| RSV14 | 110111 | | | _ | Conclusion | · · | | | |
| RSV14 | RSV/14 | | 1 | 4 | Increase in CPK | 5 | 8 | | |
| RSV14 | 110111 | | | | | Ť | | | |
| Cohort | RSV/14 | | 1 | 5 | | 5 | 8 | | |
| RSV14 | 110114 | | | Ů | 0001 | | | 26-07- | 02-08- |
| Cohort | RSV/14 | | 1 | 6 | Leukonenia | 5 | 8 | 20-07- | |
| RSV14 | 110114 | | ' | 0 | | | | | |
| Cohort | DS\/1/ | | 1 | 7 | | 5 | 15 | | |
| RSV14 | 113714 | | ' | , | leitila | | 13 | | |
| Cohort | DS\/1/ | | 1 | Ω | Bronchitie | 1 | 16 | | |
| RSV14 | 113714 | | ' | 0 | | - | 10 | | |
| Cohort | DS\/1/ | | 1 | ۵ | | 1 | 15 | | |
| RSV14 | 113714 | | ' | 3 | | <u>'</u> | 13 | | |
| Cohort | DQ\/1/ | | 1 | 10 | | 1 | 16 | | |
| RSV14 | N3V14 | | ' | 10 | | <u>'</u> | 10 | | |
| RSV14 | DQ\/1/ | | 1 | 2 | | 2 | 4 | | |
| RSV14 | N3V14 | | ' | 3 | vaccination site | | 4 | | |
| Cohort C | DCV/44 | | 4 | 11 | Inorogo TTDA | _ | 20 | | |
| RSV14 | K5V14 | | <u> </u> | 11 | increase i i PA | 5 | 29 | | |
| RSV14 | DOVAA | | | 40 | 11 | _ | _ | | |
| RSV14 | K5V14 | | 1 | 12 | | 3 | | | 2017 |
| RSV14 | D0\/4.4 | | _ | 40 | | | , | - | |
| RSV14 | RSV14 | | 1 | 13 | sensitivity | 1 | 4 | 2017 | |
| RSV14 | DOVAA | | | 4.4 | 0 | _ | 20 | | |
| RSV14 | RSV14 | | 1 | 14 | Common cold | 4 | 38 | | |
| Cohort C | DO) /4.4 | | _ | 4.5 | D terri | ١, | 40 | | |
| RSV14 | RSV14 | | 1 | 15 | | 4 | 46 | | |
| RSV14 | D0) // / | | | 4.0 | | | 00 | | |
| RSV14 | RSV14 | | 1 | 16 | vaccination site | 2 | 29 | 2017 | |
| RSV14 | D0) // / | | | 4- | | _ | | 13-09- | |
| RSV14 | RSV14 | | 1 | 17 | Leukopenia | 5 | 5/ | 2017 | |
| Cohort A | 50111 | | | | | _ | | | |
| RSV14 | RSV14 | | 1 | 18 | Neutropenia | 5 | 5/ | | |
| Cohort C | 50111 | | | | l | _ | | | |
| RSV14 A | RSV14 | | 1 | 19 | Leukopenia | 5 | 181 | | |
| Cohort Sensitivity 1 | D0) // / | | | | | _ | 404 | | |
| RSV16 B | RSV14 | | 1 | 20 | | 5 | 181 | | |
| Cohort B | | | | | | | _ | | |
| RSV16 B | RSV16 | | 1 | 1 | | 1 | 0 | | |
| Pruritus Decreased Decre | | | | _ | | | _ | | |
| RSV16 B | RSV16 | | 1 | 2 | | 1 | 1 | | |
| Cohort Left axillary ymphadenopath Decreased | 50146 | | | | | | _ | 06-10- | |
| Name | KSV16 | В | 1 | 3 | | 2 | 4 | 201/ | 2017 |
| RSV16 B | | | | | | | | | |
| Cohort Left axillary ymphadenopath Decreased 10-10- Continu ESV16 B | 50111 | | | | Iymphadenopath | | _ | | |
| Name | RSV16 | В | 1 | 4 | У | 1 | 4 | 2017 | 2017 |
| RSV16 B 1 5 y 1 7 2017 2017 RSV16 B 1 6 haemoglobin 5 8 2017 es Cohort Vaccine site 14-10-20-10-20-10-20-10-10-10-10-10-10-10-10-10-10-10-10-10 | | | | | | | | | |
| Cohort B | | | | | | 1 | | | |
| RSV16 B 1 6 haemoglobin 5 8 2017 es RSV16 B 1 7 sensitivity 1 12 2017 2017 Cohort Vaccination site 14-10-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-01-04-04-01-04-01-04-04-04-04-04-04-04-04-04-04-04-04-04- | RSV16 | | 1 | 5 | , | 1 | 7 | | |
| Cohort Sensitivity 1 12 2017 2010- | | | | | | | | | |
| RSV16 B 1 7 sensitivity 1 12 2017 2017 RSV16 B 1 8 crust 1 12 2017 2018 Cohort Vaccination site 1 12 2017 2018 RSV16 B 1 9 abscess 1 13 2017 2017 Cohort Vaccination site 1 16 2017 2017 RSV16 B 1 10 abscess 1 16 2017 2017 Cohort Vaccination site 20-10- 20-10- 20-10- | RSV16 | | 1 | 6 | | 5 | 8 | | |
| Cohort RSV16 B | | | | | | 1 | | | |
| RSV16 B 1 8 crust 1 12 2017 2018 RSV16 B 1 9 abscess 1 13 2017 2017 Cohort Vaccination site 1 16 2017 2017 RSV16 B 1 10 abscess 1 16 2017 2017 Cohort Vaccination site 20-10- 20-10- | RSV16 | | 1 | 7 | | 1 | 12 | | |
| Cohort Vaccination site 15-10- 15-10- 15-10- | | | | | Vaccination site | | | | |
| RSV16 B 1 9 abscess 1 13 2017 2017 Cohort Vaccination site 18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10-18-10- | RSV16 | | 1 | 8 | | 1 | 12 | | |
| RSV16 B 1 10 abscess 1 16 2017 2017 Cohort Vaccination site b 20-10- 20-10- | | | _ | _ | | | | | |
| RSV16 B 1 10 abscess 1 16 2017 2017 Cohort Vaccination site 20-10- 20-10- | RSV16 | | 1 | 9 | | 1 | 13 | | |
| Cohort Vaccination site 20-10- 20-10- | | Cohort | | | | | | | |
| | RSV16 | | 1 | 10 | | 1 | 16 | | |
| RSV16 B 1 11 abscess 1 18 2017 2017 | | Cohort | | | | | | | |
| | RSV16 | В | 1 | 11 | abscess | 1 | 18 | 2017 | 2017 |

| ĺ | Cohort | | | Vaccination site | 1 | | 26-10- | 26-10- |
|---|---|---|---|---|---|---|---|---|
| RSV16 | В | 1 | 12 | abscess | 1 | 24 | 2017 | 2017 |
| | Cohort | | | Increase in | | | 31-10- | 11-12- |
| RSV16 | В | 1 | 13 | SGPT | 5 | 29 | 2017 | 2017 |
| | | | | Left axillary | | | | |
| | Cohort | | | lymphadenopath | | | 27-10- | 27-10- |
| RSV16 | В | 1 | 14 | у | 1 | 25 | 2017 | 2017 |
| 50146 | Cohort | | | | | | 18-01- | 20-01- |
| RSV16 | В | 1 | 15 | Common cold | 4 | 108 | 2018 | 2018 |
| | Cohort | | | Increase in | _ | | 02-04- | Continu |
| RSV16 | В | 1 | 16 | SGPT | 5 | 182 | 2018 | es |
| D0) /47 | Cohort | | _ | Erythema | | | 03-10- | 04-10- |
| RSV17 | В | 1 | 1 | vaccination site | 1 | 1 | 2017 | 2017 |
| D0)/47 | Cohort | | 0 | Vaccine site | | _ | 03-10- | 15-10- |
| RSV17 | В | 1 | 2 | sensitivity | 1 | 1 | 2017 | 2017 |
| DO) (47 | Cohort | | 0 | Induration | | _ | 03-10- | 06-10- |
| RSV17 | В | 1 | 3 | vaccination site | 1 | 1 | 2017 | 2017 |
| DC)/47 | Cohort | | | Pain vaccination | _ | | 03-10- | 15-10- |
| RSV17 | В | 1 | 4 | site | 1 | 1 | 2017 | 2017 |
| DC)/47 | Cohort | | 5 | Fatiana | 3 | 1 | 03-10-<br>2017 | 03-10- |
| RSV17 | B<br>Cohort | 1 | 5 | Fatigue | 3 | ı | 07-10- | 2017<br>08-10- |
| DC\/17 | B | 1 | 6 | Erythema vaccination site | 1 | 5 | 2017 | 2017 |
| RSV17 | Cohort | 1 | 0 | Decrease | | 5 | 10-10- | 16-10- |
| RSV17 | B | 1 | 7 | haemoglobin | 5 | 8 | 2017 | 2017 |
| KSVII | Cohort | ' | , | naemogiobin | J | 0 | 10-10- | 16-10- |
| RSV17 | В | 1 | 8 | Increase in CPK | 5 | 8 | 2017 | 2017 |
| KSVII | Cohort | 1 | 0 | Vaccination site | | 0 | 12-10- | 13-10- |
| RSV17 | В | 1 | 9 | abscess | 1 | 10 | 2017 | 2017 |
| 13717 | Cohort | | 9 | Vaccination site | <u> </u> | 10 | 13-10- | 20-10- |
| RSV17 | В | 1 | 10 | crust | 1 | 11 | 2017 | 2017 |
| 110117 | Cohort | | 10 | Vaccination site | | '' | 16-10- | 29-10- |
| RSV17 | В | 1 | 11 | abscess | 1 | 14 | 2017 | 2017 |
| 110117 | Cohort | | | Decrease | <u> </u> | 17 | 30-10- | 04-12- |
| RSV17 | В | 1 | 12 | haemoglobin | 5 | 28 | 2017 | 2017 |
| 110111 | Cohort | | | Hadmoglobin | | | 30-10- | 04-12- |
| RSV17 | В | 1 | 13 | Leukopenia | 5 | 28 | 2017 | 2017 |
| | Cohort | | | | | | 30-10- | 04-12- |
| RSV17 | В | 1 | 14 | Increase in CPK | 5 | 28 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 20-11- | 11-02- |
| RSV17 | В | 1 | 15 | crust | 1 | 49 | 2017 | 2018 |
| | Cohort | | | Vaccination site | | | 11-12- | 07-02- |
| RSV17 | В | 1 | 16 | abscess | 1 | 70 | 2017 | 2018 |
| | Cohort | | | Decreased | | | 31-01- | Continu |
| RSV17 | В | 1 | 17 | haemoglobin | 5 | 121 | 2018 | es |
| | Cohort | | | Vaccine site | | | 04-10- | 11-10- |
| RSV18 | В | 2 | 1 | sensitivity | 1 | 1 | 2017 | 2017 |
| l | Cohort | | | Erythema | | | 04-10- | 07-10- |
| RSV18 | В | 2 | 2 | vaccination site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Induration | | | 05-10- | 13-10- |
| RSV18 | В | 2 | 3 | vaccination site | 1 | 2 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 10-10- | 11-10- |
| RSV18 | В | 2 | 4 | site | 1 | 7 | 2017 | 2017 |
| D01/16 | Cohort | _ | _ | Vaccination site | | _ | 09-10- | 15-10- |
| RSV18 | В | 2 | 5 | abscess | 1 | 6 | 2017 | 2017 |
| D0) (46 | Cohort | | _ | District. | _ | _ | 10-10- | 11-10- |
| RSV18 | В | 2 | 6 | Diarrhea | 3 | 7 | 2017 | 2017 |
| D0)/40 | Cohort | | <del>_</del> | Hypercholestero | _ | _ | 12-10- | Continu |
| RSV18 | В | 2 | 7 | lemia | 5 | 9 | 2017 | es |
| DCV/40 | Cohort | | _ | Diarrhag | | 40 | 13-10- | 13-10- |
| RSV18 | B | 2 | 8 | Diarrhea | 3 | 10 | 2017 | 2017 |
| DCV/40 | Cohort | | _ | Diarrhag | | 40 | 16-10- | 16-10- |
| RSV18 | B | 2 | 9 | Diarrhea | 3 | 13 | 2017<br>14-10- | 2017 |
| DQ\/40 | Cohort | 2 | 10 | Vaccination site | | 4.4 | | 31-12- |
| RSV18 | В | 2 | 10 | crust | 1 | 11 | 2017 | 2017 |

| i | 1 0 1 1 1 | 1 1 | | l per en en en en en en | I 1 | İ | 1 40 40 | 1 40 40 |
|---|---|---|---|---|---|---|---|---|
| RSV18 | Cohort<br>B | 2 | 11 | Pain vaccination | 4 | 10 | 13-10-<br>2017 | 13-10-<br>2017 |
| K5V18 | _ | 2 | 11 | site | 1 | 10 | | |
| D0\/40 | Cohort | | 40 | Vaccine site | | 40 | 13-10- | 19-10- |
| RSV18 | В | 2 | 12 | sensitivity | 1 | 10 | 2017 | 2017 |
| D0\/40 | Cohort | | 40 | D'andres | _ | 0.5 | 28-10- | 28-10- |
| RSV18 | В | 2 | 13 | Diarrhea | 3 | 25 | 2017<br>31-10- | 2017 |
| DC)/40 | Cohort | | 4.4 | Diamela a a | _ | 20 | | 31-10- |
| RSV18 | B | 2 | 14 | Diarrhea | 3 | 28 | 2017<br>31-10- | 2017<br>15-11- |
| RSV18 | Cohort<br>B | 2 | 15 | Left thigh cellulitis | 4 | 28 | 2017 | 2017 |
| KSVIO | Cohort | 2 | 15 | Celiulius | 4 | 20 | 05-12- | 18-01- |
| RSV18 | В | 2 | 16 | Hyperglycemia | 5 | 63 | 2017 | 2018 |
| KSVIO | Cohort | 2 | 10 | Пурегујусенна | J | 03 | 01-01- | 01-01- |
| RSV18 | В | 2 | 17 | Headache | 4 | 90 | 2018 | 2018 |
| 13710 | Cohort | 2 | 17 | Decreased | 7 | 30 | 18-01- | 26-03- |
| RSV18 | В | 2 | 18 | haemoglobin | 5 | 107 | 2018 | 2018 |
| 1.0710 | Cohort | | 10 | Hacmoglobin | J | 107 | 18-01- | Continu |
| RSV18 | В | 2 | 19 | Increase in CPK | 5 | 107 | 2018 | es |
| 110110 | Cohort | | 10 | Vaccination site | Ŭ | 107 | 18-01- | 21-03- |
| RSV18 | В | 2 | 20 | crust | 1 | 107 | 2018 | 2018 |
| 110110 | Cohort | _ | | or dot | | 101 | 28-02- | 28-02- |
| RSV18 | В | 2 | 21 | Headache | 4 | 148 | 2018 | 2018 |
| | Cohort | _ | | Pain vaccination | | | 03-10- | 06-10- |
| RSV24 | В | 2 | 1 | site | 1 | 0 | 2017 | 2017 |
| | Cohort | _ | <u> </u> | Vaccine site | | | 03-10- | 06-10- |
| RSV24 | В | 2 | 2 | sensitivity | 1 | 0 | 2017 | 2017 |
| | Cohort | | | , | | | 03-10- | 03-10- |
| RSV24 | В | 2 | 3 | Headache | 3 | 0 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 04-10- | 10-10- |
| RSV24 | В | 2 | 4 | vaccination site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Induration | | | 04-10- | 08-10- |
| RSV24 | В | 2 | 5 | vaccination site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 08-10- | 08-10- |
| RSV24 | В | 2 | 6 | site | 1 | 5 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 08-10- | 18-10- |
| RSV24 | В | 2 | 7 | sensitivity | 1 | 5 | 2017 | 2017 |
| | Cohort | | | | | | 13-10- | 13-10- |
| RSV24 | В | 2 | 8 | Headache | 3 | 10 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 14-10- | 23-10- |
| RSV24 | В | 2 | 9 | abscess | 1 | 11 | 2017 | 2017 |
| DO: 40.4 | Cohort | | 40 | Pain vaccination | | | 11-10- | 17-10- |
| RSV24 | В | 2 | 10 | site | 1 | 8 | 2017 | 2017 |
| DOV (0.4 | Cohort | | 4.4 | Induration | | 40 | 13-10- | 13-10- |
| RSV24 | B | 2 | 11 | vaccination site | 1 | 10 | 2017<br>22-10- | 2017<br>22-10- |
| DCV/24 | Cohort | 2 | 12 | Llaadaaba | 3 | 10 | | |
| RSV24 | B<br>Cohort | 2 | 12 | Headache | ა | 19 | 2017<br>24-10- | 2017 |
| RSV24 | B | 2 | 13 | Headache | 3 | 21 | 24-10- | 24-10-<br>2017 |
| 110124 | Cohort | ۷ | 13 | Vaccination site | 3 | ۷۱ | 18-10- | 20-11- |
| RSV24 | B | 2 | 14 | crust | 1 | 15 | 2017 | 20-11- |
| 10024 | Cohort | 2 | 14 | Guat | 1 | 13 | 29-10- | 31-10- |
| RSV24 | В | 2 | 15 | Common cold | 4 | 26 | 2017 | 2017 |
| 1.072-7 | Cohort | | 10 | Vaccination site | | 20 | 25-10- | 26-10- |
| RSV24 | В | 2 | 16 | abscess | 1 | 22 | 2017 | 2017 |
| | Cohort | - | | Vaccination site | | | 29-10- | 29-10- |
| RSV24 | В | 2 | 17 | abscess | 1 | 26 | 2017 | 2017 |
| | Cohort | | | | | | 31-10- | 29-11- |
| RSV24 | В | 2 | 18 | Proteinuria | 5 | 28 | 2017 | 2017 |
| | Cohort | | | Muscle | | | 18-01- | 23-01- |
| RSV24 | В | 2 | 19 | contracture back | 4 | 107 | 2018 | 2018 |
| | Cohort | | | Pain vaccination | | | 05-10- | 05-10- |
| RSV25 | В | 1 | 1 | site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 05-10- | 05-10- |
| RSV25 | В | 1 | 2 | sensitivity | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 06-10- | 12-10- |
| RSV25 | В | 1 | 3 | vaccination site | 1 | 2 | 2017 | 2017 |

| ı | Laura | i | Ī | L. v | i | Ī | 1 00 40 | 1 44 40 |
|---|---|---|---|---|---|---|---|---|
| DO) (05 | Cohort | _ | | Vaccination site | _ | | 06-10- | 11-10- |
| RSV25 | В | 1 | 4 | abscess | 1 | 2 | 2017 | 2017 |
| 501/05 | Cohort | | _ | Induration | | | 07-10- | 11-10- |
| RSV25 | В | 1 | 5 | vaccination site | 1 | 3 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 08-10- | 27-11- |
| RSV25 | В | 1 | 6 | crust | 1 | 4 | 2017 | 2017 |
| | Cohort | | | Decreased | | | 11-10- | 04-12- |
| RSV25 | В | 1 | 7 | haemoglobin | 5 | 7 | 2017 | 2017 |
| | Cohort | | | Hypophosphate | | | 11-10- | 31-10- |
| RSV25 | В | 1 | 8 | mia | 5 | 7 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 18-10- | 18-10- |
| RSV25 | В | 1 | 9 | vaccination site | 1 | 14 | 2017 | 2017 |
| | Cohort | | | Induration | | | 18-10- | 18-11- |
| RSV25 | В | 1 | 10 | vaccination site | 1 | 14 | 2017 | 2017 |
| | Cohort | - | | Hypophosphate | | | 04-12- | 02-04- |
| RSV25 | В | 1 | 11 | mia | 5 | 61 | 2017 | 2018 |
| 110120 | Cohort | | | Decreased | | 0.1 | 22-01- | Continu |
| RSV25 | В | 1 | 12 | haemoglobin | 5 | 110 | 2018 | es |
| 110725 | Cohort | | 12 | Increase in | <u> </u> | 110 | 22-01- | 02-04- |
| RSV25 | В | 1 | 13 | SGPT | 5 | 110 | 2018 | 2018 |
| K3V23 | | 1 | 13 | | 3 | 110 | 04-10- | 07-10- |
| RSV26 | Cohort<br>B | , | 1 | Pain vaccination | | 0 | | |
| K5V26 | | 1 | 1 | site | 1 | 0 | 2017 | 2017 |
| 501100 | Cohort | | | Vaccine site | | | 04-10- | 08-10- |
| RSV26 | В | 1 | 2 | sensitivity | 1 | 0 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 05-10- | 20-10- |
| RSV26 | В | 1 | 3 | vaccination site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 10-10- | 17-10- |
| RSV26 | В | 1 | 4 | sensitivity | 1 | 6 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 11-10- | 15-10- |
| RSV26 | В | 1 | 5 | abscess | 1 | 7 | 2017 | 2017 |
| | Cohort | | | Decreased | | | 11-10- | 18-10- |
| RSV26 | В | 1 | 6 | haemoglobin | 5 | 7 | 2017 | 2017 |
| | Cohort | | | | | | 04-10- | 04-10- |
| RSV26 | В | 1 | 7 | Fatigue | 3 | 0 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 11-10- | 13-10- |
| RSV26 | В | 1 | 8 | site | 1 | 7 | 2017 | 2017 |
| | Cohort | | - | Pain vaccination | | | 15-10- | 15-10- |
| RSV26 | В | 1 | 9 | site | 1 | 11 | 2017 | 2017 |
| 110120 | Cohort | | | Ulcer | | - '' | 17-10- | 18-10- |
| RSV26 | В | 1 | 10 | vaccination site | 2 | 13 | 2017 | 2017 |
| 110720 | Cohort | ' | 10 | vaccination site | | 10 | 18-10- | 03-11- |
| RSV26 | В | 1 | 11 | Pyuria | 5 | 14 | 2017 | 2017 |
| N3V20 | Cohort | 1 | 11 | Vaccination site | J | 14 | 15-10- | 13-01- |
| DOVOC | | , | 40 | | | 44 | 2017 | |
| RSV26 | B | 1 | 12 | crust | 1 | 11 | | 2018<br>05-12- |
| DOV (00 | Cohort | | 40 | E | _ | 00 | 03-11- | |
| RSV26 | B | 11 | 13 | Eosinophilia | 5 | 30 | 2017 | 2017 |
| DOVOC | Cohort | _ | | Haadaak - | | | 29-11- | 29-11- |
| RSV26 | В | 1 | 14 | Headache | 4 | 56 | 2017 | 2017 |
| DO: (2.2 | Cohort | | | | | | 10-12- | 16-12- |
| RSV26 | В | 1 | 15 | Common cold | 4 | 67 | 2017 | 2017 |
| | Cohort | | _ | Hypercholestero | | | 26-01- | Continu |
| RSV26 | В | 1 | 16 | lemia | 5 | 114 | 2018 | es |
| | Cohort | | | Increase in | | | 26-01- | Continu |
| RSV26 | В | 1 | 17 | SGPT | 5 | 114 | 2018 | es |
| | Cohort | | | | | | 02-04- | Continu |
| RSV26 | В | 1 | 18 | Pyuria | 5 | 180 | 2018 | es |
| | Cohort | | | Increase in | | | 02-04- | Continu |
| RSV26 | В | 1 | 19 | SGOT | 5 | 180 | 2018 | es |
| | Cohort | | | Induration | | | 18-10- | 20-10- |
| RSV27 | В | 1 | 1 | vaccination site | 1 | 14 | 2017 | 2017 |
| | Cohort | | - | Erythema | | | 05-10- | 06-10- |
| RSV27 | В | 1 | 2 | vaccination site | 1 | 1 | 2017 | 2017 |
| | Cohort | · | _ | Induration | | | 05-10- | 10-10- |
| RSV27 | В | 1 | 3 | vaccination site | 1 | 1 | 2017 | 2017 |
| 1.0 121 | Cohort | <u>'</u> | | Pain vaccination | <u>'</u> | - ' | 04-10- | 17-10- |
| RSV27 | B | 1 | 4 | site | 1 | 0 | 2017 | 2017 |
| NOVZI | טן | | 4 | ગા <del>ડ</del> | | U | 2017 | 2017 |

| ı | 1011 | ı | Ī | l | ı | Ī | | 1 44 40 |
|---|---|---|---|---|---|---|---|---|
| DOV /0.7 | Cohort | | _ | Vaccine site | _ | | 04-10- | 14-10- |
| RSV27 | В | 1 | 5 | sensitivity | 1 | 0 | 2017 | 2017 |
| DO: (07 | Cohort | | 0 | Pruritus | | _ | 09-10- | 10-10- |
| RSV27 | В | 1 | 6 | vaccination site | 2 | 5 | 2017 | 2017 |
| DO: (07 | Cohort | | _ | Erythema | | _ | 09-10- | 21-10- |
| RSV27 | В | 1 | 7 | vaccination site | 1 | 5 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 12-10- | 18-10- |
| RSV27 | В | 1 | 8 | abscess | 1 | 8 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 18-10- | 09-03- |
| RSV27 | В | 1 | 9 | crust | 1 | 14 | 2017 | 2018 |
| | Cohort | | | Induration | | | 24-10- | 25-10- |
| RSV27 | В | 1 | 10 | vaccination site | 1 | 20 | 2017 | 2017 |
| | Cohort | | | | | | 06-12- | 26-01- |
| RSV27 | В | 1 | 11 | Hyperglycemia | 5 | 63 | 2017 | 2018 |
| | Cohort | | | | | | 25-01- | 25-01- |
| RSV27 | В | 1 | 12 | Headache | 4 | 113 | 2018 | 2018 |
| | Cohort | | | Decreased | | | 26-01- | 03-04- |
| RSV27 | В | 1 | 13 | haemoglobin | 5 | 114 | 2018 | 2018 |
| | Cohort | | | | | | 03-04- | Continu |
| RSV27 | В | 1 | 14 | Proteinuria | 5 | 181 | 2018 | es |
| | Cohort | | | Vaccine site | | | 10-10- | 12-10- |
| RSV30 | В | 1 | 1 | sensitivity | 1 | 0 | 2017 | 2017 |
| | Cohort | | | • | | | 10-10- | 18-10- |
| RSV30 | В | 1 | 2 | Headache | 3 | 0 | 2017 | 2017 |
| | Cohort | | | | | - | 11-10- | 11-10- |
| RSV30 | В | 1 | 3 | Fatigue | 3 | 1 | 2017 | 2017 |
| | Cohort | - | _ | Pruritus | | - | 11-10- | 13-10- |
| RSV30 | В | 1 | 4 | vaccination site | 2 | 1 | 2017 | 2017 |
| 110100 | Cohort | | | vaccination one | | | 12-10- | 12-10- |
| RSV30 | В | 1 | 5 | Hypertension | 3 | 2 | 2017 | 2017 |
| 110100 | Cohort | | | Пурсполого | | | 10-10- | 10-10- |
| RSV30 | B | 1 | 6 | Left axillary pain | 2 | 0 | 2017 | 2017 |
| 110700 | Cohort | | | Vaccination site | | | 21-10- | 26-10- |
| RSV30 | В | 1 | 7 | crust | 1 | 11 | 2017 | 2017 |
| 110730 | Cohort | ' | , | Pain vaccination | - | - '' | 18-10- | 22-10- |
| RSV30 | В | 1 | 8 | site | 1 | 8 | 2017 | 2017 |
| 110100 | Cohort | · | | Vaccine site | · | J | 17-10- | 23-10- |
| RSV30 | В | 1 | 9 | sensitivity | 1 | 7 | 2017 | 2017 |
| 110100 | Cohort | | Ū | COHOLIVILY | · | | 20-10- | 24-10- |
| RSV30 | В | 1 | 10 | Headache | 3 | 10 | 2017 | 2017 |
| 110100 | Cohort | | 10 | Ticadaciic | | 10 | 13-10- | 13-10- |
| RSV30 | B | 1 | 11 | Myalgia | 3 | 3 | 2017 | 2017 |
| 110700 | Cohort | | | Wydigia | | | 17-10- | 18-10- |
| RSV30 | В | 1 | 12 | Myalgia | 3 | 7 | 2017 | 2017 |
| 110730 | Cohort | ' | 12 | iviyaigia | | - | 22-10- | 22-10- |
| RSV30 | В | 1 | 13 | Myalgia | 3 | 12 | 2017 | 2017 |
| 110700 | Cohort | | 10 | Vaccination site | | 12 | 19-10- | 21-10- |
| RSV30 | В | 1 | 14 | abscess | 1 | 9 | 2017 | 2017 |
| 10000 | Cohort | <u>'</u> | 14 | u030033 | <del> </del> | 3 | 25-10- | 25-10- |
| RSV30 | В | 1 | 15 | Myalgia | 3 | 15 | 2017 | 2017 |
| 110 7 30 | Cohort | <u>'</u> | 13 | iviyaiyia | J | 13 | 27-10- | 27-10- |
| RSV30 | B | 1 | 16 | Myalgia | 3 | 17 | 2017 | 2017 |
| 110 7 30 | Cohort | <u>'</u> | 10 | iviyaiyia | J | 17 | 29-10- | 29-10- |
| RSV30 | B | 1 | 17 | Myalgia | 3 | 19 | 29-10- | 29-10- |
| 110730 | Cohort | <u> </u> | 17 | Pruritus | 3 | 19 | 27-10- | 30-10- |
| RSV30 | B | 1 | 18 | vaccination site | 2 | 17 | 27-10- | 2017 |
| 1/2/20 | | 1 | 10 | | | 17 | 02-11- | 14-11- |
| RSV30 | Cohort | 1 | 19 | Vaccination site | 1 | 23 | | 2017 |
| 1/2/20 | B | | 19 | crust | | ۷3 | 2017 | |
| D67/30 | Cohort | | 00 | Common selel | | 0.4 | 13-11- | 18-11- |
| RSV30 | B | 1 | 20 | Common cold | 4 | 34 | 2017 | 2017 |
| DG//20 | Cohort | | 21 | Common cold | | 105 | 12-02- | 18-02- |
| RSV30 | B | 1 | 21 | Common cold | 4 | 125 | 2018 | 2018 |
| D67/30 | Cohort | ا ہ | 00 | Decreased | - | 171 | 02-04- | Continu |
| RSV30 | B | 1 | 22 | haemoglobin | 5 | 174 | 2018 | es<br>or 40 |
| De//22 | Cohort | | | Pain vaccination | | _ | 21-11- | 05-12- |
| RSV32 | С | 1 | 1 | site | 1 | 0 | 2017 | 2017 |

| ī | 1011 | i i | | 1 | i | i | 1 00 44 | |
|---|---|---|---|---|---|---|---|---|
| D0) (00 | Cohort | | 0 | Vaccine site | _ | 4 | 22-11- | 06-12- |
| RSV32 | C | 1 | 2 | sensitivity | 1 | 1 | 2017 | 2017 |
| | Cohort | | _ | Erythema | | | 22-11- | 24-11- |
| RSV32 | C | 1 | 3 | vaccination site | 1 | 1 | 2017 | 2017 |
| 50,400 | Cohort | | | | | _ | 22-11- | 25-11- |
| RSV32 | С | 1 | 4 | Headache | 3 | 1 | 2017 | 2017 |
| | Cohort | | | | | | 22-11- | 24-11- |
| RSV32 | С | 1 | 5 | Fatigue | 3 | 1 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 22-11- | 22-11- |
| RSV32 | С | 1 | 6 | site | 4 | 1 | 2017 | 2017 |
| | Cohort | | | | | | 23-11- | 24-11- |
| RSV32 | С | 1 | 7 | Myalgia | 3 | 2 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 26-11- | 01-12- |
| RSV32 | С | 1 | 8 | vaccination site | 1 | 5 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 27-11- | 27-11- |
| RSV32 | С | 1 | 9 | abscess | 1 | 6 | 2017 | 2017 |
| | Cohort | | | Induration | | | 23-11- | 24-11- |
| RSV32 | С | 1 | 10 | vaccination site | 1 | 2 | 2017 | 2017 |
| | Cohort | | | Induration | | | 27-11- | 28-11- |
| RSV32 | С | 1 | 11 | vaccination site | 1 | 6 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 27-11- | 30-11- |
| RSV32 | С | 1 | 12 | crust | 1 | 6 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 30-11- | 18-12- |
| RSV32 | С | 1 | 13 | abscess | 1 | 9 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 03-12- | 03-12- |
| RSV32 | С | 1 | 14 | vaccination site | 1 | 12 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 05-12- | 05-12- |
| RSV32 | С | 1 | 15 | vaccination site | 1 | 14 | 2017 | 2017 |
| | Cohort | | | Induration | | | 30-11- | 30-11- |
| RSV32 | С | 1 | 16 | vaccination site | 1 | 9 | 2017 | 2017 |
| | Cohort | | | Induration | | | 03-12- | 29-12- |
| RSV32 | С | 1 | 17 | vaccination site | 1 | 12 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 02-12- | 17-06- |
| RSV32 | С | 1 | 18 | crust | 1 | 11 | 2017 | 2018 |
| | Cohort | | | Vaccination site | | | 01-12- | 05-12- |
| RSV32 | С | 1 | 19 | abscess | 1 | 10 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 10-12- | 10-12- |
| RSV32 | С | 1 | 20 | vaccination site | 1 | 19 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 07-12- | 16-12- |
| RSV32 | С | 1 | 21 | abscess | 1 | 16 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 11-12- | 13-12- |
| RSV32 | С | 1 | 22 | sensitivity | 1 | 20 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 19-12- | 03-03- |
| RSV32 | С | 1 | 23 | abscess | 1 | 28 | 2017 | 2018 |
| | Cohort | | | Acute | | | 24-12- | 26-12- |
| RSV32 | С | 1 | 24 | gastroenteritis | 4 | 33 | 2017 | 2017 |
| | Cohort | | | Decreased | | | 22-01- | 20-03- |
| RSV32 | С | 1 | 25 | haemoglobin | 5 | 62 | 2018 | 2018 |
| | Cohort | | | | | | 22-01- | 20-03- |
| RSV32 | С | 1 | 26 | Hypoglycemia | 5 | 62 | 2018 | 2018 |
| | Cohort | | | ,, <u></u> , | | | 22-01- | 20-03- |
| RSV32 | С | 1 | 27 | Hypertension | 4 | 62 | 2018 | 2018 |
| | Cohort | | | , | | | 19-04- | 22-04- |
| RSV32 | С | 1 | 28 | Common cold | 4 | 149 | 2018 | 2018 |
| | Cohort | | - | | | | 07-05- | 22-05- |
| RSV32 | С | 1 | 29 | Common cold | 4 | 167 | 2018 | 2018 |
| | Cohort | | | | | - | 14-05- | Continu |
| RSV32 | С | 1 | 30 | Hypoglycemia | 5 | 174 | 2018 | es |
| | Cohort | | | 71 - 3 7 | | | 14-05- | Continu |
| RSV32 | C | 1 | 31 | Hyponatremia | 5 | 174 | 2018 | es |
| . 10 102 | Cohort | <u>'</u> | - 01 | Pain vaccination | | 17-7 | 21-11- | 22-11- |
| RSV33 | Conort | 1 | 1 | site | 1 | 0 | 2017 | 2017 |
| 110 000 | Cohort | ' | I | Vaccine site | <u>'</u> | U | 21-11- | 23-11- |
| RSV33 | Conort | 1 | 2 | sensitivity | 1 | 0 | 2017 | 2017 |
| 110 000 | Cohort | ' | | Jonottvity | <u>'</u> | U | 21-11- | 21-11- |
| RSV33 | Conort | 1 | 3 | Fatigue | 3 | 0 | 2017 | 2017 |
| 110100 | _ U | 1 | <u> </u> | ı alıyu <del>c</del> | <u> </u> | U | 2017 | 2017 |

| i | 1011 | 1 1 | Ī | l = " | I | Ī | | 1 04 44 |
|---|---|---|---|---|---|---|---|---|
| RSV33 | Cohort | 1 | 4 | Erythema vaccination site | 1 | 2 | 23-11-<br>2017 | 24-11-<br>2017 |
| NOVOO | Cohort | 1 | 4 | Puncture site | <u>'</u> | | 26-11- | 03-12- |
| RSV33 | C | 1 | 5 | ecchymosis | 4 | 5 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 26-11- | 02-12- |
| RSV33 | С | 1 | 6 | sensitivity | 1 | 5 | 2017 | 2017 |
| | Cohort | | | • | | | 26-11- | 29-11- |
| RSV33 | С | 1 | 7 | Headache | 3 | 5 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 26-11- | 30-11- |
| RSV33 | С | 1 | 8 | abscess | 1 | 5 | 2017 | 2017 |
| DCVGG | Cohort | | 0 | \/a:ti-a | _ | 40 | 01-12- | 01-12- |
| RSV33 | C<br>Cohort | 1 | 9 | Vomiting | 3 | 10 | 2017<br>01-12- | 2017<br>01-12- |
| RSV33 | Conort | 1 | 10 | Diarrhea | 3 | 10 | 2017 | 2017 |
| 110 7 3 3 | Cohort | | 10 | Diamica | J | 10 | 01-12- | 02-12- |
| RSV33 | C | 1 | 11 | Headache | 3 | 10 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 28-11- | 04-12- |
| RSV33 | С | 1 | 12 | crust | 1 | 7 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 06-12- | 30-12- |
| RSV33 | С | 1 | 13 | crust | 1 | 15 | 2017 | 2017 |
| DO: (00 | Cohort | | | Pain vaccination | | | 24-11- | 24-11- |
| RSV33 | C | 1 | 14 | site | 1 | 3 | 2017 | 2017 |
| RSV33 | Cohort<br>C | 1 | 15 | Pain vaccination | 1 | 6 | 27-11-<br>2017 | 02-12-<br>2017 |
| RSV33 | Cohort | ' | 15 | site Pain vaccination | ı | | 05-12- | 05-12- |
| RSV33 | C | 1 | 16 | site | 1 | 14 | 2017 | 2017 |
| 110700 | Cohort | | 10 | ono | ' | | 06-12- | 20-12- |
| RSV33 | C | 1 | 17 | Hypokalemia | 5 | 15 | 2017 | 2017 |
| | Cohort | | | Erythema | - | - | 28-11- | 28-11- |
| RSV33 | С | 1 | 18 | vaccination site | 1 | 7 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 30-11- | 30-11- |
| RSV33 | С | 1 | 19 | vaccination site | 1 | 9 | 2017 | 2017 |
| 50,400 | Cohort | | | Induration | | _ | 28-11- | 28-11- |
| RSV33 | C | 1 | 20 | vaccination site | 1 | 7 | 2017 | 2017 |
| RSV33 | Cohort<br>C | 1 | 21 | Decreased hemoglobin | 5 | 29 | 20-12-<br>2017 | 24-01-<br>2018 |
| 113733 | Cohort | ' | 21 | Hemoglobin | J | 29 | 20-12- | 24-01- |
| RSV33 | C | 1 | 22 | Increase in CPK | 5 | 29 | 2017 | 2018 |
| 1.0100 | Cohort | | | Vaccination site | Ť | | 02-01- | 05-02- |
| RSV33 | С | 1 | 23 | crust | 1 | 42 | 2018 | 2018 |
| | Cohort | | | | | | 20-03- | 18-05- |
| RSV33 | С | 1 | 24 | Pyuria | 5 | 119 | 2018 | 2018 |
| DO: (00 | Cohort | | 0.5 | | | 450 | 23-04- | 07-05- |
| RSV33 | Cohort | 1 | 25 | Common cold | 4 | 153 | 2018<br>10-05- | 2018<br>25-05- |
| RSV33 | Cohort<br>C | 1 | 26 | Common cold | 4 | 170 | 2018 | 2018 |
| 110 7 3 3 | Cohort | | 20 | Pain vaccination | | 170 | 21-11- | 02-12- |
| RSV34 | C | 2 | 1 | site | 1 | 0 | 2017 | 2017 |
| | Cohort | | | Vaccine site | | | 22-11- | 26-11- |
| RSV34 | С | 2 | 2 | sensitivity | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 22-11- | 24-11- |
| RSV34 | С | 2 | 3 | vaccination site | 1 | 1 | 2017 | 2017 |
| 50101 | Cohort | | | Induration | | | 23-11- | 23-11- |
| RSV34 | C | 2 | 4 | vaccination site | 1 | 2 | 2017 | 2017 |
| RSV34 | Cohort<br>C | 2 | 5 | Pruritus<br>vaccination site | 2 | 3 | 24-11-<br>2017 | 26-11-<br>2017 |
| K3V34 | Cohort | 2 | 5 | vaccination site | | 3 | 27-11- | 04-12- |
| RSV34 | C | 2 | 6 | Headache | 3 | 6 | 2017 | 2017 |
| | Cohort | _ | | Decreased | Ť | | 28-11- | 06-12- |
| RSV34 | C | 2 | 7 | hemoglobin | 5 | 7 | 2017 | 2017 |
| | Cohort | | | Pruritus | | | 04-12- | 05-12- |
| RSV34 | С | 2 | 8 | vaccination site | 2 | 13 | 2017 | 2017 |
| 5015 | Cohort | | | | _ | | 06-12- | 21-12- |
| RSV34 | C | 2 | 9 | Proteinuria | 5 | 15 | 2017 | 2017 |
| DC\/0.4 | Cohort | | 40 | Increase in | _ | 4.5 | 06-12- | 21-12- |
| RSV34 | С | 2 | 10 | SGOT | 5 | 15 | 2017 | 2017 |

| Ì | | 1 1 | | i i | | i | 00.40 | I 00 40 |
|---|---|---|---|---|---|---|---|---|
| RSV34 | Cohort | 2 | 12 | Fatigue | 3 | 12 | 03-12-<br>2017 | 03-12-<br>2017 |
| K3V34 | Cohort | 2 | 12 | raligue | 3 | 12 | 04-12- | 07-12- |
| RSV34 | Conort | 2 | 13 | Myalgia | 3 | 13 | 2017 | 2017 |
| 110 7 34 | Cohort | | 13 | iviyaigia | 3 | 13 | 10-12- | 13-12- |
| RSV34 | C | 2 | 14 | Sickness | 3 | 19 | 2017 | 2017 |
| 110134 | Cohort | | | Olokiicaa | | 10 | 06-12- | 08-12- |
| RSV34 | C | 2 | 15 | Headache | 3 | 15 | 2017 | 2017 |
| 110134 | Cohort | | 10 | Vaccination site | | 10 | 04-12- | 04-12- |
| RSV34 | C | 2 | 16 | abscess | 1 | 13 | 2017 | 2017 |
| | Cohort | _ | | Vaccination site | | | 21-12- | 20-02- |
| RSV34 | С | 2 | 17 | abscess | 1 | 30 | 2017 | 2018 |
| | Cohort | | | Hypophosphate | | | 21-12- | 18-01- |
| RSV34 | С | 2 | 18 | mia | 5 | 30 | 2017 | 2018 |
| | Cohort | | | Decreased | | | 21-12- | 18-01- |
| RSV34 | С | 2 | 19 | hemoglobin | 5 | 30 | 2017 | 2018 |
| | Cohort | | | | | | 21-12- | 18-01- |
| RSV34 | С | 2 | 20 | Eosinophilia | 5 | 30 | 2017 | 2018 |
| | Cohort | | | Hyperbilirubine | | | 18-01- | 20-03- |
| RSV34 | С | 2 | 21 | mia | 5 | 58 | 2018 | 2018 |
| | Cohort | | | | | | 18-01- | 20-03- |
| RSV34 | С | 2 | 22 | Hypoglycemia | 5 | 58 | 2018 | 2018 |
| | Cohort | | | Pain vaccination | | | 15-02- | 20-02- |
| RSV34 | С | 2 | 23 | site | 1 | 86 | 2018 | 2018 |
| 501/0/ | Cohort | | | Pruritus | | | 15-02- | 26-02- |
| RSV34 | C | 2 | 24 | vaccination site | 2 | 86 | 2018 | 2018 |
| DO: (0.4 | Cohort | | 0.5 | Vaccination site | | 0.4 | 20-02- | 23-04- |
| RSV34 | C | 2 | 25 | crust | 1 | 91 | 2018 | 2018 |
| DC)/24 | Cohort | | 00 | l la a da aba | 4 | 00 | 27-02- | 27-02- |
| RSV34 | Cohort | 2 | 26 | Headache | 4 | 98 | 2018<br>20-03- | 2018<br>23-05- |
| RSV34 | Cohort<br>C | 2 | 27 | Eosinophilia | 5 | 119 | 20-03- | 2018 |
| 13734 | Cohort | 2 | 21 | Thrombocytope | J | 119 | 20-03- | 23-05- |
| RSV34 | Conort | 2 | 28 | nia | 5 | 119 | 20-03- | 2018 |
| 110134 | Cohort | | | IIIG | | 113 | 06-12- | 21-12- |
| RSV34 | C | 2 | 29 | increase in CPK | 5 | 15 | 2017 | 2017 |
| | Cohort | _ | | Vaccine site | | | 27-11- | 20-01- |
| RSV36 | C | 1 | 1 | sensitivity | 1 | 0 | 2017 | 2018 |
| | Cohort | | | | | | 27-11- | 27-11- |
| RSV36 | С | 1 | 2 | Headache | 3 | 0 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 28-11- | 05-12- |
| RSV36 | С | 1 | 3 | vaccination site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 28-11- | 08-12- |
| RSV36 | С | 1 | 4 | site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 01-12- | 05-12- |
| RSV36 | С | 1 | 5 | abscess | 1 | 4 | 2017 | 2017 |
| DC: /02 | Cohort | | _ | E.C. | _ | | 01-12- | 01-12- |
| RSV36 | C | 1 | 6 | Fatigue | 3 | 4 | 2017 | 2017 |
| DC) /22 | Cohort | | - | Vaccination site | | -, | 04-12- | 14-12- |
| RSV36 | Cohort | 1 | 7 | crust | 1 | 7 | 2017 | 2017<br>02-01- |
| RSV36 | Cohort | 1 | 8 | Decreased | 5 | 8 | 05-12-<br>2017 | 02-01-<br>2018 |
| 13730 | Cohort | 1 | 0 | haemoglobin | ິນ | Ö | 05-12- | 11-12- |
| RSV36 | Conort | 1 | 9 | Increase in CPK | 5 | 8 | 2017 | 2017 |
| 110 7 30 | Cohort | <del> </del> | <u> </u> | Ulcer | J | J | 15-12- | 28-12- |
| RSV36 | C | 1 | 10 | vaccination site | 2 | 18 | 2017 | 2017 |
| | Cohort | <del> </del> | | . 300 | _ | | 01-01- | 01-01- |
| RSV36 | C | 1 | 11 | Urethritis | 4 | 35 | 2018 | 2018 |
| - | Cohort | | | | | | 02-01- | 25-01- |
| RSV36 | C | 1 | 12 | Increase in CPK | 5 | 36 | 2018 | 2018 |
| | Cohort | | | Vaccination site | | | 29-12- | 30-01- |
| RSV36 | С | 1 | 13 | crust | 1 | 32 | 2017 | 2018 |
| | Cohort | | | | | | 25-01- | 27-03- |
| RSV36 | С | 1 | 14 | Pyuria | 5 | 59 | 2018 | 2018 |
| | Cohort | | | Decreased | | | 25-01- | Continu |
| RSV36 | С | 1 | 15 | haemoglobin | 5 | 59 | 2018 | es |

| l | Cohort | | | Increase in | 1 | | 25-01- | 27-03- |
|---|---|---|---|---|---|---|---|---|
| RSV36 | С | 1 | 16 | SGOT | 5 | 59 | 2018 | 2018 |
| | Cohort | | | Increase in | | | 25-01- | 27-03- |
| RSV36 | С | 1 | 17 | SGPT | 5 | 59 | 2018 | 2018 |
| | Cohort | | | | | | 27-03- | 28-05- |
| RSV36 | С | 1 | 18 | Hypokalemia | 5 | 120 | 2018 | 2018 |
| | Cohort | | | | | | 27-11- | 27-11- |
| RSV38 | С | 2 | 1 | Hypotension | 3 | 0 | 2017 | 2017 |
| | Cohort | _ | _ | Vaccine site | | _ | 27-11- | 01-12- |
| RSV38 | C | 2 | 2 | sensitivity | 1 | 0 | 2017 | 2017 |
| D0) (00 | Cohort | | | Pain vaccination | _ | | 27-11- | 30-11- |
| RSV38 | Cohort | 2 | 3 | Site | 1 | 0 | 2017 | 2017 |
| RSV38 | Cohort<br>C | 2 | 4 | Erythema vaccination site | 1 | 1 | 28-11-<br>2017 | 29-11-<br>2017 |
| 13730 | Cohort | | 4 | Pruritus | ı | | 29-11- | 02-12- |
| RSV38 | C | 2 | 5 | vaccination site | 2 | 2 | 2017 | 2017 |
| 110730 | Cohort | | | Vaccine site | | | 03-12- | 04-01- |
| RSV38 | C | 2 | 6 | sensitivity | 1 | 6 | 2017 | 2018 |
| | Cohort | _ | - | Traumatic | | | 02-12- | 09-01- |
| RSV38 | C | 2 | 7 | wound, left foot | 4 | 5 | 2017 | 2018 |
| | Cohort | | | Decreased | | | 05-12- | 11-12- |
| RSV38 | С | 2 | 8 | haemoglobin | 5 | 8 | 2017 | 2017 |
| | | | | Increase in | | | | |
| | Cohort | | | alkaline | | | 05-12- | Continu |
| RSV38 | С | 2 | 9 | phosphatases | 5 | 8 | 2017 | es |
| | Cohort | | | Pain vaccination | | | 05-12- | 21-12- |
| RSV38 | С | 2 | 10 | site | 1 | 8 | 2017 | 2017 |
| 50,400 | Cohort | | | Pruritus | | | 06-12- | 08-12- |
| RSV38 | С | 2 | 11 | vaccination site | 2 | 9 | 2017 | 2017 |
| DCV/20 | Cohort | 0 | 40 | 0 | , | 44 | 08-12- | 22-12- |
| RSV38 | Cohort | 2 | 12 | Common cold Vaccination site | 4 | 11 | 2017<br>05-12- | 2017<br>07-12- |
| RSV38 | Conort | 2 | 13 | abscess | 1 | 8 | 2017 | 2017 |
| 13730 | Cohort | | 13 | Vaccination site | | 0 | 08-12- | 26-12- |
| RSV38 | C | 2 | 14 | crust | 1 | 11 | 2017 | 20-12- |
| 110700 | Cohort | _ | | Vaccination site | | | 09-12- | 10-12- |
| RSV38 | C | 2 | 15 | abscess | 1 | 12 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 14-12- | 14-12- |
| RSV38 | С | 2 | 16 | abscess | 1 | 17 | 2017 | 2017 |
| | Cohort | | | | | | 15-12- | 15-12- |
| RSV38 | С | 2 | 17 | Headache | 3 | 18 | 2017 | 2017 |
| | Cohort | | | | | | 15-12- | 15-12- |
| RSV38 | С | 2 | 18 | Fatigue | 3 | 18 | 2017 | 2017 |
| | Cohort | _ | | Ulcer | _ | | 27-12- | 05-01- |
| RSV38 | С | 2 | 19 | vaccination site | 2 | 30 | 2017 | 2018 |
| DO: (00 | Cohort | | | | | 00 | 23-12- | 23-12- |
| RSV38 | Cobord | 2 | 20 | Headache | 3 | 26 | 2017 | 2017 |
| RSV38 | Cohort<br>C | 2 | 21 | Diarrhea | 3 | 25 | 22-12-<br>2017 | 22-12-<br>2017 |
| K3V30 | Cohort | 2 | 21 | Vaccination site | 3 | 25 | 05-01- | 21-01- |
| RSV38 | Conort | 2 | 22 | crust | 1 | 39 | 2018 | 2018 |
| 13730 | Cohort | | 22 | Crust | | 39 | 13-12- | 13-12- |
| RSV38 | C | 2 | 23 | Headache | 3 | 16 | 2017 | 2017 |
| 110 700 | Cohort | | 20 | Ticadaciic | | 10 | 20-12- | 20-12- |
| RSV38 | C | 2 | 24 | Headache | 3 | 23 | 2017 | 2017 |
| | Cohort | | | | | | 07-05- | 07-05- |
| RSV38 | C | 2 | 25 | Headache | 4 | 161 | 2018 | 2018 |
| | Cohort | | | | | | 28-05- | 28-05- |
| RSV38 | С | 2 | 26 | Headache | 4 | 182 | 2018 | 2018 |
| | Cohort | | | Vaccine site | | | 28-11- | 16-12- |
| RSV40 | С | 1 | 1 | sensitivity | 1 | 0 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 04-12- | 08-12- |
| RSV40 | С | 1 | 2 | site | 1 | 6 | 2017 | 2017 |
| D0\//2 | Cohort | | _ | Erythema | | _ | 04-12- | 07-12- |
| RSV40 | С | 1 | 3 | vaccination site | 1 | 6 | 2017 | 2017 |

| | Cohort | ĺ | | Induration | ĺ | | 06-12- | 06-12- |
|---|---|---|---|---|---|---|---|---|
| RSV40 | С | 1 | 4 | vaccination site | 1 | 8 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 04-12- | 31-12- |
| RSV40 | С | 1 | 5 | abscess | 1 | 6 | 2017 | 2017 |
| DC)/40 | Cohort | | | Vaccination site | | 7 | 05-12- | 31-12- |
| RSV40 | C<br>Cohort | 1 | 6 | crust | 1 | 7 | 2017<br>06-12- | 2017<br>09-12- |
| RSV40 | Conort | 1 | 7 | Increase in CPK | 5 | 8 | 2017 | 2017 |
| 110140 | Cohort | | , | Decreased | 3 | | 09-12- | 30-01- |
| RSV40 | C | 1 | 8 | haemoglobin | 5 | 11 | 2017 | 2018 |
| | Cohort | | | Pain vaccination | | | 12-12- | 17-12- |
| RSV40 | С | 1 | 9 | site | 1 | 14 | 2017 | 2017 |
| | Cohort | | | | | | 13-12- | 16-12- |
| RSV40 | C | 1 | 10 | Tonsillitis | 4 | 15 | 2017 | 2017 |
| DCV/40 | Cohort | 4 | 11 | Contusion right | , | 10 | 16-12- | 18-12- |
| RSV40 | C Cohort | 1 | 11 | hand<br>Erythema | 4 | 18 | 2017<br>24-12- | 2017 |
| RSV40 | Conort | 1 | 13 | vaccination site | 1 | 26 | 2017 | 24-12- |
| 110140 | Cohort | | 10 | Ulcer | | 20 | 01-01- | 15-01- |
| RSV40 | C | 1 | 14 | vaccination site | 2 | 34 | 2018 | 2018 |
| | Cohort | | | | | | 10-12- | 10-12- |
| RSV40 | С | 1 | 15 | Malaise | 3 | 12 | 2017 | 2017 |
| | Cohort | | | | | | 27-12- | 27-12- |
| RSV40 | С | 1 | 16 | Diarrhea | 3 | 29 | 2017 | 2017 |
| D0\/40 | Cohort | | 47 | D'andra | | 0.4 | 29-12- | 30-12- |
| RSV40 | Cabant | 1 | 17 | Diarrhea | 4 | 31 | 2017 | 2017<br>10-12- |
| RSV40 | Cohort<br>C | 1 | 18 | Hoodoobo | 3 | 12 | 10-12-<br>2017 | 2017 |
| K3V40 | Cohort | <u>'</u> | 10 | Headache | 3 | 12 | 26-12- | 27-12- |
| RSV40 | C | 1 | 19 | Myalgia | 3 | 28 | 2017 | 2017 |
| 110110 | Cohort | | | , | | | 02-01- | 02-01- |
| RSV40 | С | 1 | 20 | Diarrhea | 4 | 35 | 2018 | 2018 |
| | Cohort | | | | | | 30-12- | 30-12- |
| RSV40 | С | 1 | 21 | Sickness | 4 | 32 | 2017 | 2017 |
| D0\/40 | Cohort | | 00 | 0 | | 00 | 27-12- | 15-01- |
| RSV40 | C Cohort | 1 | 22 | Common cold | 4 | 29 | 2017<br>03-01- | 2018<br>30-01- |
| RSV40 | Conort | 1 | 23 | Increase in CPK | 5 | 36 | 2018 | 2018 |
| 110140 | Cohort | | 25 | mercase in or it | 3 | | 01-02- | 08-02- |
| RSV40 | C | 1 | 24 | Diarrhea | 4 | 65 | 2018 | 2018 |
| | Cohort | | | | | | 01-03- | 14-04- |
| RSV40 | С | 1 | 26 | Anxiety | 4 | 93 | 2018 | 2018 |
| | Cohort | | | | | | 16-05- | 16-05- |
| RSV40 | C | 1 | 27 | Insomnia | 4 | 169 | 2018 | 2018 |
| DC)/44 | Cohort | | | Vaccine site | | 0 | 28-11- | 09-12- |
| RSV41 | C<br>Cohort | 1 | 1 | sensitivity | 1 | 0 | 2017<br>29-11- | 2017 |
| RSV41 | Conort | 1 | 2 | Pain vaccination site | 1 | 1 | 2017 | 30-11-<br>2017 |
| 110141 | Cohort | | | Vaccination site | | | 30-11- | 02-12- |
| RSV41 | C | 1 | 3 | abscess | 1 | 2 | 2017 | 2017 |
| | Cohort | | | Induration | | | 01-12- | 01-12- |
| RSV41 | С | 1 | 4 | vaccination site | 1 | 3 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 04-12- | 05-12- |
| RSV41 | C | 1 | 5 | abscess | 1 | 6 | 2017 | 2017 |
| DC\/44 | Cohort | | _ | Pain vaccination | _ | _ | 05-12- | 07-12- |
| RSV41 | C Cohort | 1 | 6 | site Vaccination site | 1 | 7 | 2017<br>03-12- | 2017<br>03-12- |
| RSV41 | Conort | 1 | 7 | crust | 1 | 5 | 2017 | 2017 |
| 1,0 4 7 1 | Cohort | <u>'</u> | · · · · · · | Decreased | ' | | 06-12- | Continu |
| RSV41 | C | 1 | 8 | haemoglobin | 5 | 8 | 2017 | es |
| | Cohort | | | Erythema | _ | | 06-12- | 06-12- |
| RSV41 | С | 1 | 9 | vaccination site | 1 | 8 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 06-12- | 22-12- |
| RSV41 | C | 11 | 10 | crust | 1 | 8 | 2017 | 2017 |
| DC\/44 | Cohort | _ | 4.4 | Urticorio | | 40 | 10-12- | 10-12- |
| RSV41 | С | 1 | 11 | Urticaria | 4 | 12 | 2017 | 2017 |

| | | | | 1 | i | • | | |
|---|---|---|---|---|---|---|---|---|
| 501/44 | Cohort | | 40 | | | 00 | 18-12- | 19-12- |
| RSV41 | С | 1 | 12 | Headache | 3 | 20 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 18-12- | 20-12- |
| RSV41 | С | 1 | 13 | abscess | 1 | 20 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 24-12- | 08-02- |
| RSV41 | С | 1 | 14 | crust | 1 | 26 | 2017 | 2018 |
| | Cohort | | | Vaccine site | | | 23-12- | 25-12- |
| RSV41 | С | 1 | 15 | sensitivity | 1 | 25 | 2017 | 2017 |
| | Cohort | | | Pain vaccination | | | 23-12- | 24-12- |
| RSV41 | С | 1 | 16 | site | 1 | 25 | 2017 | 2017 |
| | Cohort | | | | | | 12-01- | 29-01- |
| RSV41 | С | 1 | 17 | Common cold | 4 | 45 | 2018 | 2018 |
| | Cohort | | | | | | 16-01- | 18-01- |
| RSV41 | С | 1 | 18 | Myalgia | 4 | 49 | 2018 | 2018 |
| | Cohort | | | Increase in | | | 23-01- | 02-04- |
| RSV41 | С | 1 | 19 | SGOT | 5 | 56 | 2018 | 2018 |
| | Cohort | | | | | | 23-01- | 02-04- |
| RSV41 | С | 1 | 20 | Increase in CPK | 5 | 56 | 2018 | 2018 |
| | Cohort | | | | | | 29-01- | 08-02- |
| RSV41 | C | 1 | 21 | Tonsillitis | 4 | 62 | 2018 | 2018 |
| | Cohort | 1 | | 10110111110 | | | 08-02- | 07-03- |
| RSV41 | C | 1 | 22 | Common cold | 4 | 72 | 2018 | 2018 |
| 110111 | Cohort | | | Vaccination site | | | 11-02- | 10-06- |
| RSV41 | C | 1 | 23 | crust | 1 | 75 | 2018 | 2018 |
| 110141 | Cohort | ' | | Crust | <u> </u> | 7.5 | 02-04- | 28-05- |
| RSV41 | Conort | 1 1 | 24 | Hyperglycemia | 5 | 125 | 2018 | 2018 |
| 13741 | Cohort | <u>'</u> | 24 | ттуретутусенна | J | 123 | 02-04- | 28-05- |
| RSV41 | | | 25 | I ly man atranaia | _ | 105 | | |
| R5V41 | Cabant | 1 | 25 | Hypernatremia | 5 | 125 | 2018 | 2018<br>12-05- |
| DC)/44 | Cohort | | 00 | Dua malaitia | | 450 | 27-04- | |
| RSV41 | C | 1 | 26 | Bronchitis | 4 | 150 | 2018 | 2018 |
| DO) (40 | Cohort | | | Vaccine site | _ | | 04-12- | 17-12- |
| RSV42 | С | 1 | 1 | sensitivity | 1 | 0 | 2017 | 2017 |
| 501110 | Cohort | | | Pain vaccination | | _ | 05-12- | 10-12- |
| RSV42 | С | 1 | 2 | site | 1 | 1 | 2017 | 2017 |
| 501110 | Cohort | | _ | Erythema | | _ | 05-12- | 06-12- |
| RSV42 | С | 1 | 3 | vaccination site | 1 | 1 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | _ | 06-12- | 11-12- |
| RSV42 | С | 1 | 4 | abscess | 1 | 2 | 2017 | 2017 |
| | Cohort | | | General | | | 05-12- | 06-12- |
| RSV42 | С | 1 | 5 | discomfort | 4 | 1 | 2017 | 2017 |
| | | | | Left axillary | | | | |
| | Cohort | | | lymphadenopath | | | 07-12- | 13-12- |
| RSV42 | С | 1 | 6 | у | 1 | 3 | 2017 | 2017 |
| | Cohort | | | | | | 06-12- | 06-12- |
| RSV42 | С | 1 | 7 | Headache | 3 | 2 | 2017 | 2017 |
| | Cohort | | | Erythema | | | 09-12- | 12-12- |
| RSV42 | С | 1 | 8 | vaccination site | 1 | 5 | 2017 | 2017 |
| | Cohort | | | | | | 05-12- | 05-12- |
| RSV42 | С | 1 | 9 | Hypotension | 3 | 1 | 2017 | 2017 |
| 1 | Cohort | | | | | | 11-12- | 18-12- |
| RSV42 | С | 1 | 10 | Pyuria | 5 | 7 | 2017 | 2017 |
| 1 | Cohort | Ι Τ | | Vaccination site | | | 15-12- | 15-12- |
| RSV42 | С | 1 | 11 | abscess | 1 | 11 | 2017 | 2017 |
| | Cohort | | | Vaccination site | | | 11-12- | 23-03- |
| RSV42 | С | 1 | 12 | crust | 1 | 7 | 2017 | 2018 |
| | Cohort | | | | | | 29-12- | 03-01- |
| RSV42 | С | 1 | 13 | Pyuria | 5 | 25 | 2017 | 2018 |
| | Cohort | | | | | | 29-12- | 03-01- |
| RSV42 | С | 1 | 14 | Hematuria | 5 | 25 | 2017 | 2018 |
| | Cohort | | | Decreased | | | 29-12- | 05-04- |
| RSV42 | С | 1 | 15 | hemoglobin | 5 | 25 | 2017 | 2018 |
| | Cohort | 1 | | - | | | 03-01- | 07-02- |
| RSV42 | С | 1 | 16 | Proteinuria | 5 | 30 | 2018 | 2018 |
| | | 1 | | Precordial pain | | | | 1 |
| | | | | secondary to | | | | 1 |
| 1 | Cohort | | | supraventricular | | | 24-01- | 26-01- |
| RSV42 | С | 1 | 17 | tachycardia | 4 | 51 | 2018 | 2018 |



16 September 2019

#### 16. REFERENCE LIST

- 1. Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, et al. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. (2010) May 1;375(9725):1545-1555. doi: 10.1016/S0140-6736(10)60206-1. PubMed PMID: WOS:000277655100027; English.
- Collins PL, Melero JA. Progress in understanding and controlling respiratory syncytial virus: still crazy after all these years. Virus Res. (2011) Dec;162(1-2):80-99. doi: 10.1016/j.virusres.2011.09.020. PubMed PMID: 21963675; PubMed Central PMCID: PMC3221877.
- 3. Hall CB. The burgeoning burden of respiratory syncytial virus among children. Infect Disord Drug Targets. (2012);12(92-97).
- 4. Huang K, Incognito L, Cheng X, Ulbrandt ND, Wu H. Respiratory syncytial virus-neutralizing monoclonal antibodies motavizumab and palivizumab inhibit fusion. J Virol (2010);84(16):8132-40.
- 5. Kim HW, Canchola JG, Brandt CD. Respiratory syncytial virus disease in infants despite prior administration of antigenic inactivated vaccine. Am J Epidemiol (1969);89(4):422-34.
- 6. Kim HW, Canchola JG, Brandt CD, Pyles G, Chanock RM, Jensen K, et al. Respiratory syncytial virus disease in infants despite prior administration of antigenic inactivated vaccine. Am J Epidemiol (1969);89(4):422-34.
- 7. Kruijsen D, Schijf MA, Lukens MV, Uden NOv, Kimpen JL, Coenjaerts FE, et al. Local innate and adaptive immune responses regulate inflammatory cell influx into the lungs after vaccination with formalin inactivated RSV. Vaccine. (2011);29(15):2730-41.
- 8. Bendelja K, Gagro A, Bace A, Lokar-Kolbas R, Krsulovic-Hresic V, Drazenovic V, et al. Predominant type-2 response in infants with respiratory syncytial virus (RSV) infection demonstrated by cytokine flow cytometry. Clin Exp Immunol (2000);121(2):332-8.
- 9. AOYAGI M, SHIMOJO N, SEKINE K, NISHIMUTA T, KOHNO Y. Respiratory syncytial virus infection suppresses IFN-γ production of γδ T cells. Clin Exp Immunol (2003);131(2):312–317.

- 10. PATH. Respiratory syncytial virus. Vaccine development against a major cause of childhood respiratory illness. <a href="http://sites.path.org/vaccinedevelopment/respiratory-syncytial-virus-rsv">http://sites.path.org/vaccinedevelopment/respiratory-syncytial-virus-rsv</a>. Accesed 17 Febreary 2017. (2016.).
- 11. Bueno SM, Gonzalez PA, Cautivo KM, Mora JE, Leiva ED, Tobar HE. Protective T cell immunity against respiratory syncytial virus is efficiently induced by recombinant BCG Proc Natl Acad Sci USA. (2008);105(52):20822-7.
- 12. Abubakar I, Pimpin L, Ariti C, Beynon R, Mangtani P, Sterne JA, et al. Systematic review and meta-analysis of the current evidence on the duration of protection by bacillus Calmette-Guérin vaccination against tuberculosis. Health Technol Assess. (2013);17(37):1-372.
- 13. Marchant A, Goetghebuer T, Ota MO, Wolfe I, Ceesay SJ, De Groote D, et al. Newborns develop a Th1-type immune response to Mycobacterium bovis bacillus Calmette-Guerin vaccination. J Immunol. (1999);163(4):2249–55.
- 14. Cautivo KM, Bueno SM, Cortes CM, Wozniak A, Riedel CA, Kalergis AM. Efficient lung recruitment of respiratory syncytial virusspecific Th1 cells induced by recombinant bacillus Calmette-Guerin promotes virus clearance and protects from infection J Immunol. (2010);185(12):7633-45.
- 15. Céspedes PC, Rey-Jurado E, Espinoza JA, Rivera CA, Canedo-Marroquín G, Bueno SM, et al. A single, low dose of a cGMP recombinant BCG vaccine elicits protective T cell immunity against the human respiratory syncytial virus infection and prevents lung pathology in mice. Vaccine. (2016).
- 16. Soto JA, Galvez NMS, Rivera CA, Palavecino CE, Céspedes PF, Rey-Jurado E, et al. Recombinant BCG induces protective cellular and humoral immunity reducing the lung pathology caused by respiratory viruses.
- 17. Declaración de Helsinki de la Asociación Médica Mundial: Recomendaciones para guiar a los médicos en la investigación biomédica con seres humanos, adoptada por la 18ª Asamblea Médica Mundial (Helsinki, junio 1964) y enmendada por la 29ª Asamblea Médica Mundial (Tokio, octubre 1975), a la 35ª Asamblea Médica Mundial (Venecia, octubre 1983), la 41ª Asamblea Médica Mundial (Hong Kong, septiembre 1989) y la 52ª Asamblea General (Edimburgo, octubre 2000).

- 18. Maecker HT. Multiparameter Flow Cytometry Monitoring of T Cell Responses. , . Vol. vol 485. Humana Press. 2009. (In: Prasad V.R. KGVe, editor. HIV Protocols. Methods In Molecular Biology<sup>TM</sup>).
- 19. Chen JJ, Chan P, Paes B, Mitchell I, Li A, Lanctôt KL, et al. Serious Adverse Events in the Canadian Registry of Children Receiving Palivizumab (CARESS) for Respiratory Syncytial Virus Prevention. PLoS One. (2015);10(8):e0134711.
- 20. Whelan KT, Pathan AA, Sander CR, Fletcher HA, Poulton I, Alder NC, et al. Safety and Immunogenicity of Boosting BCG Vaccinated Subjects with BCG: Comparison with Boosting with a New TB Vaccine, MVA85A. Plos one. (2009);4(6): e5934. doi:10.1371/journal.pone.0005934.
- 21. Bont L, Versteegh J, Swelsen WT, Heijnen CJ, Kavelaars A, Brus F, et al. Natural reinfection with respiratory syncytial virus does not boost virus-specific T-cell immunity. Pediatric research. (2002) Sep;52(3):363-7. doi: 10.1203/00006450-200209000-00009. PubMed PMID: 12193668.
- 22. Hall CB, Walsh EE, Long CE, Schnabel KC. Immunity to and frequency of reinfection with respiratory syncytial virus. J Infect Dis (1991);163:4.